

| Sponsor | Mirum Pharmaceuticals, Inc. |
|---|---|
| Protocol Title: | Randomized Double-blind Placebo-controlled Phase 3 Study to Evaluate the Efficacy and Safety of Maralixibat in the Treatment of Children with Progressive Familial Intrahepatic Cholestasis (PFIC) – MARCH-PFIC |
| Protocol Number: | MRX-502 |
| Premier Research PCN: | MIRU8967 |
| Document Version: | Final Version 2.0 |
| Document Date: | 29Sep2022 |

## **Approvals**

| Role | Signatures |
|---|---|
| | Print Name: Jana Steinmetz |
| Biostatistician | Sign Name: DocuSigned by: Jana Steinmety Signer Name: Jana Steinmetz Signing Reason: I am the author of this document Signing Time: 29-Sep-2022 17:56:37 EDT 9302752519E1436089832B622B6DE775 |
| | Print Name: Mary Poole |
| Peer Reviewer | Sign Name: DocuSigned by: Many Poole Signer Name: Mary Poole Signing Reason: I have reviewed this document Signing Time: 30-Sep-2022 15:51:33 EDT 85955933B2AB4430B05982AEEF99AC8B |





| Role | Signatures |
|---|---|
| | Print Name: Will Garner |
| Mirum Pharmaceuticals, Inc. Representative | Sign Name: DocuSigned by: Will Garner Signer Name: Will Garner Signing Reason: I approve this document Signing Time: 30-Sep-2022 17:39:35 EDT 2924BA8492304DB89A4DF5C7F56C3585 |
| | Print Name: Tiago Nunes |
| Mirum Pharmaceuticals, Inc. Representative | Sign Name: DocuSigned by: Virtago Mures Signer Name: Tiago Nunes Signing Reason: I approve this document Signing Time: 03-Oct-2022 00:52:11 PDT 2C1A401070C04C91B99CAA4F3DFC580F |



# **Document History**

| Version | Date | Change(s) | Author |
|---|---|---|---|
| 1.0 | 21Sep2022 | Initial version | Jana Steinmetz |
| 2.0 | 29Sep2022 | Minor: Update document header to read | Jana Steinmetz |
| | | 'Protocol Number MRX-502 (Amendment 4)' | |
| | | across all pages; some pages in Version 1.0 did | |
| | | not include '(Amendment 4)' | |





## **Table of Contents**

| Approvals | 1 |
|-------------------------------------------------------|----|
| Document History | 3 |
| Table of Contents | 4 |
| List of Tables | 6 |
| List of Figures | 7 |
| List of Abbreviations | |
| 1. Overview | |
| 2. Study Objectives and Endpoints | |
| 2.1. Study Objectives | 11 |
| 2.1.1. Primary Objective | 11 |
| 2.1.2. Secondary Objectives | 11 |
| 2.1.3. Exploratory Objectives | |
| 2.2. Study Endpoints | |
| 2.2.1. Safety Endpoints | 13 |
| 2.2.2. Efficacy Endpoints | |
| 2.2.2.1. Primary Efficacy Endpoint | 13 |
| 2.2.2.2. Secondary Efficacy Endpoints | |
| 2.2.2.3. Exploratory Efficacy Endpoints | |
| 2.2.3. Other Endpoints | 17 |
| 3. Overall Study Design and Plan | |
| 3.1. Overall Design | 17 |
| 3.2. Sample Size and Power | 20 |
| 3.3. Study Population | 21 |
| 3.4. Treatments Administered | 21 |
| 3.4.1. Dose Escalation Period | |
| 3.4.2. Stable Dosing Period | 22 |
| 3.5. Method of Assigning Subjects to Treatment Groups | 22 |
| 3.6. Blinding and Unblinding | |
| 3.7. Schedule of Assessments | 23 |
| 4. Statistical Analysis and Reporting | 27 |
| 4.1. Introduction | |
| 4.2. Interim Analysis and Data Monitoring | 28 |
| 5. Analysis Populations | 28 |



| | 5.1. Subject Grouping | 29 |
|---|---|---|
| 6. | General Issues for Statistical Analysis | 29 |
| | 6.1. Statistical Definitions and Algorithms | 29 |
| | 6.1.1. Baseline | 29 |
| | 6.1.2. Adjustments for Covariates | 30 |
| | 6.1.3. Multiple Comparisons | 30 |
| | 6.1.4. Handling of Dropouts or Missing Data | 31 |
| | 6.1.4.1. MMRM Analysis Method | 32 |
| | 6.1.4.2. Multiple Imputation Methods | 33 |
| | 6.1.4.3. Missing ItchRO/EDQ/PedsQL Scores | 41 |
| | 6.1.4.4. Missing Responder Definition Data | 41 |
| | 6.1.4.5. Missing Adverse Event Severity/Relationship | 42 |
| | 6.1.5. Analysis Visit Windows | 42 |
| | 6.1.6. Investigative Sites | 43 |
| | 6.1.7. Treatment Period Definitions | 43 |
| | 6.1.8. Derived Variables | 43 |
| | 6.1.9. Data Adjustments/Handling/Conventions | 50 |
| 7. | Study Subjects and Demographics | 55 |
| | 7.1. Disposition of Subjects and Withdrawals | 55 |
| | 7.2. Protocol Violations and Deviations | 56 |
| | 7.3. Demographics and Other Baseline Characteristics | 56 |
| | 7.4. Prior Medications/Therapies | 58 |
| | 7.5. Exposure and Compliance | 58 |
| 8. | Efficacy Analysis | 59 |
| | 8.1. Primary Efficacy Analysis | 59 |
| | 8.2. Secondary Efficacy Analysis | 61 |
| | 8.3. Sensitivity and Supportive Analyses for Primary and Secondary Endpoints | 62 |
| | 8.4. Adjustment for Multiplicity | 63 |
| | 8.5. Exploratory Efficacy Analysis | 63 |
| 9. | Safety and Tolerability Analysis | 64 |
| | 9.1. Adverse Events | |
| | 9.1.1. Adverse Events Leading to Discontinuation of Study Drug | |
| | 9.1.2. Deaths and Serious Adverse Events | 66 |
| | 9.1.3. Events of Clinical Interest | 66 |

AD-PR-109.02 Effective date: 17-Aug-2020



| 9.2. | Clinical Laboratory Evaluations | 6 / |
|-----------|--------------------------------------------------------|-----|
| 9.3. | Vital Signs and Weight/Height Measurements | 67 |
| 9.4. | Electrocardiograms | 67 |
| 9.5. | Liver Ultrasound | 67 |
| 9.6. | Concomitant Medications/Therapies | 67 |
| 10. O | ther Planned Analysis | 68 |
| 10.1. | Healthcare Utilization | 68 |
| 10.2. | Pharmacokinetic Analyses | 68 |
| 11. Cl | hanges from Protocol Planned Analysis | 68 |
| 12. Re | eferences | 71 |
| | ables, Listings, and Figures | |
| | Planned Table Descriptions | |
| | 1.1. Subject Data | |
| | 1.2. Efficacy Data | |
| | 1.3. Safety Data | |
| | 1.4. Other Data | |
| | Planned Figure Descriptions | |
| | 2.1. Efficacy Data | |
| 13.3. | $\mathcal{E}$ | |
| 13.4. | Standard Layout for all Tables, Listings, and Figures | |
| | 11: Listing of Safety and Efficacy Laboratory Analytes | |
| Appendix | 2: Listing of Lipid Soluble Vitamin Deficiency Events | 89 |
| List of T | Γables | |
| Table 1: | Schedule of Assessments | 24 |
| Table 2: | Analysis Visit Windows | 42 |
| Table 3: | Subject Data Summary Tables | 73 |
| Table 4: | Efficacy Data Summary Tables | 74 |
| Table 5: | Safety Data Summary Tables | 81 |
| Table 6: | Other Data Summary Tables | 82 |
| Table 7: | Efficacy Data Summary Figures | 83 |





# **List of Figures**

| Figure 1. | Study Design Flow Chart | 19 |
|-----------|-------------------------|----|
| Figure 2. | Standardized Layout | 86 |



## **List of Abbreviations**

| Abbreviation | Definition |
|---------------------------|-----------------------------------------|
| ALGS | alagille syndrome |
| APRI | AST to platelet ratio index |
| ATC | anatomical therapeutic chemical |
| BID | twice daily |
| BL | baseline |
| C4 | 7α hydroxyl-4-cholesten-3-one |
| CI | confidence interval |
| CIS | caregiver impression of severity |
| СМН | Cochran-Mantel-Haenszel |
| CSS | clinician scratch scale |
| DMC | data monitoring committee |
| ECI | events of clinical interest |
| EDQ | exploratory diary questionnaire |
| EM | expectation-maximization |
| ЕОТ | end of treatment |
| ET | early termination |
| FGF-19 | fibroblast growth factor-19 |
| FIB-4 | fibrosis-4 |
| НСС | hepatocellular carcinoma |
| INR | international normalized ratio |
| ItchRO <sup>TM</sup> | Itch Reported Outcome |
| ItchRO(Obs) <sup>TM</sup> | Observer-reported Itch Reported Outcome |
| ItchRO(Pt)TM | Patient-reported Itch Reported Outcome |
| IRT | interactive response technology |
| K-M | Kaplan-Meier |
| LLOQ | lower limit of quantitation |



| Abbreviation | Definition |
|--------------|--------------------------------------------------|
| LS | least squares |
| LSV | lipid soluble vitamin |
| MAR | missing at random |
| MCMC | Markov-Chain Monte-Carlo |
| MELD | Model for End-Stage Liver Disease |
| MI | multiple imputation |
| MMRM | mixed-effects model for repeated measurements |
| MNAR | missing not at random |
| nt-PFIC2 | non-truncating PFIC2 |
| Obs | observer |
| PEBD | partial external biliary diversion |
| PedsQL | pediatric quality of life |
| PELD | Pediatric End-Stage Liver Disease |
| PFIC | progressive familial intrahepatic cholestasis |
| PIS | patient impression of severity |
| PRO | patient reported outcomes |
| Pt | patient |
| PT | preferred term |
| QTcB | QT interval corrected using Bazett's formula |
| QTcF | QT interval corrected using Fridericia's formula |
| REML | restricted maximum likelihood |
| SAE | serious adverse event |
| sBA | serum bile acid |
| SD | standard deviation |
| SE | standard error |
| SI | International System of Units |
| SOC | system organ class |



| Abbreviation | Definition |
|--------------|---------------------------------------------|
| t-PFIC2 | truncating PFIC2 |
| TEAE | treatment-emergent adverse event |
| TESAE | treatment-emergent serious adverse event |
| TSB | otal serum bilirubin |
| UDCA | ursodeoxycholic acid |
| ULN | upper limit normal |
| ULOQ | upper limit of quantitation |
| VAP | validation analysis plan |
| WHO | World Health Organization |
| WHO-DD | World Health Organization - Drug Dictionary |



#### 1. Overview

This statistical analysis plan (SAP) describes the planned analysis and reporting for Mirum Pharmaceuticals, Inc. protocol number MRX-502 (Randomized Double-blind Placebo-controlled Phase 3 Study to Evaluate the Efficacy and Safety of Maralixibat in the Treatment of Subjects with Progressive Familial Intrahepatic Cholestasis [PFIC]), Amendment 4, dated 10-May-2022. Reference materials for this statistical plan include the protocol and the accompanying sample data collection documents. Operational aspects related to collection and timing of planned clinical assessments are not repeated in this SAP unless relevant to the planned analysis.

The structure and content of this SAP provides sufficient detail to meet the requirements identified by the Food and Drug Administration (FDA), European Medicines Agency (EMA), and International Conference on Harmonization (ICH) of Technical Requirements for Registration of Pharmaceuticals for Human Use: Guidance on Statistical Principles in Clinical Trials (ICH, 1998). All work planned and reported for this SAP will follow internationally accepted guidelines, published by the American Statistical Association (ASA, 2018) and the Royal Statistical Society (RSS, 2014), for statistical practice.

The planned analyses identified in this SAP may be included in clinical study reports (CSRs), regulatory submissions, or future manuscripts. Also, post-hoc exploratory analyses not necessarily identified in this SAP may be performed to further examine study data. Any post-hoc or unplanned, exploratory analysis performed will be clearly identified as such in the final CSR.

The statistical plan described hereafter is an a priori plan. It will be submitted to file prior to any unblinded inferential or descriptive analysis of data pertaining to Mirum Pharmaceuticals, Inc.'s study MRX-502.

### 2. Study Objectives and Endpoints

### 2.1. Study Objectives

### 2.1.1. Primary Objective

The primary objective is to evaluate the efficacy of maralixibat vs. placebo on the *severity of pruritus* in the primary cohort, as defined in Section 5.1.

### 2.1.2. Secondary Objectives

The secondary objectives are:

- To evaluate the efficacy of maralixibat vs. placebo on total serum bile acid (sBA) levels in the primary cohort
- To evaluate the efficacy of maralixibat vs. placebo on the *severity of pruritus* in the PFIC cohort, as defined in Section 5.1



- To evaluate the efficacy of maralixibat vs. placebo on total sBA levels in the PFIC cohort
- To evaluate the efficacy of maralixibat vs. placebo on the ItchRO(Obs) responder rate in the primary cohort.
- To evaluate the efficacy of maralixibat vs. placebo on the sBA responder rate in the primary cohort.
- To evaluate the efficacy of maralixibat vs. placebo on the ItchRO(Obs) responder rate in the PFIC cohort.
- To evaluate the efficacy of maralixibat vs. placebo on the sBA responder rate in the PFIC cohort.
- To evaluate the safety, tolerability, and pharmacokinetics (PK) of maralixibat vs. placebo in all participants who received at least 1 dose of study medication (Safety Population)

### 2.1.3. Exploratory Objectives

The exploratory objectives are:

- To evaluate the efficacy of maralixibat vs placebo in the primary cohort and in the PFIC cohort on the following parameters:
  - Liver biochemistry
  - Non-invasive fibrosis markers: Fibrosis-4 (FIB-4), AST to Platelet Ratio Index (APRI), pediatric end-stage liver disease (PELD) score, model for end-stage liver disease (MELD) score
  - Other measures of pruritus including ItchRO(Obs), for parameters not utilized for primary and secondary objectives, ItchRO(Pt), CSS and other Patient Reported Outcomes (PRO), including Caregiver Impression of Severity (CIS), Patient Impression of Severity of Pruritus (PIS), and Exploratory Diary Questionnaire (EDQ)
  - o Responder rates for pruritus severity and total sBA
  - Health-related quality of life
  - Quality of sleep
  - Subject growth
  - o Markers of bile acid metabolism: Bile acid subspecies, C4, FGF-19, autotaxin
  - Time to liver-associated events
- To evaluate the impact of maralixibat on healthcare utilization
- To evaluate the correlation between sBA and severity of pruritus in terms of levels and changes from baseline



### 2.2. Study Endpoints

### 2.2.1. Safety Endpoints

The safety and tolerability endpoints of this study include the following:

- Incidence of adverse events (AEs) including serious, related to study drug, leading to withdrawal, events of clinical interest, along with AEs by severity and by relationship to study drug
- Change from baseline in clinical laboratory values
- Change from baseline in physical examination findings (including body weight, height, and BMI)
- Change from baseline in vital signs
- Change from baseline in electrocardiogram (ECG) measures
- Concomitant treatment usage

Vital signs include heart rate, respiratory rate, body temperature, and blood pressure.

Safety laboratory tests, and associated units of measure, that will be used for reporting are listed in Appendix 1. Note that bilirubin (total and direct), alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), GGT, FGF-19, and total sBA are considered as both safety and efficacy laboratory tests.

### 2.2.2. Efficacy Endpoints

For the sequential (hierarchical) testing and the specific study populations used for each primary and secondary endpoints, please refer to Section 6.1.3 (Multiple Comparisons).

### 2.2.2.1. Primary Efficacy Endpoint

The primary efficacy endpoint of this study is defined as the mean change in the average morning ItchRO(Obs) severity score between baseline and Week 15 through Week 26, using 4-week average morning ItchRO(Obs) severity scores in the primary cohort.

### 2.2.2.2. Secondary Efficacy Endpoints

The secondary efficacy endpoints of this study include the following:

- Mean change in total sBA level between baseline and average of Weeks 18, 22, and 26 in the primary cohort (considered as the <u>key</u> secondary endpoint)
- Mean change in the average morning ItchRO(Obs) severity score between baseline and Week 15 through Week 26, using 4-week average morning ItchRO(Obs) severity scores in the PFIC cohort



- Mean change in total sBA level between baseline and average of Weeks 18, 22, and 26 in the PFIC cohort
- Proportion of ItchRO(Obs) responders from Week 15 to Week 26 (reference Section 6.1.8) in the primary cohort
- Proportion of sBA responders from Week 18 to Week 26 (reference Section 6.1.8) in the primary cohort
- Proportion of ItchRO(Obs) responders from Week 15 to Week 26 (reference Section 6.1.8) in the PFIC cohort
- Proportion of sBA responders from Week 18 to Week 26 (reference Section 6.1.8) in the PFIC cohort

### 2.2.2.3. Exploratory Efficacy Endpoints

The exploratory efficacy endpoints of this study will be evaluated in the primary cohort and the PFIC cohort, unless otherwise noted, and include the following:

- Mean change from baseline in total sBA level to Weeks 2, 6, 10, 14, 18, 22, and 26
- Mean change from baseline in liver-associated laboratory test levels (i.e., ALT, AST, ALP, total bilirubin, direct bilirubin, GGT, albumin) to Weeks 2, 6, 10, 14, 18, 22, 26, and average of Weeks 18, 22, and 26
- Mean change from baseline in FIB-4, APRI, MELD and PELD score to Weeks 2, 6, 10, 14, 18, 22, 26, and average of Weeks 18, 22, and 26
- Mean change from baseline in average morning ItchRO(Obs) severity scores to Week 6, 10, 14, 18, 22, and 26, using 6-week average for Week 6 and 4-week average afterwards
- Mean change from baseline in average evening ItchRO(Obs) severity scores to Weeks 6, 10, 14, 18, 22, 26, using 6-week average for Week 6 and 4-week average afterwards, and Weeks 15 to 26 combined
- Mean change from baseline in average highest daily ItchRO(Obs) severity scores to Weeks 6, 10, 14, 18, 22, 26, using 6-week average for Week 6 and 4-week average afterwards, and Weeks 15 to 26 combined
- Mean change from baseline in average morning ItchRO(Obs) frequency scores to Weeks 6, 10, 14, 18, 22, 26, using 6-week average for Week 6 and 4-week average afterwards, and Weeks 15 to 26 combined
- Mean change from baseline in average evening ItchRO(Obs) frequency scores to Weeks 6, 10, 14, 18, 22, 26, using 6-week average for Week 6 and 4-week average afterwards, and Weeks 15 to 26 combined



- Mean change from baseline in average highest daily ItchRO(Obs) frequency scores to Weeks 6, 10, 14, 18, 22, 26, using 6-week average for Week 6 and 4-week average afterwards, and Weeks 15 to 26 combined
- Mean change from baseline in average morning ItchRO(Pt) severity scores to Weeks 6, 10, 14, 18, 22, 26, using 6-week average for Week 6 and 4-week average afterwards, and Weeks 15 to 26 combined
- Mean change from baseline in average evening ItchRO(Pt) severity scores to Weeks 6, 10, 14, 18, 22, 26, using 6-week average for Week 6 and 4-week average afterwards, and Weeks 15 to 26 combined
- Mean change from baseline in average highest daily ItchRO(Pt) severity scores to Weeks 6, 10, 14, 18, 22, 26, using 6-week average for Week 6 and 4-week average afterwards, and Weeks 15 to 26 combined
- Mean change from baseline in average morning ItchRO(Pt) frequency scores to Weeks 6, 10, 14, 18, 22, 26, using 6-week average for Week 6 and 4-week average afterwards, and Weeks 15 to 26 combined
- Mean change from baseline in average evening ItchRO(Pt) frequency scores to Weeks 6, 10, 14, 18, 22, 26, using 6-week average for Week 6 and 4-week average afterwards, and Weeks 15 to 26 combined
- Mean change from baseline in average highest daily ItchRO(Pt) frequency scores to Weeks 6, 10, 14, 18, 22, 26, using 6-week average for Week 6 and 4-week average afterwards, and Weeks 15 to 26 combined
- Number of days with a morning ItchRO(Obs) severity score ≤1 at the participant level for the last 84 days (i.e., study day 99 through 182, inclusive) of the study
- Mean change from baseline in CSS at Weeks 2, 4, 6, 10, 14, 18, 22, 26, and Weeks 18, 22, and 26 combined
- Mean change from baseline in CIS at Weeks 4, 6, 10, 14, 18, 22, 26, and Weeks 18, 22, and 26 combined
- Mean change from baseline in PIS at Weeks 4, 6, 10, 14, 18, 22, 26, and Weeks 18, 22, and 26 combined
- Mean change from baseline in average morning EDQ(Obs) severity scores to Weeks 6, 10, 14, 18, 22, 26, using 6-week average for Week 6 and 4-week average afterwards, and Weeks 15 to 26 combined
- Mean change from baseline in average evening EDQ(Obs) severity scores to Weeks 6, 10, 14, 18, 22, 26, using 6-week average for Week 6 and 4-week average afterwards, and Weeks 15 to 26 combined



- Mean change from baseline in average highest daily EDQ(Obs) severity scores to Weeks 6, 10, 14, 18, 22, 26, using 6-week average for Week 6 and 4-week average afterwards, and Weeks 15 to 26 combined
- Number and proportion of participants achieving morning ItchRO(Obs) severity scores ≤1 for more than 50% of the time from post-baseline to Week 6, Weeks 7 to 10, Weeks 11 to 14, Weeks 15 to 18, Weeks 19 to 22, Weeks 23 to 26, and Week 15 to Week 26
- Mean change from baseline over time in quality of life as measured by the PedsQL (parent) total scale score at Weeks 4, 6, 10, 14, 18, 22, 26, and Weeks 18, 22, and 26 combined
- Mean change from baseline in average morning EDQ(Obs) sleep disturbance scores to Weeks 6, 10, 14, 18, 22, and 26, using 6-week average for Week 6 and 4-week average afterwards, and Weeks 15 to 26 combined
- Proportion of participants with improvement from baseline (i.e., change from baseline <0) in morning EDQ(Obs) sleep disturbance score at Weeks 6, 10, 14, 18, 22, and 26, using 6-week average scores for Week 6 and 4-week average scores afterwards
- Proportion of morning EDQ(Obs) sleep disturbance scores ≤2 at the participant level post-baseline through Week 26
- Mean change from baseline in height z-score and weight z-score at Weeks 2, 4, 6, 10, 14, 18, 22, 26, and Weeks 18, 22, and 26 combined
- Mean change and % change from baseline in total sBA level to Weeks 2, 6, 10, 14, 18, 22, 26, and Weeks 18, 22, and 26 combined
- Number and proportion of subjects with total sBA % decrease from baseline to Weeks 2, 6, 10, 14, 18, 22, and 26 within the following categories: >75%, 0-75%, and <0%
- Mean change from baseline in C4, FGF-19, and autotaxin to Weeks 6, 10, 18, and 26 in the primary cohort
- Time to first liver-associated event (PEBD surgery, listing for liver transplantation, liver decompensation [hepatic encephalopathy, variceal bleeding, ascites, and spontaneous bacterial peritonitis] events, HCC, death)

Severity scores for the EDQ are based on the EDQ(Obs) question of "How bad was your child's itch at its worst?" and on the EDQ(Pt) question of "How bad was your itch at its worst". "Non-severity" scores are based on all other EDQ questions.

To assess possible improvements in sleep, the sleep-related question from the EDQ(Obs) questionnaire will be summarized. For EDQ(Obs), sleep disturbance is assessed on the morning diary through the question, "Because of itch, my child had trouble staying asleep". Responses are scored on a 5-point scale, where 1=Never, 2=Rarely, 3=Sometimes, 4=Often, and 5=Almost Always. For the EDQ sleep-related question, 6-week average scores will be derived for Weeks 1-6 and 4-week average scores will be derived for the remaining time periods.



### 2.2.3. Other Endpoints

Other endpoints of this study include the following and will be evaluated in the primary cohort, the PFIC cohort, and all cohorts combined (i.e., all subjects):

- Impact of maralixibat treatment on healthcare utilization (incidence of PFIC-related hospitalization, total inpatient days, selected surgical procedures, emergency room visits, and caregiver days missed from work, etc.) between clinic visits from baseline through Week 27 follow-up visit.
- Plasma levels of maralixibat at pre-dose and approximately 2.5 hours after the morning dose at Week 10 and Week 26 (EOT/ET).

### 3. Overall Study Design and Plan

### 3.1. Overall Design

This is a 6-month international, multicenter, randomized, double-blind, placebo-controlled phase 3 study in participants with PFIC who are ≥12 months and <18 years of age at time of baseline. This study will be followed by a long-term extension study (MRX-503), during which all participants who complete study MRX-502 will have the opportunity to be treated with maralixibat.

Subjects in the primary cohort will be randomized in a 1:1 ratio to receive maralixibat or placebo. Subjects in the supplemental cohort will be randomized in a 1:1 ratio to receive maralixibat or placebo within the following subcohorts: a) PFIC1; b) PFIC3; c) all other supplemental cohort subjects.

For the purposes of the randomization stratification and enrollment objectives, the primary and supplemental cohorts are defined as follows:

- Primary cohort, defined as participants with genetic testing results consistent with biallelic disease-causing variation in *ABCB11* (PFIC2), based on standard of care genotyping, excluding those PFIC2 participants with complete absence of bile salt excretion pump (BSEP) function, and do not fall under the definition of the supplemental cohort.
- Supplemental cohort, defined as:
  - o Subjects with genetic testing results consistent with biallelic disease causing variation in ATP8B1 (PFIC1), ABCB4 (PFIC3), or TJP2 (PFIC4), based on standard-of-care genotyping
  - o Subjects with PFIC phenotype without a known mutation or with another known mutation not described above or with intermittent cholestasis as manifested by fluctuating sBA levels



o Subjects with PFIC after internal or external biliary diversion surgery or for whom internal or external biliary diversion surgery was reversed

Further information about the treatment allocation is provided in Section 3.5.

In the primary cohort, approximately 30 participants will be enrolled in order to achieve 26 participants (13 per treatment group) completing the study. In the supplemental cohort, overall enrollment will be capped at a maximum of 60 participants.

The primary analysis will be conducted in the ITT population of participants in the primary cohort. For analysis purposes, post-randomization cohort definitions have been defined (see Section 5.1).

The study will be divided into 4 parts:

- 1. Screening period (up to 6 weeks)
- 2. Dose Escalation period (4-6 weeks)
- 3. Stable Dosing period (20-22 weeks)
- 4. Safety Follow-up period (7 days from the last dose of study drug for participants not continuing into the extension study [MRX-502])



Figure 1. Study Design Flow Chart



<sup>&</sup>lt;sup>a</sup> Dose escalation may occur over 4-6 weeks depending on tolerability. Stable dosing will occur over 20-22 weeks, depending on the duration of the dose escalation period.
<sup>b</sup> Safety follow-up visit for subjects not continuing into the extension study (MRX-503).

BID=twice daily; Scr=screening; V=visit; W=week

Subjects randomized to placebo will remain on placebo for the entire duration of the study. The Dose Escalation period will consist of the following weekly steps:

Dose level 1: 150 µg/kg maralixibat BID for 1 week

Dose level 2: 300 μg/kg maralixibat BID for 1 week

Dose level 3: 450 µg/kg maralixibat BID for 1 week

Dose level 4: 600 μg/kg maralixibat BID for the remaining duration of the study

Study drug is administered twice daily over a 26-week treatment period. A participant's maximum duration of participation is expected to be up to 33 weeks.

At the end of the 26-week double-blind treatment period, participants will have the opportunity to enroll into the long-term, extension study (MRX-503). Subjects who do not enroll into the treatment extension study or who discontinue at any time during this study will have a final safety follow-up phone call 7 days after the last dose of study drug. Subjects who discontinue from the study for safety reasons are followed-up as long as clinically indicated or until no further improvement with an adverse event is expected.

AD-ST-33.06 Effective date: 12-Nov-2020

Final Version 2.0 | 29-Sep-2022 | AD-PR-109.02 Effective date: 17-Aug-2020 | Page 19 of 89



The study will be conducted in approximately 40 sites in North America, Europe, Asia, and South America. Other regions may be added, if necessary, for enrollment purposes.

### 3.2. Sample Size and Power

The sample size was calculated to ensure enrollment of an adequate number of PFIC2 participants who fulfill criteria for the primary cohort (primary endpoint). The sample size is chosen to provide at least 80% of power for the analysis of the primary endpoint.

The primary efficacy endpoint is the mean change from baseline in the average morning ItchRO(Obs) severity score for the last 12 weeks of the study (Weeks 15-26).

The following assumptions were made in estimating the sample size for study MRX-502:

- Between-treatment group (placebo to active) LS mean difference of 0.663
- Pooled SD of 0.563
- Effect size of 1.178 in the mean change from baseline in the 4-week average morning ItchRO(Obs) score

The estimations of LS mean difference, SD and effect size for the sample size justification are based on ItchRO(Obs) data from the maralixibat Phase 2 studies. Maralixibat-treated subjects with PFIC2 from Study LUM001-501 were compared to placebo-treated subjects with ALGS from Studies LUM001-301 and LUM001 302 as no placebo data are available from Study LUM001-501. Since impact and symptoms of itching reported by PFIC patients are also reported by ALGS patients, (i.e., mood changes, scratching, difficulty falling asleep, skin damage, blood from scratching etc.), it is reasonable to assume that the ItchRO outcomes from the ALGS placebo-controlled studies will inform outcomes for this PFIC study due to the similarities in the features of pruritus. Two fundamental assumptions were made: A) the placebo effect in subjects with ALGS is similar to the one expected in subjects with PFIC2. Subjects with ALGS in study LUM001-301/302 had a slightly higher BL ItchRO(Obs) value compared to subjects with PFIC in Study LUM001-501. As subjects with higher BL pruritus generally report a higher placebo response, the use of ALGS subjects from study LUM001-301/302 would therefore lead to a slightly more conservative assumption of the expected effect and sample size. The 2 populations were similar in the other BL characteristics. Besides from the small difference in BL characteristics there are no obvious reasons to believe why the placebo response in subjects with ALGS and PFIC should be difference. Therefore, the comparison of ALGS placebo subjects with treated PFIC subjects is considered a valid approximation for the purpose of assessing the effect size, data variability and the calculation of the sample size. B) the placebo effect does not change after 3 months of treatment; as Studies LUM001-301 and -302 were 13week studies, data beyond 13 weeks were imputed using the last observation carried forward.

With the assumed values, a total of 26 complete subjects (13 subjects in each treatment group) will be required to provide 80% power for the comparison of the primary endpoint measure between



the maralixibat treatment group and placebo, based on a 2-sided, 2-sample t-test at the 0.05 level of significance.

Including a 10% dropout rate based on the previous PFIC study and rounding up to the next even number, approximately 30 participants (15 participants in each treatment group) will be randomized in the primary cohort of the study.

### 3.3. Study Population

The study population is comprised of male and female participants with a body weight  $\geq 5.0$  kg, who are  $\geq 12$  months and  $\leq 18$  years of age at time of baseline, with a confirmed diagnosis of PFIC based on clinical/laboratory features and standard of care genotyping. Subjects will not be considered eligible for the study without having cholestasis as manifested by total sBA (primary cohort only)  $\geq 3$  x ULN (upper limit normal) and an average morning ItchRO(Obs) severity score  $\geq 1.5$  during 4 consecutive weeks leading to the baseline visit.

#### 3.4. Treatments Administered

Subjects will be randomized to one of two treatment groups:

- maralixibat
- placebo

Eligible participants will be randomly assigned to study drug in a 1:1 allocation ratio, stratified by cohort (see Section 3.1). Subjects will self-administer (or will be administered) varying volumes of ready-to-use oral solution study drug at each dosing visit, starting with the baseline visit (Visit 1/Day 0). The dosing volume is determined based on the individual body weight, the dose level according to the dose escalation plan (150, 300, 450 or 600  $\mu$ g/kg), and the strength of solution being administered (5, 10, 15, or 20 mg/mL).

Subjects will take the first dose of study drug at the baseline visit (Visit 1/Day 0) under the supervision of the Investigator or trained staff.

Study drug administration will take place during the Dose Escalation and Stable Dosing periods of the study based on a BID regimen. The morning dose should be administered approximately 30 minutes before breakfast and the evening dose approximately 30 minutes before the main evening meal. The doses will be administered prior to meals rather than q12h in order to better cover the luminal bile acid release associated with meals. Study drug should be administered approximately at the same time each day throughout the study. The interval between administration of study drug and any concomitant treatment should not change during the study.

Dosing will occur over a 26-week treatment period.



#### 3.4.1. Dose Escalation Period

For participants assigned to maralixibat, the Dose Escalation period will consist of the following weekly steps:

- Dose level 1: 150 μg/kg maralixibat BID for 1 week
- Dose level 2: 300 μg/kg maralixibat BID for 1 week
- Dose level 3: 450 μg/kg maralixibat BID for 1 week
- Dose level 4: 600 μg/kg maralixibat BID for the remaining duration of the study

Dose escalation should occur in the absence of major safety (e.g., liver parameters) or tolerability (e.g., GI-related TEAEs) concerns related or possibly related to study medication. Subjects with such safety concerns can be down-titrated to a lower, previously tolerated dose level for 1 week before continuing dose escalation. The minimum dose to continue in the study will be 150  $\mu$ g/kg maralixibat BID; subjects who cannot tolerate this dose will be discontinued from the study.

### 3.4.2. Stable Dosing Period

Investigators have up to Week 6 to determine the maximum tolerated dose; if re-challenges or further dose escalations fail, the participant will remain on the maximum tolerated dose level for the remainder of the Stable Dosing period to complete a minimum of 20 weeks of stable dosing.

During the Stable Dosing period, participants will remain on the maximum tolerated dose level for the remainder of the study. Dose reductions are allowed for safety or tolerability reasons down to a minimum level of 150  $\mu$ g/kg BID. Subjects who cannot tolerate this dose will be discontinued from the study.

### 3.5. Method of Assigning Subjects to Treatment Groups

Subjects who meet study entry criteria will be randomly assigned to maralixibat or placebo in a 1:1 allocation ratio. The randomization schedule will be computer generated by an independent biostatistician using a permuted block algorithm and will randomly allocate each treatment group to randomization numbers. The randomization numbers will be assigned sequentially through a central interactive response technology (IRT) system as participants are entered into the study. The randomization schedule will be stratified by cohort as described in Section 3.1.

The IRT system will be used for screening and enrolling participants, randomization, study drug supply dispensation and management, inventory management and supply ordering, study drug expiration tracking and management, and emergency unblinding. Individual participant treatment is automatically assigned by the IRT to participants who meet study entry criteria. The participant's randomization number represents a unique number corresponding to the treatment allocated to the participant.



At each dosing visit, the Investigator or designee will access the IRT system, and enter participant-specific information (e.g., unique participant number, age [years and months], weight, and information on dose escalation status). For randomized participants, this information will be used by the IRT to identify the appropriate strength of solution and dosing volume, and to assign a corresponding bottle number(s) to be dispensed to the participant.

Siblings enrolled in the study will be assigned in a blinded manner by the IRT system to the same treatment arm.

The randomization schedule will be prepared by Premier Research before the start of the study. No one involved in the study performance will have access to the randomization schedule before the official unblinding of treatment assignment. Subjects who discontinue from the study will not be replaced. Study center will not be a blocking factor in the randomization schedule.

### 3.6. Blinding and Unblinding

All participants, investigators, and study personnel involved in the conduct of the study, including data management, will be blinded to treatment assignment.

The treatment assignment must not be unblinded during the study except in emergency situations where the identification of the study drug is required for further treatment of the participant. The Investigator should make an effort to contact the medical monitor before unblinding occurs or as soon as possible after the Investigator has been unblinded without revealing the treatment assignment to the medical monitor. In any event, the medical monitor and Sponsor must be informed about the code break as soon as possible.

If the treatment assignment is unblinded, the date and the signature of the person who was unblinded, and the reason for unblinding are recorded in the source documents. Upon breaking the blind, the participant will be withdrawn from the study, but should be followed up for safety purposes. Unblinding will be processed through the IRT system, and instructions will be available in the user manual.

Data that may potentially unblind treatment assignment (i.e., maralixibat serum concentrations, treatment allocation, post-baseline sBA levels) will be handled with special care during the data cleaning and review process. Prior to unblinding, any data that may potentially unblind study site personnel or study team personnel will be presented as blinded information or otherwise will not be made available. If applicable, unblinded data may be made available to quality assurance representatives for the purposes of conducting independent audits.

### 3.7. Schedule of Assessments

A detailed schedule of assessment for the study is provided in Table 1.





**Table 1: Schedule of Assessments** 

| Procedures <sup>p</sup> | Screening a | Dose | e Escalation | (4-6 we | eks) | <br> | Stable Dosing (20-22 weeks) | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit/Subject Contact<br># | Screening /<br>V0 | Baseline<br>/ V1 | Subject contact | V2 | Subject contact | V3 | Subject contact | V4 | Subject contact | V5 | Subject contact | V6 | Subject contact | V7 | Subject contact | V8 | Subject contact | EOT/ET<br>V9 <sup>b</sup> | Follow-up |
| Study Week | -6 | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 8 | 10 | 12 | 14 | 16 | 18 | 20 | 22 | 24 | 26 | 27 |
| Study Day | Day -42 | 0 | 7 | 14 | 21 | 28 | 35 | 42 | 56 | 70 | 84 | 98 | 112 | 126 | 140 | 154 | 168 | 182 | 189 |
| Window (in days) | (-5) | | (±2) | (±2) | (±2) | (±2) | (±2) | (±2) | (±2) | (±3) | (±3) | (±3) | (±3) | (±3) | (±3) | (±3) | (±3) | (±3) | (±2) |
| Informed<br>Consent/Assent | X | | | | | | | | | | | | | | | | | | |
| Eligibility Assessment | X | X | | | | | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | | | | | | |
| Medical History | X | | | | | | | | | | | | | | | | | | |
| Physical & Vital signs <sup>c</sup> | X | X | | X | | X | | X | | X | | X | | X | | X | | X | |
| ECG | X | X | | | | | | | | X | | | | | | | | X | |
| Liver Ultrasound <sup>d</sup> | X | | | | | | | | | | | | | | | | | X | |
| Pregnancy Test <sup>e</sup> | S | U | | | | U | | U | | U | | U | | U | | U | | S | |
| Confirm PFIC<br>Genotype Results <sup>f</sup> | X | | | | | | | | | | | | | | | | | | |
| eDiary Device Provided<br>/ Returned <sup>g</sup> | P | | | | | | | | | | | | | | | | | R | |
| ItchRO(Obs),<br>ItchRO(Pt) & EDQ | | | | | | | Twi | ice-daily | completion ( | of ItchRO | O & EDQ | | | | | | | | |
| Review eDiary &<br>Assess Compliance | | X | | X | | X | | X | | X | | X | | X | | X | | X | |
| Randomized | | X | | | | | | | | | | | | | | | | | |
| CISh | | X | | | | X | | X | | X | | X | | X | | X | | X | |
| PISi | | X | | | | X | | X | | X | | X | | X | | X | | X | |
| PIC | | | | | | | | | | | | | | | | | | X | |
| CIC | | | | | | | | | | | | | | | | | | X | |





| Procedures <sup>p</sup> | Screening a | Dose | l<br>I | | Stable Dosing (20-22 weeks) | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit/Subject Contact<br># | Screening /<br>V0 | Baseline<br>/ V1 | Subject contact | V2 | Subject contact | V3 | Subject contact | V4 | Subject<br>contact | V5 | Subject contact | V6 | Subject contact | V7 | Subject contact | V8 | Subject contact | EOT/ET<br>V9 <sup>b</sup> | Follow-up |
| Study Week | -6 | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 8 | 10 | 12 | 14 | 16 | 18 | 20 | 22 | 24 | 26 | 27 |
| Study Day | Day -42 | 0 | 7 | 14 | 21 | 28 | 35 | 42 | 56 | 70 | 84 | 98 | 112 | 126 | 140 | 154 | 168 | 182 | 189 |
| Window (in days) | (-5) | | (±2) | (±2) | (±2) | (±2) | (±2) | (±2) | (±2) | (±3) | (±3) | (±3) | (±3) | (±3) | (±3) | (±3) | (±3) | (±3) | (±2) |
| $PedsQL^{j}$ | | X | | | | X | | X | | X | | X | | X | | X | | X | |
| Clinician Scratch Scale | X | X | | X | | X | | X | | X | | X | | X | | X | | X | |
| CBC with Differential | X | X | | X | | | | X | | X | | X | | X | | X | | X | |
| Coagulation | X | X | | X | | | | X | | X | | X | | X | | X | | X | |
| Chemistry Panel | X | X | | X | | | | X | | X | | X | | X | | X | | X | |
| Lipid Panel <sup>k</sup> | X | X | | X | | | | X | | X | | X | | X | | X | | X | |
| Urinalysis | | X | | | | | | X | | X | | | | X | | | | X | |
| FGF-19, Autotaxin, C4 <sup>k</sup> | | X | | | | | | X | | X | | | | X | | | | X | |
| sBA collection <sup>k</sup> | X | X | | X | | | | X | | X | | X | | X | | X | | X | |
| Lipid Soluble<br>Vitamins <sup>k,l</sup> | | X | | | | | | X | | X | | X | | X | | X | | X | |
| AFP Sample | | X | | | | | | | | X | | | | | | | | X | |
| PK Sample <sup>m</sup> | | | | | | | | | | X | | | | | | | | X | |
| Serum storage sample | | X | | X | | | | X | | X | | X | | X | | X | | X | |
| Healthcare Utilization | | | | X | | | | X | | X | | X | | X | | X | | X | X |
| Study drug Supplied <sup>n</sup> | | X | | X | | X | | X | | X | | X | | X | | X | | | |
| Study drug<br>Administration <sup>o</sup> | | | | | | | | | Twice-da | aily admi | nistration | | | | | | | | |
| Assess AEs | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Prior and Concomitant<br>Treatments | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |





AFP=a-fetoprotein; C4=7a-hydroxy-4-cholesten-3-one; CBC=complete blood count; CIS=Caregiver Impression of Severity; CIC=Caregiver Impression of Change; ECG=electrocardiogram; EDQ=exploratory diary questionnaire; EOT=end of treatment; ET=early termination; FGF-19=fibroblast growth factor-19; ItchRO=Itch Reported Outcome; P=Provided; PedsQL=Pediatric Quality of Life Inventory; PIC=Patient Impression of Change; PIS=Patient Impression of Severity of Pruritus; PK=pharmacokinetic; R=Returned; S=Serum; U= Urine; V=visit

- <sup>a</sup> Subjects who initially fail to meet eligibility criteria may be re-assessed during the 6-week screening period prior to being captured as a screen failure. Subjects may also be re-screened
- b Study sites should record dates of any future scheduled procedures related to PFIC (e.g., PEBD, ileal exclusion, liver transplant, or listed for liver transplant), if known at this visit
- Blood pressure, heart rate, temperature, respiration rate. Height and weight will be measured by trained staff using standardized methodology, incl. calibrated stadiometer or headboard and calibrated balance, respectively
- d Screening ultrasound not required if an ultrasound or liver MRI less than 6 months old is available
- <sup>e</sup> Females of childbearing potential only; result must be reviewed prior to dispensing study drug
- f Genotyping results will be reviewed by Sponsor or designee
- g Caregivers and age-appropriate participants will be instructed to complete their eDiary twice daily (morning and evening)
- h To be completed by caregivers for all participants
- To be completed only by participants aged ≥9 years at screening
- To be completed by participants and caregivers using the age-appropriate PedsQL module
- <sup>k</sup> Subjects should make every effort to fast at least 6 hours prior to collection. Water intake is permitted if necessary but not recommended
- Blood samples must be drawn before administration of vitamin supplementation
- $^{\mathrm{m}}$  PK samples will be drawn pre-dose, and approximately 2.5 hours after the morning dose
- <sup>n</sup> If needed, study drug may be supplied via direct-to-patient shipments in between site visits, see Section 6.4 of the protocol (amendment 4).
- O Subjects will self-administer (or will be administered) the first dose of study drug in the clinic on Visit 1/Day 0 after breakfast under the supervision of the Investigator or trained site staff.
- P See Appendix 10 of the protocol (amendment 4) for management of study procedures during pandemic.



### 4. Statistical Analysis and Reporting

#### 4.1. Introduction

Data processing, tabulation of descriptive statistics, calculation of inferential statistics, and graphical representations will be performed primarily using SAS (release 9.4 or higher). If the use of other software is warranted, the final statistical methodology report will detail what software was used for what purposes.

Continuous (quantitative) variable summaries will include the number of participants with non-missing values (n), mean, 2-sided 95% CI for the mean, standard deviation (SD) and/or standard error (SE) if appropriate, median, minimum, and maximum.

Categorical (qualitative) variable summaries will include the frequency and percentage of participants who are in the particular category for each possible value. In general, the denominator for the percentage calculation will be based upon the total number of participants in the analysis population (and cohort where applicable) with available data for each treatment group, unless otherwise specified.

The minimum and maximum will be reported with the same degree of precision (i.e., the same number of decimal places) as the observed data. Measures of location (mean and median) will be reported to 1 degree of precision more than the observed data and measures of spread (i.e., SD or SE) will be reported to 2 degrees of precision more than the observed data. Confidence intervals (CIs) for the mean are reported to the same degree of precision as the mean.

The minimum and maximum values for derived and select observed values will be reported as follows, with measures of location and spread following the above rules. Derived values for corrected sodium (mEq/L), calculated osmolarity (mOsm/kg), osmolar gap (mOsm/kg), anion gap (mEq/L), MELD and PELD scores will be presented as integers. Derived values for PedsQL summary and total scale scores will be presented to 1 decimal place. Serum bile acid levels (total and sub-species), and derived values of height, weight, and BMI z-scores, EDQ and ItchRO average scores, FIB-4, APRI, retinol:RBP molar ratio (mol/mol), and ratio of α-tocopherol to the sum of cholesterol and triglycerides (mg/g), will be reported to 2 decimal places.

Percentages will be presented to 1 decimal place, unless otherwise specified. Where the number of participants in a particular category is zero, a percentage (i.e., 0.0%) will not be displayed.

Unless otherwise indicated, all testing of statistical significance will be 2-sided, and a difference resulting in a p-value of  $\leq 0.05$  will be considered statistically significant. Corresponding 95% confidence intervals (CIs) will be presented for statistical tests.

A p-value of  $\leq 0.10$  but > 0.05 will be considered evidence of a trend.





To control for the overall type I error rate, hierarchical testing based on a fixed sequence procedure will be used. If statistical significance is declared for the primary efficacy analysis, formal hypothesis testing will be done for the secondary efficacy endpoints in the pre-specified sequence until a non-significant result is reached. All other p-values from secondary endpoints, after a non-significant p-value is reached, will be considered nominal and will be interpreted with appropriate caution when considering the extent to which results from secondary endpoints provide support for evidence of efficacy.

### 4.2. Interim Analysis and Data Monitoring

No interim analyses are planned.

A data monitoring committee (DMC) will be involved in the management of this study. DMC meetings will be held periodically for the duration of the study. The purpose of the DMC is to review the progress of the study, with regard to safety and make recommendations to the Sponsor to stop or modify the study if safety concerns are identified. In addition to scheduled meetings, the DMC will convene for ad hoc meetings in case of any safety concerns arising during the conduct of the study.

Further details regarding the DMC can be found in the DMC charter, which will be available prior to the enrollment of the first participant. There is no study stop planned based on the efficacy results during the study and no alpha spending will occur prior to the completion of the study.

### 5. Analysis Populations

The following analysis populations are planned for this study:

- **Safety Population:** The Safety Population will consist of all participants who receive at least 1 dose of study drug.
- **Intent-To-Treat (ITT) Population:** The ITT Population will consist of all randomized participants.
- **Per Protocol (PP) Population**: The PP Population will consist of all participants in the ITT Population who receive at least 1 dose of study drug and do not have any important protocol violations or deviations that have a potential impact on the efficacy analysis. Important protocol violations/deviations will be identified prior to database lock.

Membership in the analysis populations will be determined prior to database lock.





The primary efficacy endpoint and the key secondary efficacy endpoint (i.e., change from baseline in sBA) will be analyzed for the ITT and PP analysis populations. The other secondary and exploratory efficacy endpoints will be analyzed in the ITT population.

The number of participants excluded from each analysis will be presented.

Safety, tolerability, and PK analyses will be conducted in the Safety Population.

Because PFIC is a rare disease, siblings are allowed to enroll in this study. Each sibling will be considered for each analysis population described above. A sensitivity analysis on the primary efficacy endpoint and the key secondary efficacy endpoint will include only 1 sibling in the ITT analysis population. The choice of sibling will be made at random. The method of choosing a sibling is described in Section 6.1.9.

### 5.1. Subject Grouping

The following subject cohorts will be used for the analysis of the various endpoints in this study. Subject cohorts are identified according to the centrally adjudicated PFIC type which are recorded on the Genotype Adjudication file (see Section 6.1.9).

- **Primary cohort**: All non-truncated PFIC2 (nt-PFIC2) participants.
- **PFIC cohort**: PFIC1, nt-PFIC2, PFIC3, PFIC4, PFIC5 and PFIC6 participants (i.e., all genotypes <u>except</u> for truncating PFIC2 [t-PFIC2] participants, and participants with heterozygosis, low or fluctuating sBAs, a history of surgery, or where there is no established variant linked to PFIC disease)
- Full cohort: All participants enrolled.

Each of the above-defined cohorts, with the exception of the Full cohort, will exclude any participants with previous documented surgery to address PFIC at baseline.

### 6. General Issues for Statistical Analysis

### 6.1. Statistical Definitions and Algorithms

#### 6.1.1. Baseline

In general, baseline values are defined as data measured or collected at the baseline visit, Visit 1 (Day 0), before the first dose of study drug is administered. If data is not measured or collected at the baseline visit, then the last non-missing measurement before receiving the first dose of study drug is used as the baseline value.





Baseline and all post-baseline sBA samples are assayed at Frontage Laboratories, while screening sBA samples are assayed at ACM Global Laboratories. Only pre-dose samples assayed at Frontage Laboratories will be used as a baseline sample.

Baseline ItchRO and EDQ average morning, evening, and highest scores (observer and patient) are constructed as the average of 4 weekly (7-day) average scores in the period consisting of the 28 days immediately before the date of first dose of study drug. The numerator and denominators used in the derivation of weekly average and time period scores are based on the number of non-missing daily and weekly scores, respectively.

For liver-biochemistry laboratory parameters (i.e., ALT, AST, ALP, total bilirubin, direct bilirubin, GGT, and albumin) baseline is defined as the average of data collected between Screening and Visit 1 (Day 0), or the last non-missing measurement before receiving the first dose of study drug if only one value is available. Pre-dose measurements obtained from a local laboratory will only be used if no other data are available. For the derived non-invasive fibrosis markers of APRI, FIB-4, PELD, and MELD, the same (derived/average) liver-biochemistry baseline value will be used.

### **6.1.2.** Adjustments for Covariates

Efficacy variables that are continuous measures assessed over time will be analyzed using a mixed-effects model for repeated measures (MMRM) with change from baseline as the dependent variable and fixed, categorical effects of treatment group, analysis visit, and treatment group-by-visit interaction as well as the continuous, fixed covariates of baseline and baseline-by-visit interaction.

For the PFIC cohort (as defined in Section 5.1), PFIC type will also be used as a covariate in the MMRM analysis. For this analysis, due to the small sample sizes, PFIC4, PFIC5, and PFIC6 will be grouped together. Within the PFIC cohort, 4 levels of PFIC types are included in the covariate: nt-PFIC2, PFIC1, PFIC3, and other (PFIC4, PFIC5, and PFIC6 group).

No other covariates will be included in the analyses of the efficacy endpoints.

### 6.1.3. Multiple Comparisons

The type I error rate of  $\alpha = 0.05$  will be maintained for the study by using sequential (hierarchical) testing for primary and secondary efficacy endpoints.

The testing will be done in the following order, noting the primary and PFIC cohorts are defined in Section 5.1:

1. Primary: Mean change in the average morning ItchRO(Obs) severity score between baseline and Week 15 through Week 26 in the primary cohort



- 2. Key Secondary: Mean change in total sBA level between baseline and average of Weeks 18, 22, and 26 in the primary cohort
- 3. Secondary: Mean change in the average morning ItchRO(Obs) severity score between baseline and Week 15 through Week 26 in the PFIC cohort
- 4. Secondary: Mean change in total sBA level between baseline and average of Weeks 18, 22, and 26 in the PFIC cohort
- 5. Secondary: Proportion of ItchRO(Obs) responders from Week 15 to Week 26 (reference Section 6.1.8) in the primary cohort
- 6. Secondary: Proportion of sBA responders from Week 18 to Week 26 (reference Section 6.1.8) in the primary cohort
- 7. Secondary: Proportion of ItchRO(Obs) responders from Week 15 to Week 26 in the PFIC cohort
- 8. Secondary: Proportion of sBA responders from Week 18 to Week 26 in the PFIC cohort

Because the testing is sequential, the type I error rate of  $\alpha = 0.05$  is maintained. Failure at any stage in the sequence implies no type I error control for the additional subsequent tests. All p-values for each comparison without adjustments will be provided in the summary tables for informational purposes.

### 6.1.4. Handling of Dropouts or Missing Data

While all possible efforts will be made to ensure that participants stay in the study and all data is collected as scheduled, the occurrence of missing data cannot be completely eliminated.

The primary analysis population for all efficacy analyses will be the ITT Population. For the analysis of primary efficacy endpoint and the key secondary efficacy endpoint, based on the ITT Population over the primary and PFIC cohorts (separately), several methods will be used to handle missing data for average morning ItchRO(Obs) severity and total sBA, including:

- MMRM
- multiple imputation (MI) using standard MAR approach
- MI using tipping point approach

The MMRM method will be used for the primary analysis on all continuous, repeated efficacy measures. Sensitivity analyses using the 2 MI methods will be performed on the primary efficacy endpoint and the key secondary efficacy endpoint to assess the robustness of alternate imputation assumptions.





The above procedures are described in the below sub-sections, along with the handling of missing individual ItchRO and EDQ scores, PedsQL scale scores, and adverse event severity and relationship to study drug.

### 6.1.4.1. MMRM Analysis Method

Efficacy variables that are continuous measures assessed over time will be analyzed using a MMRM model as the primary analysis method, with change from baseline as the dependent variable and fixed, categorical effects of treatment group, visit, and treatment group-by-visit interaction as well as the continuous, fixed covariates of baseline and baseline-by-visit interaction. For PFIC cohort analyses, PFIC type (i.e., PFIC1, nt-PFIC2, PFIC3, and the combination of PFIC4, PFIC5, and PFIC6) will also be included in the MMRM model as a covariate.

The MMRM method has been demonstrated extensively as an appropriate choice for the primary analysis in longitudinal confirmatory clinical trials with continuous endpoints (Mallinckrodt et al, 2008). This analysis method, which is from a broader class of direct-likelihood analyses methods, makes use of fully and partially observed data sequences from individual participants by estimating the covariance between data from different time points (Molenberghs et al, 2007). Further, it is often useful to implement MMRM using an unstructured approach to modeling both the treatment-by-time means and the variances and covariances, leading to what is essentially a multivariate normal model wherein treatment group means at the primary time point are adjusted to reflect both the actual observed data and the projected outcomes from the participants with missing data (Cnaan et al, 1997, Molenberghs et al, 2004, Molenberghs et al, 2007).

As a direct likelihood method, the MMRM method is a preferred approach for handling missing data in such designs and will be used as the primary analysis method for all efficacy and safety endpoints where assessments are made over time. MMRM is a full multivariate model in nature, which avoids potential bias as a predetermined model and operates in a more general missing at random (MAR) framework (Mallinckrodt et al, 2001). Data are considered MAR if, conditional upon the independent variables in the analytic model, the missingness depends on the observed outcomes of the variable being analyzed but does not depend on the unobserved outcomes of the variable being analyzed. This assumption implies that the behavior of the post dropout observations can be predicted from the observed variables, and therefore that treatment effect can be estimated without bias using the observed data (EMA, 2010). For studies of missing data in a controlled clinical trial setting, MAR is usually considered as a plausible underlying missing mechanism (Molenberghs et al, 2007; Siddiqui et al, 2009, Mallinckrodt et al, 2008, Mallinckrodt et al, 2013). The assumption of MAR is often reasonable because, particularly in longitudinal studies wherein the evolution of treatment effects is assessed by design over time, the observed data and the models used to analyze them can explain much of the missingness (Little et al, 1987, Verbeke et al, 2000). This point may be especially relevant in well-controlled studies, in which extensive efforts are made to observe all outcomes and factors that influence



proc mixed data = example;



them while participants are following protocol-defined procedures. Thus, longitudinal clinical trials by their very design aim to reduce the amount of missing not at random (MNAR) data (missingness explained by unobserved responses), thereby increasing the plausibility of MAR (Mallinckrodt et al, 2008).

The following SAS pseudocode will be used for the MMRM models:

```
class <subjectid> <visit> <treatment>;
   model chg = <baseline score> <treatment> <visit> <treatment>*<visit> <baseline score>*<visit> /
              *** PFIC type is included in the model for analyses of the PFIC cohort ***;
   repeated <visit> / subject = <subjectid>(<treatment>) type = un;
   Ismeans <treatment>*<visit> / cl pdiff;
lsmestimate <treatment>*<visit> 'Weeks 15-18 MRX LS Mean=0' 0 0 1 0 0 0 0 0 0 0 0 divisor=1 / cl;
lsmestimate <treatment>*<visit> 'Weeks 15-18 Placebo LS Mean=0' 0 0 0 0 0 0 0 0 0 0 0 divisor=1 / cl;
lsmestimate <treatment>*<visit> 'Weeks 15-18 MRX LS Mean = Placebo LS Mean' 0 0 1 0 0 0 0 0 -1 0 0 0
divisor=1 / cl;
lsmestimate <treatment>*<visit> 'Weeks 19-22 MRX LS Mean=0' 00010000000 divisor=1 / cl;
lsmestimate <treatment>*<visit> 'Weeks 19-22 Placebo LS Mean=0' 0 0 0 0 0 0 0 0 0 0 0 0 divisor=1 / cl;
lsmestimate <treatment>*<visit> 'Weeks 19-22 MRX LS Mean = Placebo LS Mean' 0 0 0 1 0 0 0 0 -1 0 0
divisor=1 / cl;
lsmestimate <treatment>*<visit> 'Weeks 23-26 MRX LS Mean=0' 0 0 0 0 1 0 0 0 0 0 0 divisor=1 / cl;
```

lsmestimate <treatment>\*<visit> 'Weeks 23-26 Placebo LS Mean=0' 0 0 0 0 0 0 0 0 0 0 1 0 divisor=1 / cl; Ismestimate <treatment>\*<visit> 'Weeks 23-26 MRX LS Mean = Placebo LS Mean' 0 0 0 0 1 0 0 0 0 -1 0 divisor=1 / cl;

lsmestimate <treatment>\*<visit> 'Weeks 15-26 MRX LS Mean=0' 0 0 1 1 1 0 0 0 0 0 0 0 divisor=3 / cl; lsmestimate <treatment>\*<visit> 'Weeks 15-26 Placebo LS Mean=0' 0 0 0 0 0 0 0 1 1 1 0 divisor=3 / cl; lsmestimate <treatment>\*<visit> 'Weeks 15-26 MRX LS Mean = Placebo LS Mean' 0 0 1 1 1 0 0 0 -1 -1 -1 0 divisor=3 / cl: run;

#### Multiple Imputation Methods 6.1.4.2.

Although the assumption of MAR, as used for the primary efficacy analysis method, is often reasonable in clinical trials, the possibility of MNAR data cannot be ruled out. Therefore, analysis valid under MNAR will also be performed. Both MNAR- and MAR-based analyses using MI methods will be the basis upon which sensitivity of the analysis to missing data are assessed.

Any participant who withdraws or is discontinued from the study or who misses a scheduled visit or assessment up through Week 26 will have their primary and key secondary efficacy missing data analyzed as imputed using MI techniques. This analysis will be presented as a sensitivity analysis.





Multiple imputation is a simulation-based approach where missing values are replaced using an appropriate stochastic model given the observed data and covariates, creating multiple completed data sets. These completed datasets are then analyzed using standard analysis methods (MMRM for this study), and the different parameter estimates across the datasets are then combined to produce unique point estimates, standard errors, and confidence intervals taking into account the uncertainty of the imputation process.

In most randomized clinical trials that collect data over time, the great majority of missing data follow a monotone pattern. That is, once a participant has missing data for some visit, data will be missing for all subsequent visits. Typically, there is also a small amount of non-monotone missing data (i.e., some participants have missing values for intermediate visits, but have non-missing data at subsequent visits).

The following 2 MI analysis models, one based on the standard MAR approach and the other based on the MNAR approach, will be used to examine robustness of the primary analysis results.

### **Standard MAR Imputation**

The MAR imputation model will impute missing values using a regression-based multiple imputation model (Little et al, 1996). For participants with complete data up to a particular timepoint (e.g., time period average score for the primary endpoint and analysis visit for the key secondary endpoint), a multiple regression model will be fit that includes the outcome at that time point as the dependent variable and observed data (e.g., outcomes at previous time points, treatment, and baseline) as independent variables. Separate models will be similarly constructed for each time point. Using these regression models, a missing value for a participant at a particular time point will be imputed as a draw from the predictive distribution given the outcomes at previous time points (some possibly imputed), treatment group, etc. This process will be repeated a given number of times (as specified below), resulting in the same number of complete analysis data sets. The MMRM analyses will be performed separately for each of the completed analysis data sets, and the results will be combined into one multiple imputation inference (Little et al, 1996, Schafer, 1997). This strategy is appropriate for data sets that have a monotone missing data pattern. If the data set does not precisely have this pattern, a monotone data augmentation method, as described below in Step 1, will be used to impute the small amount of missing data that is required to make the missing data pattern monotone before applying the MI algorithm described above.

Multiple imputation based on a standard MAR imputation approach will be performed in SAS using a general three-step approach:

Step 1: If the data has a non-monotone pattern of missingness, then a monotone data augmentation method using Markov-Chain Monte-Carlo (MCMC) will be used to impute data that is missing and required to make the missing data pattern monotone. Twenty datasets with a





monotonic missing pattern will be generated. This method will use a non-informative Jeffreys prior to derive the posterior mode from the expectation-maximization (EM) algorithm as the starting values for the MCMC method. Intermittent missing values will be imputed using the MCMC method assuming a multivariate normal distribution over all variables included in the imputation model (i.e., treatment group, baseline, and each post-baseline visit). The MCMC statement of the MI procedure in SAS (PROC MI) will specify the CHAIN=MULTIPLE option, so that the procedure uses multiple chains and completes the default 200 burn-in iterations before each imputation, and the IMPUTE=MONOTONE option to create the 20 partially imputed datasets with a monotone missing pattern. The seed of the pseudorandom number generator used to randomly generate imputations for the missing values in Step 1 is 3590145.

Assumptions underlying the partial imputation step are such that participants with missing data follow the same model as other participants in their respective treatment arm that have complete data.

If the raw data has a monotone pattern of missingness, then the same procedures described above can be followed to create 20 identical datasets that will be used as an input dataset for the next step.

Pseudocode for imputation of primary efficacy missing data is provided below:

Step 2: Using a standard MAR-based MI approach, the remaining missing data will be imputed using a method for monotone missingness. The dataset that contains the multiple (20) partially imputed datasets is first sorted by imputation number and treatment group. The MI procedure used to complete the imputation will use a BY imputation number statement and request one imputed dataset within each BY group. The variables in the imputation model include treatment group, baseline, and each post-baseline visit. The final 20 fully imputed datasets will be generated using a regression-based multiple imputation model (PROC MI statement MONOTONE REGRESSION). For participants with complete data up to a particular visit, a multiple regression model will be fit that includes the outcome at that visit as the dependent variable and outcomes at previous visits and treatment group as independent variables. Using these regression models, a missing value for a participant at a particular time point will be imputed as a draw from the predictive distribution given the outcomes at previous time points (some possibly imputed) and treatment group. The seed number of 9482038 will be used for the imputation procedure described in Step 2.





For both Steps 1 and 2, minimum and maximum values for average ItchRO severity scores (i.e., 0 and 4) will be specified in the MI procedure to avoid imputed values outside the possible range of values. When an intended imputed value is less than the minimum or greater than the maximum value specified, the MI procedure in SAS will redraw another value for imputation.

Pseudocode for this step is below:

```
proc sort data= example 1;
       by <imputationnumber> <treatment>;
run;
proc mi data= example_1 nimpute=1 seed=9482038 minimum = 0 maximum = 4 out= example_2;
       by <imputationnumber>;
       monotone regression;
       var <treatment> <baseline score> <week 1-6>...... <week 23-26>;
run;
```

Step 3: MMRM analyses will be performed separately for each of the 20 complete analysis datasets, and the results will be combined into one multiple imputation inference (estimated treatment effect, standard error, p-value and associated 95% confidence interval) using the SAS MIANALYZE procedure. The treatment difference will be tested at the 2-sided 0.05 level and corresponding 95% CIs will be calculated. In the case that there is no missing data for a particular visit, p-values and 95% confidence intervals will come from the MMRM analysis on the observed data.

SAS pseudocode for the MMRM analysis is as follows:

```
ods output | Ismestimates = Ism diff;
proc mixed data = example 3;
        by <imputationnumber>;
        class <subjectid> <treatment> <visit>;
        model chg = <baseline score> <treatment> <visit> <treatment>*<visit> <baseline score>*<visit>
/ddfm = kr; *** PFIC type is included in the model for analyses of the PFIC cohort ***;
<visit> / subject = <subjectid>(<treatment>) type = un;
   lsmeans <treatment>*<visit> / cl pdiff;
lsmestimate <treatment>*<visit> 'Weeks 15-18 MRX LS Mean=0' 0 0 1 0 0 0 0 0 0 0 0 0 divisor=1 / cl;
lsmestimate <treatment>*<visit> 'Weeks 15-18 Placebo LS Mean=0' 0 0 0 0 0 0 0 0 1 0 0 0 divisor=1 /
cl;
Ismestimate <treatment>*<visit> 'Weeks 15-18 MRX LS Mean = Placebo LS Mean' 0 0 1 0 0 0 0 0 -1 0 0 0
divisor=1 / cl;
lsmestimate <treatment>*<visit> 'Weeks 19-22 MRX LS Mean=0' 00010000000 divisor=1 / cl;
lsmestimate <treatment>*<visit> 'Weeks 19-22 Placebo LS Mean=0' 0 0 0 0 0 0 0 0 0 0 0 0 divisor=1 / cl;
```




lsmestimate <treatment>\*<visit> 'Weeks 19-22 MRX LS Mean = Placebo LS Mean' 0 0 0 1 0 0 0 0 0 -1 0 0 divisor=1 / cl;

run;

```
proc mianalyze data=diff;
  by <visit>;
  modeleffects estimate;
STDERR stderr;
  ods output parameterestimates=dif_2;
run;

proc mianalyze data=lsm;
  by <visit> <treatment>;
  modeleffects estimate;
  stderr stderr;
  ods output parameterestimates=lsmn_2;
run;
```

Pseudocode for imputation of key secondary efficacy missing data is provided below. There is a potential need to add option MAXITER=nnn to the MI procedure if the analysis fails to converge with 200 iterations.

```
Step 1:
```

XX will be determined based on the proportion of missing data across visits. The minimum and maximum values for total sBA level will be specified as the minimum and maximum values of the calculated results.





```
Step 2:
proc sort data= example_1;
       by <imputationnumber> <treatment>;
run;
proc mi data= example 1 nimpute=1 seed=9482038 minimum = yy maximum = yy out= example 2;
       by <imputationnumber>;
       monotone regression;
       var <treatment> <baseline> <week 2>..... <week 26>;
run;
Step 3:
ods output Ismestimates= Ism diff;
proc mixed data = example 3;
       by <imputationnumber>;
       class <subjectid> <treatment> <visit> ;
       model chg = <baseline> <treatment> <visit> <treatment>*<visit> <baseline> *<visit> /ddfm = kr;
       *** PFIC type is included in the model for analyses of the PFIC cohort ***;
       repeated <visit> / subject = <subjectid>(<treatment>) type = un;
       lsmeans <treatment>*<visit> / cl pdiff;
lsmestimate <treatment>*<visit> 'Week 18 MRX LS Mean=0' 0 0 1 0 0 0 0 0 0 0 0 0 0 0 divisor=1 / cl;
lsmestimate <treatment>*<visit> 'Week 18 Placebo LS Mean=0' 0 0 0 0 0 0 0 0 0 0 0 0 0 divisor=1 / cl;
lsmestimate <treatment>*<visit> 'Week 18 MRX LS Mean = Placebo LS Mean' 0 0 1 0 0 0 0 0 0 -1 0 0 0 0
divisor=1 / cl;
lsmestimate <treatment>*<visit> 'Week 22 MRX LS Mean=0' 0000100000000 divisor=1 / cl;
lsmestimate <treatment>*<visit> 'Week 22 Placebo LS Mean=0' 0 0 0 0 0 0 0 0 0 0 0 1 0 0 divisor=1 / cl;
Ismestimate <treatment>*<visit> 'Week 22 MRX LS Mean = Placebo LS Mean' 0 0 0 0 1 0 0 0 0 0 -1 0 0
divisor=1 / cl;
lsmestimate <treatment>*<visit> 'Week 26 MRX LS Mean=0' 000001000000 divisor=1 / cl;
lsmestimate <treatment>*<visit> 'Week 26 Placebo LS Mean=0' 0 0 0 0 0 0 0 0 0 0 0 1 0 divisor=1 / cl;
lsmestimate <treatment>*<visit> 'Week 26 MRX LS Mean = Placebo LS Mean' 0 0 0 0 0 1 0 0 0 0 0 -1 0
divisor=1 / cl:
lsmestimate <treatment>*<visit> 'Weeks 18-26 MRX LS Mean=0' 00101100000000 divisor=3 /
| Ismestimate <treatment>*<visit> 'Weeks 18-26 Placebo LS Mean=0' 0 0 0 0 0 0 0 0 1 0 1 1 0 divisor=3
cl;
lsmestimate <treatment>*<visit> 'Weeks 18-26 MRX LS Mean = Placebo LS Mean' 0 0 1 0 1 1 0 0 0 -1 0 -1
-10 divisor=3 / cl;
run;
```





```
proc mianalyze data=diff;
  by <visit>;
  modeleffects estimate;
STDERR stderr;
  ods output parameterestimates=dif_2;
run;

proc mianalyze data=lsm;
  by <visit> <treatment>;
  modeleffects estimate;
  stderr stderr;
  ods output parameterestimates=lsmn_2;
run;
```

# **Tipping Point Analysis**

As a sensitivity analysis to the standard MAR imputation approach, a tipping point analysis will be performed in order to determine the inflection point at which the inference under the MNAR assumption changes substantially. This will be used to check the robustness of the imputation.

The sensitivity analysis will be performed by using a specified sequence of shift parameters, which will adjust the imputed values for observations in each treatment group. The range of shift parameters to be included in this analysis are -2 to 2 by 0.2. Thus, the value at which the results of the analysis are shifted from significant (i.e.,  $\alpha \le 0.05$ ) to non-significant (i.e.,  $\alpha > 0.05$ ) will be determined.

A heatmap figure will be generated to display p-values corresponding to all combinations of shifts from the imputed data.

The seed number of 2740211 will be used for the imputation procedure described in Step 2.

Steps 1 and 3 of the analysis will be the same as for the multiple imputation analysis as described in the Standard MAR Imputation above. However, Step 2 of the analysis is the step that the shift parameters will be applied. Pseudocode for Step 2 is as follows:

```
proc mi data=example_1 seed=2740211 nimpute =1 OUT= example_2;
    class <treatment>;
    by <imputationnumber>;
    monotone regression;
    var <baseline score> <week 1-6>...... <week 23-26>;
    mnar adjust ( <week 1-6>/ shift=YY adjustobs=(treatment ='active') );
    mnar adjust ( <week 1-6>/ shift =YY adjustobs =( treatment ='placebo') );
    mnar adjust ( <week 7-10>/ shift =YY adjustobs =( treatment ='active'));
```





```
mnar adjust ( <week 7-10>/ shift =YY adjustobs =( treatment ='placebo') );
mnar adjust ( <week 11-14>/ shift =YY adjustobs =( treatment ='active') );
mnar adjust ( <week 11-14>/ shift =YY adjustobs =( treatment ='placebo') );
mnar adjust ( <week 15-18>/ shift =YY adjustobs =( treatment ='active') );
mnar adjust ( <week 15-18>/ shift =YY adjustobs =( treatment ='placebo') );
mnar adjust ( <week 19-22>/ shift =YY adjustobs =( treatment ='active') );
mnar adjust ( <week 19-22>/ shift =YY adjustobs =( treatment ='placebo') );
mnar adjust ( <week 23-26>/ shift =YY adjustobs =( treatment ='placebo') );
run;
```

YY will encompass the range of shift parameters as pre-specified above.

proc mi data=example\_1 seed=2740211 nimpute =1 OUT= example\_2;

For the secondary endpoint the planned range of shift parameters to be included in this analysis are -100 to 100 by 1.

Pseudocode for Step 2 for imputation of key secondary efficacy missing data is as follows:

```
class <treatment>;
        by <imputationnumber>;
        monotone regression;
        var <baseline> <week 2>...... <week 26>;
        mnar adjust ( <week 2>/ shift=YY adjustobs=(treatment ='active') );
        mnar adjust ( <week 2>/ shift =YY adjustobs =( treatment ='placebo') );
        mnar adjust ( <week 6>/ shift =YY adjustobs =( treatment ='active'));
        mnar adjust ( <week 6>/ shift =YY adjustobs =( treatment ='placebo') );
        mnar adjust ( <week 10>/ shift =YY adjustobs =( treatment ='active') );
        mnar adjust ( <week 10>/ shift =YY adjustobs =( treatment ='placebo') );
        mnar adjust ( <week 14>/ shift = YY adjustobs =( treatment ='active') );
        mnar adjust ( <week 14>/ shift =YY adjustobs =( treatment ='placebo') );
        mnar adjust ( <week 18>/ shift =YY adjustobs =( treatment ='active') );
        mnar adjust ( <week 18>/ shift =YY adjustobs =( treatment ='placebo') );
        mnar adjust ( <week 22>/ shift =YY adjustobs =( treatment ='active') );
        mnar adjust ( <week 22>/ shift =YY adjustobs =( treatment ='placebo') );
        mnar adjust ( <week 26>/ shift =YY adjustobs =( treatment ='active') );
        mnar adjust ( <week 26>/ shift =YY adjustobs =( treatment ='placebo') );
run;
```





## 6.1.4.3. Missing ItchRO/EDQ/PedsQL Scores

In deriving the highest daily ItchRO/EDQ severity/frequency score, if either the morning or evening reports are not completed, the available score is used as the highest daily score. If both morning and evening reports are not completed, the highest daily score for that day is treated as missing data.

For weekly (7-day) morning/evening/highest ItchRO(Obs)/ItchRO(Pt)/EDQ(Obs)/EDQ(Pt) severity/frequency scores, if >50% (i.e., >3 of 7) of the daily scores are missing, the average score for that weekly time period will be treated as missing.

For 4- and 6-week time period ItchRO/EDQ scores (i.e., baseline, post-baseline to Week 6, Week 7 to 10, Week 11 to 14, Week 15 to 18, Week 19 to 22, and Week 23 to 26), if >50% of the weekly scores are missing, the respective time period score will be treated as missing. Thus, to derive a 4-week time period score, 2 or more of the respective weekly scores must be non-missing; for a 6-week time period score, 3 or more weekly scores must be non-missing.

For Pediatric Quality of Life Inventory (PedsQL) scale scores, if >50% of the items in the scale are missing, the scale score is not computed.

# 6.1.4.4. Missing Responder Definition Data

For the sBA responder endpoint, a participant is defined as a non-responder if the baseline value is missing OR sBA values are missing at all of the 3 time points (i.e., Weeks 18, 22, and 26).

For the ItchRO responder endpoint, a participant is defined as a non-responder from Week 15 to 26 if the 4-week average baseline score is missing OR all of the three 4-week average (post-baseline) scores (i.e., Weeks 15-18, 19-22, and 23-26) are missing.

For the number of days the morning ItchRO(Obs) severity score is  $\leq 1$  over the last 84 days (i.e., study day 99 through 182, inclusive, relative to the day of 1<sup>st</sup> dose of study drug), days with missing data would <u>not</u> be considered to have met the " $\leq 1$ " criteria for that day. In computing the total number of days that the score is  $\leq 1$  within the specified time period (for each participant), missing data will be treated as having a score of >1.

For the number and proportion of participants achieving morning ItchRO(Obs) severity scores  $\leq 1$  for more than 50% of the time within pre-specified time periods, days with missing data would <u>not</u> be considered to have met the " $\leq 1$ " criteria for that day. In computing the % of time the score is  $\leq 1$  within each time period for each participant, the denominator of the proportion would include all days within the specified time period (i.e., days with missing and non-missing data), while the numerator only includes those days that the score is 0 or 1.



For the proportion of participants with improvement from baseline in EDQ sleep scores, a participant is defined as having no improvement (i.e., non-responder) for an analysis visit if the 4-week average baseline score is missing OR the 4-week (or 6-week for the first time period) average sleep score at the analysis visit is missing.

For the proportion of EDQ sleep scores ≤2, missing scores are treated as a non-responder (i.e., >2).

# 6.1.4.5. Missing Adverse Event Severity/Relationship

For analysis purposes, the following rules will be applied for missing AE severity or relationship to study drug. An AE that does not have a recorded relationship to study drug value will be considered as "Related" to study drug. If the severity of an AE is missing, the severity will be reported as "Missing".

# 6.1.5. Analysis Visit Windows

Analyses of all visit-based efficacy and safety variables will be performed using the analysis visit windows defined by study day relative to the first dose of study drug as outlined below in Table 2. Scheduled visits will be selected over unscheduled visits. The below table addresses scheduled post-baseline in-clinic visits; baseline assessments are described in Section 6.1.1.

**Table 2: Analysis Visit Windows** 

| Analysis<br>Visit | Analysis<br>Visit Name | Target Day<br>of Planned<br>Visit | Assessment Window (Study Days1) |
|---|---|---|---|
| 2 | Week 2 | 14 | $1^2 - 20$ |
| 4 | Week 4 | 28 | 21 - 34 |
| 6 | Week 6 | 42 | 35 - 55 |
| 10 | Week 10 | 70 | 56 - 83 |
| 14 | Week 14 | 98 | 84 - 111 |
| 18 | Week 18 | 126 | 112 - 139 |
| 22 | Week 22 | 154 | 140 - 167 |
| 26 | Week 26 | 182 | 168 - x |

<sup>&</sup>lt;sup>1</sup> Study day relative to the date of first dose of study drug.

For those participants who discontinue early from the study, Table 2 will also be used to assign the appropriate analysis visit.

<sup>&</sup>lt;sup>2</sup>Only data collected post-dose on Day 1 will be considered.

x = last dose date plus 7 days





The study day will be calculated for each scheduled or ET post-baseline visit and compared to the assessment window presented in Table 2 to define the visit window used for analyses. The analysis visit windows only apply to those visits that are applicable to the specific assessment. For example, if the scheduled or ET visit falls at Week 4 but a specific assessment (e.g., sBA sample) was not scheduled at that visit (see Table 1, Schedule of Assessments), then that assessment will not be used for analyses.

If more than 1 assessment occurs within a single visit window, then the analysis will use the assessment closest to the target day. If 2 assessments within the same visit window are equidistant from the target day, then the analysis will use the later assessment.

Efficacy assessments performed >7 days after the last dose of study drug will not be included in any efficacy analyses.

## **6.1.6.** Investigative Sites

An investigative site is defined as a single principal investigator (including sub-investigators) who enroll participants for the study. If an investigator has multiple practice locations, these locations are considered a single investigative site.

There is the potential that a participant could be transferred to a principal investigator that did not enroll the participant. Unless otherwise specified, the investigative site of the enrolling investigator will be used for the unique participant ID.

The primary presentations and analyses will be based on data pooled across investigative sites.

#### 6.1.7. Treatment Period Definitions

- "Dose Escalation Period" is defined for analysis purposes as the period of time between the first dose of study drug and the end of study Week 6 (i.e., through the Week 6 visit date).
- "Stable Dosing Period" is defined for analysis purposes as the period of time between the beginning of Week 7 (i.e., Week 6 visit date plus 1 day) and the EOT visit (inclusive).

#### 6.1.8. Derived Variables

Select derived variables will be rounded for presentation purposes (see Section 4.1).

#### • Age (years) at baseline

The reported age in years at baseline will be used.



#### Age (months) at baseline

The reported age in years and months at baseline will be used:

Age (months) at baseline = (12 x Reported age in years at baseline) + Reported number of months at baseline

#### • Date of Birth

```
Date of Birth = Baseline Visit Date - [ 365.25 x ( Age in yrs + (months/12) ) ]
```

Age in years and months at baseline, as reported on the CRF, is used. If only age in years (at baseline) is reported, then 6 months will be used.

If the derived date of birth is later than the PFIC diagnosis date, the earliest complete medical history event start date, or the earliest complete reported prior/concomitant treatment start date, will be used to derive the date of birth by selecting the earliest of these 3 dates.

- **Age Group at baseline**: 1 if age (full years) at baseline is 1 to < 6 years 2 if age (full years) at baseline is 6 to <13 years 3 if age (full years) at baseline is 13 to 18 years
- UDCA usage at baseline: A subject reporting the use of UDCA, based on ATC Class Level 5 (chemical substance), with a start date on or prior to the first dose of study drug and either be ongoing or have a stop date on or after the first dose of study drug would be considered as using UDCA at baseline.
- **Rifampicin usage at baseline**: A subject reporting the use of Rifampicin, based on ATC Class Level 5 (chemical substance), with a start date on or prior to the first dose of study drug and either be ongoing or have a stop date on or after the first dose of study drug would be considered as using Rifampicin at baseline.
- Time since original diagnosis of PFIC (months) = (date of first dose date of original diagnosis of PFIC) / 30.4375
- Change from baseline = post-baseline value at time point value at baseline
   For average ItchRO and EDQ scores, "value" is the average score as defined below.
- % Change from baseline = 100 x change from baseline / value at baseline



## **Highest daily ItchRO and EDQ scores** = maximum of morning and evening scores

If either the morning or evening reports are not completed, the available score is used as the highest daily score. If both morning and evening reports are not completed, the highest daily score for that day is treated as missing data.

### **Baseline ItchRO and EDQ scores:**

Baseline morning, evening, and highest ItchRO and EDQ scores used for analysis purposes are calculated using the daily scores from the 28 days (4 weeks) immediately before the date of first dose. Pre-dose weekly scores are first calculated for each of the 4-week, 7-day periods. The "first" 7-day period (immediately before the first dose date) is considered 'Week -1', whereas the "last" 7-day period is considered as 'Week -4'. For each subject and ItchRO/EDQ efficacy variable, a baseline score is derived as the average of the 4 pre-dose weekly average scores.

The handling of missing daily and weekly average scores is addressed in Section 6.1.4.3. The numerator and denominators used in the derivation of weekly average and time period scores are based on the number of non-missing daily and weekly scores, respectively.

# Post-baseline ItchRO and EDQ scores:

Post-baseline morning, evening, and highest ItchRO and EDQ scores used for analysis purposes are calculated using the daily scores from the 182 days (26 weeks) immediately after the date of first dose. Post-dose weekly scores are first calculated for each of the 26-week, 7-day periods. The first 7-day period is considered 'Week 1', whereas the last 7-day period is considered as 'Week 26'. For each subject and ItchRO/EDQ efficacy variable, post-baseline scores are derived as the average of the 4- or 6-week post-dose weekly average scores for the following time periods: post-baseline to Week 6 (42 days), Week 7 to 10 (28 days), Week 11 to 14 (28 days), Week 15 to 18 (28 days), Week 19 to 22 (28 days), and Week 23 to 26 (28 days).

The handling of missing daily and weekly average scores is addressed in Section 6.1.4.3. The numerator and denominators used in the derivation of weekly average and time period scores are based on the number of non-missing daily and weekly scores, respectively.



• ItchRO(Obs) Responder is defined as a subject having a 4-week average morning ItchRO(Obs) severity change from baseline of ≤-1.0 OR an average severity score of ≤1.0.

For the purpose of determining response, the average severity score from the three 4-week periods (Weeks 15-18, 19-22, and 23-26) will be computed and used.

Before the database lock, the definition of an ItchRO(Obs) Responder may be re-defined based on outcomes of the ItchRO instrument validation performed on the analysis of data blinded to treatment. This blinded analysis, performed according to the Validation Analysis Plan (VAP), will be used to estimate a threshold of clinically meaningful change (i.e., responder definition) in the 4-week average morning ItchRO(Obs) pruritus scores. Details of the analysis will be included in a standalone VAP; results will be presented in a standalone validation analysis report.

• sBA Responder is defined as a subject having an average sBA level of <102 μmol/L (applies only if baseline sBA level was ≥102 μmol/L), OR a ≤-75% average percent change from baseline.

For the purpose of determining response, the average sBA value from Weeks 18, 22, and 26 values will be computed and used.

• FIB-4 = 
$$\frac{\textit{Age (years) x AST}\left(\frac{\textit{U}}{\textit{L}}\right)}{\textit{platelet count}\left(\frac{10^3}{\textit{µL}}\right)x\sqrt{\textit{ALT}}\left(\frac{\textit{U}}{\textit{L}}\right)}} \text{ , where age is years at sample collection time point}$$

• **APRI** = 
$$100 \text{ x} \frac{\text{AST} \left(\frac{U}{L}\right) / \text{AST ULN} \left(\frac{U}{L}\right)}{\text{platelet count} \left(\frac{10^3}{\mu L}\right)}$$
, where ULN = upper limit normal

• Ratio of Alpha Tocopherol to the sum of Cholesterol and Triglycerides (mg/g) = 1000 x alpha tocopherol (mg/dL) / [cholesterol (mg/dL) + triglycerides (mg/dL)]

For alpha tocopherol concentrations reported as below the minimum quantitation limit, half of the minimum quantitation limit is used in the calculation.

- Corrected Sodium (mEq/L) = sodium (mEq/L) + (0.002 x triglycerides [mg/dL])
- Retinol: RBP Molar Ratio (mol/mol) =  $0.0734 \text{ x retinol} (\mu g/dL) / \text{RBP} (mg/dL)$
- Anion Gap (mEq/L) = Sodium (mEq/L) Chloride (mEq/L) Bicarbonate (mEq/L)



## Osmolar Gap (mOsm/kg) = MO - CO,

where MO = measured osmolality (mOsm/kg), CO = calculated osmolality (mOsm/kg)=  $[2 \times (Sodium (mEq/L) + Potassium (mEq/L))] + [Glucose (mg/dL) / 18]$ + [BUN (mg/dL) / 2.8]

#### PELD/MELD Scores

Pediatric end-stage liver disease (PELD) score will be calculated for children under 12 years of age at the baseline visit. For children 12 years or older at the baseline visit, the model for end-stage liver disease (MELD) score will be calculated.

PELD Score =  $4.80 \times \ln(\text{total bilirubin } \lceil \text{mg/dL} \rceil) + 18.57 \times \ln(\text{INR}) - 6.87 \times \ln(\text{albumin})$ [g/dL]) + 4.36 (if patient <1 year: scores for patients listed for liver transplantation before the patient's first birthday continue to include the value assigned for age (<1 year) until the patient reaches the age of 24 months) + 6.67 (if the patient has growth failure, where growth failure is defined as a weight z-score <-2.00)

Laboratory values in the PELD equation that are <1.0 will be set to 1.0 for the calculation of the PELD score.

MELD Score =  $3.78 \times \ln (\text{total bilirubin [in mg/dL]}) + 11.2 \times \ln(\text{INR}) + 9.57 \times$ ln(creatinine [in mg/dL]) + 6.43.

Laboratory values in the MELD equation that are <1.0 will be set to 1.0 and serum creatinine values greater than 4.0 mg/dL (equivalent of 353.6 µmol/L) will be set to 4.0 for calculation of the MELD score.

Scores from PELD and MELD will be summarized separately.

#### **Treatment Duration (days) =**

Date of last dose of study drug – Date of first dose of study drug + 1 day

For participants who are missing the date of last dose of study drug, the last known contact date will be used in the calculation of treatment duration.



# **Study Drug Exposure (days) =**

Treatment duration (days) – Number of days that a participant reported missing both morning and evening doses (between the date of first and last dose)

For participants who are missing the date of last dose of study drug, the last known contact date will be used in the calculation of study drug exposure.

Compliance (%) = 100 x Study drug exposure (days) / Treatment duration (days)

Study drug compliance will not be calculated for participants whose date of last study drug is unknown.

**Total Dose** ( $\mu g/kg$ ) =  $\sum$  [ Number of doses taken<sub>i</sub> x Dose received ( $\mu g/kg$ )<sub>i</sub>] where,

i = 1 to k, (k = number of time periods participant is receiving a constant dose)

Average Daily Dose ( $\mu g/kg/day$ ) = Total Dose ( $\mu g/kg$ ) / Treatment Duration (days)

Dose variables (total dose and average daily dose) not calculated for placebo participants.

### **PedsQL Scoring Algorithm**

For each item of the PedsQL instrument (parent and participant), a 5-point response scale is used (0 = never, 1 = almost never, 2 = sometimes, 3 = often, 4 = almost always). Items are reverse-scored and linearly transformed to a 0-100 scale (0  $\rightarrow$  100, 1  $\rightarrow$  75, 2  $\rightarrow$  50,  $3 \rightarrow 25, 4 \rightarrow 0$ ), so that higher scores indicate better HRQoL (less negative impact). Scale scores are computed as the sum of the items divided by the number of items answered (this accounts for missing data). If more than 50% of the items in the scale are missing, the scale score is not computed. See PedsQL (2021) reference in Section 12 for scoring instructions on the PedsQL.

PedsQL scale scores are computed for the following:

- > Total Scale Score computed as the sum of the items over the number of items answered on the PedsQL Generic Core Scales (up to 45 items)
- ➤ Physical Health Summary Score computed as the sum of the items over the number of items answered in the Physical Functioning Scale (and Physical Symptoms Scale for infants) from the PedsQL Generic Core Scales (up to 19 items)



- Psychosocial Health Summary Score computed as the sum of the items over the number of items answered in the Emotional, Social, and Nursery/Day Care/School Functioning Scales for children ages 2 to 18 years or Emotional, Social, and Cognitive Functioning Scales for infants (<2 years) from the PedsQL Generic Core Scales (up to 26 items)</p>
- Multidimensional Fatigue Scale Score computed as the sum of the items over the number of items answered in the PedsQL Multidimensional Fatigue Scales (18 items)
- Family Impact Total Scale Score computed as the sum of the items over the number of items answered in the PedsQL Family Impact module (36 items)
- ➤ Parent Functioning Summary Score computed as the sum of the items over the number of items answered in the Physical, Emotional, Social, and Cognitive Functioning Scales from the PedsQL Family Impact module (20 items)
- Family Impact Summary Score computed as the sum of the items over the number of items answered in the Daily Activities and Family Relationships Scales from the PedsQL Family Impact module (8 items)

Total scale, physical health summary, psychosocial health summary, and multidimensional fatigue scale scores are computed individually for the parent and participant reports. Family impact and parent functioning total scale and summary scores are based on parent-reported items.

• Treatment-Emergent Adverse Event (TEAE) = In general, TEAEs are defined as AEs that start or deteriorate on or after the first dose of study drug and no later than 7 days following the last dose of study drug (for participants not participating in the extension study) or reported through the Week 26/EOT visit (for participants participating in the extension study). For participants with > 7 days of study drug interruption/withdrawal, the definition of a TEAE considers both the date of the last dose prior to drug interruption and the actual last dose (see Section 6.1.9).

Any event which started before the first dose and worsens in either intensity or frequency or changes from non-serious to serious on or after the first dose date will also be designated as a TEAE.

For any participants who die during the study and the date of death is between the date of first dose of study drug and the date of study discontinuation (as entered by the site), inclusive, all AEs (including those resulting in death) that occur during the study will be considered as TEAEs irrespective of the last dose and will be included in the TEAE summaries.





# Body Weight, Height and BMI Z-Scores

Height, weight, and body mass index (BMI) z-scores are based on a participant's sex and age at each scheduled visit. For participants less than 24 months of age, the World Health Organization (WHO) growth charts will be used to derive z-scores (WHO, 2000). For participants at least 24 months of age, the Center for Disease Control (CDC) growth charts will be used to derive z-scores (CDC, 2000).

- Length of Stay for Hospitalizations (days) = Date of discharge Date of admission + 1 day
- Time to Liver-Associated Event (days) = Date of liver-associated event Date of first dose of study drug

#### 6.1.9. Data Adjustments/Handling/Conventions

All collected data will be presented in listings. Data not subject to analysis according to this plan will not appear in any tables or graphs but will be included in the data listings.

All p-values will be displayed in four decimals and rounded using standard scientific notation (e.g., 0.xxxx). If a p-value less than 0.0001 occurs it will be shown in tables as <0.0001.

### PFIC Type and Subtype

The PFIC type (and BSEP subtype for PFIC2) is centrally assessed by a blinded PFIC genetics expert based on a review of the genotype report. Analyses will be performed according to centrally adjudicated PFIC type which will be recorded on the Genotype Adjudication file, and not what is reported within the IRT system or on the eCRF. A listing of any discrepancies between the PFIC type recorded in IRT or the eCRF and the centrally adjudicated PFIC type will be presented.

#### Subject Age

The age of a participant at screening will be used to determine the age-specific module or instrument for the appropriate ItchRO and EDQ clinical outcome questionnaire or assessment (i.e., ItchRO, EDQ, PedsQL, PIS). The same module or instrument will be completed for the duration of the study, regardless of subsequent birthdays throughout the study.

The PIC will be completed by subjects who are 9 years of age or older at the Week 26 (EOT) visit.





## **Handling of Siblings**

Because PFIC is a rare disease, siblings are allowed to enroll in the study. Siblings enrolled in the study will be assigned in a blinded manner to the same treatment arm. The data from all enrolled participants (including siblings) will be used for all primary efficacy and safety analysis. The data for only 1 sibling will be used for a sensitivity analysis on the primary efficacy endpoint and the key secondary efficacy endpoint for the primary and PFIC cohorts, independently, in the ITT Population. The choice of sibling to use in the sensitivity analysis will be made at random, unless only 1 sibling is evaluable in the specific cohort and ITT Population and the other sibling is not. In this case, the evaluable sibling will be used in the sensitivity analyses. Sibling selection for the purposes of the sensitivity analysis will be completed prior to data lock.

### Adverse Event and Concomitant Medication Coding

Adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 22.1. Prior and concomitant medications will be coded using World Health Organization Drug Dictionary (WHO-DD Enhanced version September 2019), Anatomical Therapeutic Chemical (ATC) level 2 for ATC class and level 5 (clinical substance) for preferred term.

# Prior and Concomitant Treatment Definition and Data Handling

A concomitant treatment refers to all treatment, including concomitant therapies as well as herbal treatments, vitamins, behavioral treatment, non-pharmacological treatment, such as psychotherapy, taken between the dates of the first dose of study drug and the end of the participant's participation in the study (Week 26 or Week 27), inclusive. For participants not continuing into the extension study, this period of participation is from the first day of screening through the last contact at Week 27. For participants continuing into the extension study, this period is from the first day of screening through the Week 26 visit.

Treatments that started before the first dose of study drug are considered prior treatments whether or not they were stopped prior to the first dose of study drug. Any treatment continuing or starting after the first dose of study drug will be considered as concomitant. If a treatment starts prior to the first dose of study drug and continues after the first dose of study drug, the medication will be considered as both prior and concomitant.

Medications that treat pruritus include ATC preferred terms of rifampicin, phenobarbital, alimemazine, brompheniramine maleate, cetirizine hydrochloride, desloratadine, dexchlorpheniramine maleate, dimetindene maleate, ketotifen fumarate, levocetirizine dihydrochloride, loratadine, mequitazine, promethazine, promethazine hydrochloride, ornithine aspartate, ursodeoxycholic acid, colestyramine, naltrexone, naltrexone hydrochloride, and sertraline.





For participants participating in the extension study, concomitant treatments that are ongoing as of the Week 26 visit are closed-out with a stop date of "ongoing". Concomitant treatments that are continuing from the core study (MRX-502) are copied into the extension study database with start dates entered as the original start date in the core study.

## TEAE Data Handling

If an event worsens in severity during the study, the lower grade event is marked as "Not recovered/not resolved" on the AE case report form (CRF) and an end date entered. A new event is recorded on the AE CRF with a start date that matches the end date, and the term recorded includes "Worsened" (e.g., "Worsened Headaches"). If an event becomes serious, the date that the event became serious is recorded on the AE CRF as the End Date of that AE and the Start Date of the corresponding serious adverse event (SAE).

For participants participating in the extension study, AEs that are ongoing as of the Week 26 visit are closed-out with a stop date of "ongoing". Adverse events that are continuing from the core study (MRX-502) are copied into the extension study database with start dates entered as the original start date in the core study.

#### **Events of Clinical Interest**

The following events have been defined as events of clinical interest (ECI) due to the nature of PFIC disease as well as of maralixibat:

- Diarrhoea events
- Lipid soluble vitamin (LSV) deficiency events
- Elevated transaminases events
- Elevated bilirubin events

PFIC is associated with LSV deficiency and fluctuating transaminase elevations. Maralixibat is associated with gastrointestinal disturbances such as diarrhoea.

AD-PR-109.02 Effective date: 17-Aug-2020

The list of PTs used to identify LSV deficiency events are provided in Appendix 2.

Diarrhoea events include PTs of:

- 'Diarrhoea',
- 'Intermittent Diarrhoea',
- 'Increased stool frequency'
- 'Gastroenteritis'



#### Elevated transaminases events include PTs of:

- 'Elevated liver enzymes'
- 'Transaminases abnormal'
- 'Transaminases increased'
- 'Alanine aminotransferase increased',
- 'Aspartate aminotransferase increased'
- 'Aspartate aminotransferase abnormal'
- 'Alanine aminotransferase abnormal'

#### Elevated bilirubin events include the PT of:

- 'Blood bilirubin increased',
- 'Blood bilirubin abnormal'
- 'Hyperbilirubinaemia'

### Partial Date Imputation

If partial dates occur, the convention for replacing missing dates for the purpose of calculating derived variables is as follows:

#### Partial PFIC Diagnosis Dates

For partial original PFIC diagnosis dates: (a) if only the day is missing, and the month and year match the first dose date, then the day is assigned the first day of the month (01); otherwise the day assigned is 15; and (b) if both the day and month are missing then the day/month assigned is the first day of July (01JUL), as long as the date is before the first dose date; otherwise, the day/month assigned is the first day of January (01JAN).

#### Partial AE or Medication Dates

Adverse events or medications with entirely missing start dates will be classified as treatmentemergent or concomitant, as appropriate.

For partial AE or concomitant treatment start dates: (a) if only the day is missing, and the month and year match the first dose date and the end date is on or after the first dose date, then the date is assigned the first dose date thus the event/medication will be considered as treatment-emergent/concomitant; if the month and/or year do not match the first dose date or the end date is prior to the first dose date, then the day is assigned the first day of the month (01); (b) if both the day and month are missing, and the year matches the first dose date and the end date is on or





after the first dose date, then the date is assigned the first dose date; if the year does not match the first dose date or the end date is prior to the first dose date, then the day/month are assigned the first day of the year (01JAN).

For partial end dates: (a) if only the day is missing, then the day is assigned the last day of the month; (b) if both day and month are missing, they are assigned the last day of the year (31DEC).

#### Partial Liver-Associated Event Date

For partial liver-associated event date: (a) if only the day is missing, then the day is assigned the first day of the month (01); (b) if both the day and month are missing, and the year matches the first dose date, then the date is assigned the first dose date; if the year is after the first dose date, then the day/month are assigned the first day of the year (01JAN).

### Dates of Birth

Partial or complete dates of birth are not reported by the investigative sites. Complete date of birth is required, however, to derive a participant's weight, height, and BMI z-scores. The convention for imputing missing birth dates for the purpose of statistical analysis will be based on a subject's age in years and months at baseline, as defined in Section 6.1.8.

## Lower and Upper Limit of Quantitation

In general, for quantitative laboratory values reported as "<" or "\le " the lower limit of quantitation (LLOQ), one-half of the reported value (i.e., LLOQ/2) will be used for analysis. The exception to this data treatment is for plasma maralixibat concentrations that are reported as <LLOQ, where a value of zero will be used in calculating summary statistics.

For quantitative laboratory values reported as ">" or "\geq" the upper limit of quantitation (ULOQ), the reported value (i.e., ULOQ) will be used for analysis.

#### Laboratory Test Results

For analysis purposes, repeat laboratory test results will not be used unless the original laboratory value is missing or indicated as invalid, in which case the first non-missing repeat laboratory value will be used for data analysis.

Local laboratory results are used where central laboratory results are not available.

The International System of Units (SI) will be used in reporting all efficacy and safety laboratory values, unless otherwise specified in Appendix 1.





### Dose Used in Safety Analysis

For all safety and tolerability analyses, participants will be analyzed by the treatment received. For the maralixibat treatment group, the dose of IP received at the end of the dose-escalation period, or the last dose received if the participant discontinued from the IP during the dose escalation period, will be used for the safety analysis, where specified.

## Treatment Received in Adverse Event Listings

For all AE listings, treatment received at the start of the event will be presented. For subjects on maralixibat, dose in units of  $\mu g/kg/day$  will be reported. For AEs that started within 7 days after the last dose of study drug, the last treatment received is listed. For AEs that started >7 days after the last dose of study drug, treatment received is blank. For AEs that started prior to the first dose of study drug, NT (Not Treated) will be listed.

### Treatment Duration and Exposure

For participants who are missing the date of last study drug application, for any reason, the last known contact date will be used in the calculation of treatment duration and study drug exposure. Study drug compliance will not be calculated for those participants whose date of last study drug administration is unknown.

#### Censoring for Time to First Liver-Associated Event

If a subject does not report a liver-associated event, then the time to first liver-associated event is censored at the last contact date.

### 7. Study Subjects and Demographics

Subject disposition, demographics, disease history and baseline disease, important protocol deviations, prior medications, and study drug exposure and compliance will be summarized, unless otherwise noted, by randomized treatment group and overall for the primary cohort, the PFIC cohort, and all cohorts combined (all subjects) in the Safety Population.

#### 7.1. Disposition of Subjects and Withdrawals

Subject disposition will be tabulated in all subjects, including screen failures.

Subject disposition will include tabulations of the number and proportion of participants in each of the analysis populations, completed study treatment, and discontinued early from the study (along with reasons for withdrawal). Percentages will be based on the number of participants in the Safety Population. The participant disposition tabulation will also include the number of participants screened for eligibility, the number of screen failures, the number of participants





randomly assigned to study treatment, and the number of families with siblings enrolled in the study, along with the total number of siblings.

The number and proportion of randomized and completed participants by country and investigative site, individually, will also be tabulated. Percentages will be based on the number of participants randomly assigned to study treatment.

Study drug accountability and compliance listings will be prepared for all participants, showing when the planned dosing schedule was not followed, along with the date and type of dosing deviation. Other disposition and study conduct information, including important protocol deviations will be listed.

#### 7.2. Protocol Violations and Deviations

Protocol deviations will be tracked, recorded, and reviewed prior to database lock, following the Protocol Deviation Guidance Plan for this study.

Protocol deviations will be classified as "Important" or "Not Important". An important deviation poses as a relevant operational/study conduction deviation, a possible safety issue to the participant, or it has a potential impact on the statistical analysis of the clinical data. A non-important deviation is identified as any protocol deviation that does not meet the criteria for an important deviation. Potentially important deviations will be reviewed by the Sponsor and Premier to determine the final classification as per the final Protocol Deviation Guidance Plan.

The number and proportion of participants with important protocol violations/deviations will be tabulated by category/type and treatment group in the Safety Population, for the primary cohort, the PFIC cohort, and all cohorts combined (all subjects). These protocol violations/deviations will also be presented in a participant listing by randomized treatment group.

The final decision regarding inclusion and exclusion of participants from the analysis populations will be based on a final listing of protocol deviations. This will be determined during a (blinded) review meeting before any unblinding occurs or database freeze/lock, with input from the Clinical and Biostatistics team members and approval from the Sponsor.

Additionally, inclusion and exclusion criteria not met and reasons for screen failures will be listed.

### 7.3. Demographics and Other Baseline Characteristics

Summary statistics for age at baseline, sex, race, ethnicity, region, height, height z-score, weight, weight z-score, BMI, and BMI z-score will be presented.

Tabulations for age group categories, defined as 1 to <6, 6 to <13, and 13-18 years of age, will also be presented. Given the small number of participants in the study, age categories may be





combined for presentation and analysis (e.g., <9 and  $\ge9$ ). Unless otherwise noted, age is the participant's age at the baseline visit for all evaluations and presentations.

Subjects reporting more than 1 race will be counted in a "More than one race" category for purposes of tabulating summary statistics for race.

#### Disease History and Baseline Disease Characteristics

Summary statistics will also be presented for the following baseline variables:

- PFIC type
- BSEP phenotype
- time since original diagnosis of PFIC (months)
- participants with liver masses detected on ultrasound
- participants with baseline UDCA usage
- participants with baseline Rifampicin usage
- participants above and below the median baseline sBA level; where the median is calculated separately for the primary cohort, PFIC cohort, and all subjects
- baseline pruritus assessments:
  - clinician scratch scale (CSS) score
  - patient impression of severity (PIS)
  - caregiver impression of severity (CIS)
  - ItchRO (Obs) 4-week morning average severity score
  - ItchRO (Pt) 4-week morning average severity score
  - ItchRO (Obs) 4-week evening average severity score
  - ItchRO (Pt) 4-week evening average severity score
  - ItchRO (Obs) 4-week highest daily average severity score
  - ItchRO (Pt) 4-week highest daily average severity score
  - ItchRO (Obs) 4-week morning average frequency score
  - ItchRO (Pt) 4-week morning average frequency score
  - ItchRO (Obs) 4-week evening average frequency score
  - ItchRO (Pt) 4-week evening average frequency score
  - ItchRO (Obs) 4-week highest daily average frequency score
  - ItchRO (Pt) 4-week highest daily average frequency score



- baseline levels of biochemical markers of cholestasis and liver disease and other important baseline laboratory tests:
  - total serum bile acids (sBA)
  - ALT
  - ALP
  - AST
  - GGT
  - bilirubin (total and direct)
  - albumin
  - FGF-19
  - autotaxin
  - 7α hydroxyl-4-cholesten-3-one (C4)
  - 25-hydroxyvitamin D
  - alpha tocopherol
  - prothrombin intl. normalized ratio
  - vitamin A
  - APRI
  - FIB-4
  - PELD score
  - MELD score

Subject demographics and baseline characteristics, and medical and surgical history information and prior medications, will be presented in a participant listing by randomized treatment group.

### 7.4. Prior Medications/Therapies

Prior treatments will be summarized descriptively by treatment group using the number and proportion of participants by ATC Class Level 2 (therapeutic main group) and ATC Class Level 5 (chemical substance).

Prior treatments will be presented separately from concomitant treatments.

### 7.5. Exposure and Compliance

Treatment exposure will be calculated for each participant exposed to maralixibat during the study and summarized descriptively. This analysis will be conducted for the overall 26-week treatment period.





Treatment exposure summaries will include total treatment duration (days), treatment exposure (days), total dose ( $\mu$ g/kg), and average daily dose ( $\mu$ g/kg/day).

Treatment compliance (%) will also be summarized. For a given day, a participant is considered compliant with treatment if any amount of study drug was administered. In addition to the presentation of descriptive statistics on compliance rates, treatment compliance will also be categorized and summarized as <80%, 80-<90%, and 90-100%.

Study drug accountability will be presented in a participant listing by randomized treatment group. Dosing details will be listed separately.

# 8. Efficacy Analysis

Efficacy analyses will be conducted in the ITT population separately on the primary cohort and the PFIC cohort. Analysis of the primary efficacy endpoint and the key secondary efficacy endpoint (i.e., change from baseline in sBA level) will also be performed on the primary cohort in the PP population.

Analyses on the exploratory efficacy endpoints will be performed in the ITT population separately on the primary cohort and the PFIC cohort.

The primary efficacy analysis will be performed in the primary cohort for the ITT population.

For all efficacy analyses, participants will be analyzed by the randomized treatment group assignment (maralixibat or placebo), based on the intent-to-treat principle that asserts that the effect of a treatment can be best assessed by evaluating on the basis of the intention to treat a participant (i.e., the planned treatment regimen) rather than the actual treatment given. All efficacy data will be presented in participant listings.

For the PFIC cohort analyses, PFIC type will also be used as a covariate in the MMRM analysis. For this analysis, due to the small sample sizes, PFIC4, PFIC5, and PFIC6 will be grouped together. Within the PFIC cohort, 4 PFIC types are include in the covariate: nt-PFIC2, PFIC1, PFIC3, and other (PFIC4, PFIC5, and PFIC6 group).

# 8.1. Primary Efficacy Analysis

For this study, the primary estimand is the improvement in pruritus measured as change from baseline in the average morning ItchRO(Obs) severity score in the maralixibat treatment group relative to the placebo group. In the course of the 26-week randomized treatment period, participants may be exposed to possible known or unknown inter-current events that could possibly impact the interpretation of the measures associated with the clinical question of interest, such as treatment discontinuation due to a specific adverse effect or perhaps a lack of effect. The "Hypothetical Strategy" has been adopted for handling all known inter-current events





in this study. To this end, a restricted maximum likelihood (REML)-based MMRM model conducted on the primary cohort in the ITT population will be used as the primary analysis method.

The repeated measures include post-baseline time periods during the dose escalation period (i.e., Week 1-6) and stable dosing period (i.e., Weeks 7-10, 11-14, 15-18, 19-22, and 23-26), with change from baseline in the 6- or 4-week average morning ItchRO(Obs) severity score as the dependent variable. The MMRM model will include the fixed, categorical effects of treatment group, time period, and treatment group-by-time period interaction as well as the continuous, fixed covariates of baseline 4-week average morning ItchRO(Obs) severity score and the baseline score-by-time period interaction. The MMRM analysis method is further described in Section 6.1.4.1.

The unstructured variance/covariance matrix will be used to model the variances and covariances for the six time points included in the model. The unstructured variance/covariance does not impose any restrictions on the pattern of the matrix elements. If there is a convergence issue with the unstructured covariance model, the following variance/covariance matrix structures will be used in the following order: 1) heterogeneous Toeplitz, 2) heterogeneous autoregressive of order 1, and 3) heterogeneous compound symmetry. The first variance/covariance structure which does not have a convergence problem will be the one used for the analysis. The Kenward-Roger approximation will be used to estimate denominator degrees of freedom (Kenward et al, 1997).

The primary efficacy analysis will compare maralixibat and placebo using the contrast (difference in least squares [LS] means) between treatment groups across the last 12 weeks of the study (i.e., Weeks 18, 22, and 26 combined). The analytical solution of the overall treatment effect obtained from MMRM is an equally weighted average of the 3 individual visit-specific estimates over the time period of interest (i.e., the last 12 weeks of the study). Significance tests will be based on LS means using a 2-sided significance level (2-sided 95% confidence intervals [CIs]).

The null hypothesis for the primary efficacy endpoint of the equality of maralixibat and placebo is:

H<sub>01</sub>: mean change in average morning ItchRO(Obs) severity score between baseline and Week 15 through Week 26 over the primary cohort in the two treatment groups are equal

The null hypothesis of equal treatment effect will be rejected if the statistical analysis results in a 2-sided p-value for treatment over the last 12 weeks of the study of less than or equal to 0.05. Least squares (LS) means will be calculated for each treatment group for each post-baseline time period in the model. The difference between maralixibat and placebo change from baseline in average morning ItchRO(Obs) severity score will be estimated, with the corresponding 2-sided 95% CI constructed for each time period, and the last 12 weeks (i.e., last 3 visits) of the study





combined. The change from baseline LS means with standard error, 95% CI for the LS means, p-value for testing if the LS mean is zero, LS mean difference between treatment groups (maralixibat minus placebo) with standard error, 95% CI for the LS mean difference, and p-value for testing if the treatment LS means are equal will be presented.

The trial will be claimed successful if the hypothesis of no treatment effect on the primary efficacy endpoint over the primary cohort in the ITT population is rejected at the 0.05 (2-sided) significance level.

### 8.2. Secondary Efficacy Analysis

Analysis similar to that described for the primary efficacy endpoint will be performed for each of the change from baseline secondary efficacy endpoints. For responder-type endpoints, the number and proportion of participants that are considered a "responder" will be summarized by treatment group for each analysis visit or time period, as appropriate. Barnard's exact unconditional test will be used to calculate the p-value for the difference between treatment groups.

The null hypotheses for the secondary efficacy endpoints of the equality of maralixibat and placebo are:

H<sub>02</sub>: mean change in total sBA level between baseline and average of Weeks 18, 22, and 26 over the primary cohort in the two treatment groups are equal

H<sub>03</sub>: mean change in the average morning ItchRO(Obs) severity score between baseline and Week 15 through Week 26 over the PFIC cohort in the two treatment groups are equal

H<sub>04</sub>: mean change in total sBA level between baseline and average of Weeks 18, 22, and 26 over the PFIC cohort in the two treatment groups are equal

H<sub>05</sub>: proportion of ItchRO(Obs) responders from Week 15 to Week 26 on participants in the primary cohort in the 2 treatment groups are equal

H<sub>06</sub>: proportion of sBA responders from Week 15 to Week 16 on participants in the primary cohort in the 2 treatment groups are equal

H<sub>07</sub>: proportion of ItchRO(Obs) responders from Week 15 to Week 26 on participants in the PFIC cohort in the 2 treatment groups are equal

H<sub>08</sub>: proportion of sBA responders from Week 18 to Week 26 on participants in the PFIC cohort in the 2 treatment groups are equal





A hierarchical testing procedure, as described in Section 6.1.3 will be used in the comparisons between maralixibat and placebo on the primary and secondary efficacy endpoints in the ITT population.

All tests will be performed as 2-sided tests at the 0.05 level of significance.

### 8.3. Sensitivity and Supportive Analyses for Primary and Secondary Endpoints

Sensitivity and/or supportive analysis will be performed on the primary and secondary efficacy endpoints to quantify the possible impact of missing data and the use of potentially correlated sibling data, and to demonstrate the robustness of the conclusions.

Sensitivity analysis will be performed on the primary efficacy endpoint and key secondary efficacy endpoint in the primary cohort and PFIC cohort, individually, in the ITT analysis population.

Although the assumption of MAR, as used for the primary efficacy analysis method, is often reasonable in clinical trials, the possibility of MNAR data cannot be ruled out. Sensitivity analyses to deal with missing data will use MI methods where missing values are imputed individually under both a plausible MAR and MNAR scenario. Two sensitivity analysis models, one based on the standard MAR imputation approach and the other on a tipping point analysis, will be used to examine robustness of the primary analysis results (see Section 6.1.4.2).

If siblings are evaluable for efficacy, the primary analysis method described above for the primary efficacy endpoint and the key secondary efficacy endpoint will be repeated as a sensitivity analysis in which only one of sibling pairs or multiples will be used. The choice of which sibling to use in the sensitivity analysis will be made at random before the MRX-502 study is unblinded (see Section 6.1.9).

Summary statistics on the primary efficacy endpoint and the key secondary efficacy endpoint will also be presented descriptively by treatment group and visit, overall and for each of the following subgroups on the primary cohort in the ITT analysis population:

- Region (Asia, Europe, Middle East, North America, and South and Central America)
- Age at baseline (1 year to <6 years old, 6 years to < 13 years, and 13-18 years old)
- Sex (male, female)
- Race (White, Asian, Black or African American, American Indian or Alaska Native, Multiple)
- Baseline sBA (< median, ≥ median; where only subjects in the primary cohort are used to calculate the baseline median sBA level)
- Baseline ursodeoxycholic acid (UDCA) usage (yes, no)



- Baseline Rifampicin usage (yes, no)
- BSEP type of primary cohort (non-truncating PFIC2) participants (BSEP 1, BSEP 2)

# 8.4. Adjustment for Multiplicity

A hierarchical testing procedure will be used in the comparisons between maralixibat and placebo on the primary and secondary efficacy endpoints in the ITT population using the primary analysis method (as described for the primary endpoint). The hierarchical order for testing the null hypotheses is listed in Section 6.1.3.

The effect of such a procedure maintains study-wide Type I error control, ensuring that no confirmatory claims can be based on the endpoint(s) that have a testing rank lower than that endpoint whose null hypothesis was the first that could not be rejected. Those tests will be considered as exploratory without any type I error control for the additional subsequent tests.

# 8.5. Exploratory Efficacy Analysis

Analyses will be conducted for the exploratory efficacy endpoints separately on the primary cohort and the PFIC cohort.

Analysis similar to that described for the primary efficacy endpoint (i.e., MMRM) will be performed for each exploratory endpoint that is based on change from baseline values on continuous variables. The repeated measures in the MMRM model will include the post-baseline visits as specified for each above-listed endpoint, with change from baseline value as the dependent variable. The MMRM model will include the fixed, categorical effects of treatment group, visit, and treatment group-by-visit interaction as well as the continuous, fixed covariates of baseline and the baseline-by-visit interaction. Least squares means will be calculated for each treatment group for each post-baseline visit in the model. The difference between maralixibat and placebo change from baseline in each outcome variable will be estimated, with the corresponding 2-sided 95% CI constructed for each visit. Change from baseline LS means with standard error, 95% CI for the LS means, p-value for testing if the LS mean is zero, LS mean difference between treatment groups (maralixibat minus placebo) with standard error, 95% CI for the LS mean difference, and p-value for testing if the treatment LS means are equal will be calculated for each visit. For the ItchRO (Obs and Pt) and EDQ (Obs and Pt) endpoints that compare treatment groups across the last 12 weeks of the study, the same methods as described for the primary analysis of the primary efficacy endpoint will be applied. The number of observations, mean, 95% CI on the mean, standard deviation, median, minimum, and maximum on both the observed and change from baseline values will also be summarized by treatment group for each visit including the end of study visit (Week 26/EOT).

For responder-type endpoints (i.e., efficacy variables involving binary outcomes), the number and proportion of participants that are considered a "responder" will be summarized by treatment





group for each analysis visit or time period, as appropriate. Barnard's exact unconditional test will be used to calculate the p-value for the difference between treatment groups.

For responder-type endpoints with ordinal measures, the Cochran-Mantel-Haenszel (CMH) test will be applied to test for no association between treatment group and the variable of interest. For the OL and ARW treatment phases, the number and percentage of subjects at each level of the 7-or 5-point scale, for PIC/CIC or CGTB respectively, will be presented overall and for each treatment group during the RW phase. For the RW phase, the number and percentage of subjects at each level will be presented by the randomized treatment group. For ordinal non-binary outcomes, the CMH test will be used to take the ordinal nature of the variable into account.

The number and proportion of subjects with total sBA % decrease from baseline to Weeks 2, 6, 10, 14, 18, 22, and 26 within the following categories: >75% (large decrease), 0-75% (decrease), and <0% (increase) will be analyzed using a CMH test to test for no association between treatment group and the variable of interest at each analysis visit.

A Student's t-test, assuming unequal variances, will be used to compare treatment differences on the number of days the morning ItchRO(Obs) severity score ≤ 1 over the last 84 days (i.e., study day 99 through 182, inclusive). Satterthwaite's method for computing standard error of the mean of the difference will be used. A conservative approach will be taken for subjects with missing morning severity scores during this 84-day period, including those subject that withdraw early from the study. Missing data will be treated as a severity score of >1.

Time to first liver-associated event (PEBD surgery, listing for liver transplantation, liver decompensation [hepatic encephalopathy, variceal bleeding, ascites, and spontaneous bacterial peritonitis] events, HCC, and death) will be compared among treatments using Kaplan-Meier product-limit survival curve estimates. The median and other quartiles for time to first liver-associated event, along with 2-sided 95% CIs, will be estimated based on the Kaplan-Meier method. Both a log-rank test and a Wilcoxon test will be used to test for treatment differences.

All tests will be performed as 2-sided tests at the 0.05 level of significance.

Sensitivity analyses are not planned to be performed on the exploratory efficacy endpoints.

### 9. Safety and Tolerability Analysis

All safety analyses will be performed on the Safety Population, defined as all participants who were randomized and received at least 1 dose of study drug. Analyses will be conducted separately on the primary cohort, the PFIC cohort, and all cohorts combined (all subjects).

Safety measures including AEs, clinical laboratory values, physical examination findings (including body weight, height, and BMI), vital signs, ECGs, and concomitant treatment usage will be summarized descriptively. No inferential statistical tests will be performed, unless





otherwise specified. For quantitative variables, descriptive statistics including number of observations, mean, median, standard deviation, minimum, and maximum will be presented for observed and change from baseline values at each study visit. Qualitative variables will be summarized using counts and percentages.

Safety data collected at the baseline visit (Visit 1/Day 0) or the last preceding visit if not collected at Visit 1 will be used as the baseline value for safety analyses.

All safety and tolerability data will be presented in participant listings.

#### 9.1. Adverse Events

All summaries of AEs will be based on TEAEs unless specified otherwise. TEAEs are defined as described in Section 6.1.8 (Derived Variables).

Adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). The number and proportion of participants who experience the event according to MedDRA system organ class (SOC) and preferred term (PT) will be presented by treatment group. Treatment-emergent adverse events related to study drug, AEs leading to withdrawal, SAEs, and deaths will be similarly summarized.

A summary of TEAEs will be presented by treatment group. The summary will include the total number and percent of participants reporting:

- Any TEAEs
- Any treatment-related TEAE
- Any severe TEAE
- Any severe treatment-related TEAE
- Any serious TEAE
- Any serious treatment-related TEAE
- Any TEAE leading to permanent study drug discontinuation
- TEAEs resulting in death

A participant reporting multiple cases of the same AE will be counted once within each SOC and similarly counted once within each PT. Treatment-emergent AEs summarized by SOC and PT will be sorted in alphabetical order of the SOC, and by descending frequency order of the PT within each SOC.

Additionally, the following subgroup analyses will be explored for the summary of TEAEs and the incidence of TEAEs by SOC and PT indicated above:



- Age at baseline (1 year to <6 years old, 6 years to < 13 years, and 13-18 years old)
- Sex (male, female)
- Race (available races in the study)

Missing and partially missing AE start and/or stop dates will be imputed, for the purpose of statistical analysis, according to the specifications described in Section 6.1.9.

Listings of AEs will be presented in by-participant listings, detailing the participant cohort (primary [nt-PFIC2], PFIC or other), treatment received at the start of the event including dose for active study drug, SOC, PT, verbatim term given by the investigator, onset date and study day, end date and study day, event duration, severity, relationship to study drug, outcome, action taken with study drug, seriousness, and treatment required. Events that are treatment-emergent will be flagged.

### 9.1.1. Adverse Events Leading to Discontinuation of Study Drug

AEs that lead to permanent discontinuation of study drug will be tabulated by treatment group. Subject listings of AEs that lead to permanent discontinuation of study drug will also be presented.

#### 9.1.2. Deaths and Serious Adverse Events

Treatment-emergent SAEs will be summarized in the same manner as AEs that lead to permanent discontinuation of study drug. Subject listings of all SAEs will also be presented.

Any deaths that occur during the study will be presented in a participant listing. The listing will include participant ID, participant cohort, study drug and dose received at the time of death (or the last study drug/dose received prior to death), date of death, number of days from the 1st and last dose, MedDRA PT, and relationship to study drug.

#### 9.1.3. Events of Clinical Interest

Due to the nature of PFIC disease, as well as maralixibat, the following events have been defined as ECI: diarrhoea events, LSV deficiency events, elevated transaminases, and elevated bilirubin. For each of the ECI, the PTs are described in Section 6.1.9.

The incidence of ECI will be summarized in the same manner as AEs that lead to permanent discontinuation of study drug.

The clinical protocol references adverse events of special interest; however, the study has no such events.





# 9.2. Clinical Laboratory Evaluations

Safety laboratory test results will be summarized descriptively by study visit and treatment group as observed and change from baseline values. The number and proportion of participants with clinical laboratory values below, within, or above the normal range by time point and in relation to baseline will be tabulated for each select lipid soluble vitamin laboratory analytes by treatment group in a shift table. The shift table will include the following LSVs: 25-hydroxyvitamin D (ng/mL), alpha tocopherol (mg/dL), INR, and vitamin A ( $\mu$ g/dL).

All safety laboratory test parameters will be presented by panel in participant listings.

Efficacy laboratory tests (i.e., total sBA, ALT, AST, ALP, total and direct bilirubin, GGT, C4, FGF-19, autotaxin, FIB-4, APRI, PELD and MELD) will not be included in safety summaries or listings. A separate participant listing for efficacy labs will be presented.

# 9.3. Vital Signs and Weight/Height Measurements

Vital signs (temperature, systolic and diastolic blood pressure, heart rate, and respiratory rate), weight, height, and BMI will be summarized descriptively by study visit and treatment group as observed and change from baseline values. Weight, height, and BMI measurements will also be summarized as a z-score for a participant's age and sex.

## 9.4. Electrocardiograms

Descriptive summaries will be presented for ECG measures of PR interval, QRS duration, and QT interval corrected using both Bazett's and Fridericia's formula (QTcB and QTcF). The number and proportion of participants with normal, abnormal-not clinically significant, and abnormal-clinically significant ECG results will also be summarized. These summaries will be presented by study visit and treatment group.

#### 9.5. Liver Ultrasound

Liver ultrasound (or MRI) results will be presented in participant listings.

### 9.6. Concomitant Medications/Therapies

Concomitant treatments will be summarized descriptively by treatment group using the number and proportion of participants by ATC Class Level 2 (therapeutic main group) and ATC Class Level 5 (chemical substance).

Prior treatments will be presented separately from concomitant treatments. Any treatments continuing or starting after the first dose of study drug will be considered concomitant. If a





treatment starts prior to the first dose of study drug and continues after the first dose of study drug, it will be considered both prior and concomitant.

## 10. Other Planned Analysis

Healthcare utilization and pharmacokinetic analyses will be performed on the Safety Population, conducted separately on the primary cohort, the PFIC cohort, and all cohorts combined (all subjects).

#### 10.1. Healthcare Utilization

Healthcare resource utilization variables include the number of hospitalizations, emergency room visits, the length of stay for hospitalization (days), surgeries and procedures related to the participant's PFIC condition, and the number of days the caregiver missed from work due to healthcare resource utilization events. Healthcare utilization data is collected at Weeks 2, 6, 10, 14, 18, 22, 26, and the Week 27 follow-up and covers the time period since the last on-site visit.

Subjects that visit the emergency room and the visit results in the subject being admitted to the hospital will be counted in both categories.

Number and percent of subjects and number of occurrences will be presented across the entire post-baseline study period, between clinic visits from baseline through Week 27 Follow-up, by treatment group for PFIC-related hospitalizations and ER visits. For length of hospital stays and number of days a caregiver missed work, summary statistics on a subject-level basis will be presented.

#### 10.2. Pharmacokinetic Analyses

Systemic concentrations of maralixibat in plasma will be determined at pre-dose and at approximately 2.5 hours after the morning dose at Week 10 and Week 26 (EOT/ET). Summary statistics (number of observations, mean, standard deviation, coefficient of variation, median, minimum, maximum, and geometric mean) will be determined for maralixibat concentrations at each analysis visit.

### 11. Changes from Protocol Planned Analysis

The PP Population has been re-defined as all participants in the ITT Population who receive at least 1 dose of study drug and do not have any important protocol violations or deviations that have a potential impact on the efficacy analysis.

The sensitivity analysis using placebo-based MI for handling missing data has been replaced with a tipping point approach.





The number and proportion of subjects with total sBA % decrease from baseline to Weeks 2, 6, 10, 14, 18, 22, and 26 within the following categories: >75%, 0-75%, and <0% have been added as an exploratory endpoint. The analysis will be performed using a CMH test.

The number of days morning ItchRO(Obs) severity score ≤1 for the last 12 weeks (84 days) of the study has been added as an exploratory endpoint. The analysis will be performed using a Student's t-test.

The following exploratory endpoints listed in the protocol have been removed. They may be included after the finalization of the analysis plan for adhoc or posthoc analyses:

- Proportion of participants with elevated liver biochemistry (i.e., >ULN at baseline), whose liver biochemistry normalize (≤ULN) at Weeks 2, 6, 10, 14, 18, 22, and 26
- Mean change from baseline in weekly average morning, evening, and highest daily ItchRO(Obs) severity and frequency scores, individually, to each post-baseline week, and Weeks 15 to 26 combined
- Proportion of days with a morning/evening/highest daily ItchRO(Obs)/ItchRO(Pt) severity/frequency score ≤1, individually, at the participant level from baseline to Week 6 (overall and weekly), Weeks 7-10, 11-14, 15-18, 19-22, 23-26, and 15-26
- Proportion of participants in each change from baseline category of the CSS at Weeks 2, 4, 6, 10, 14, 18, 22, and 26
- Proportion of participants in each change from baseline category of the CIS and PIS, individually, at Weeks 4, 6, 10, 14, 18, 22, and 26
- Mean change from baseline in average (6 week average for Week 6 and 4 week average afterwards) morning, evening, and highest daily EDQ(Pt) severity scores, individually, to Weeks 6, 10, 14, 18, 22, 26, and Weeks 15 to 26 combined
- Proportion of responders at Weeks 6, 10, 14, 18, 22, 26, and any of those weeks, where a responder is defined as having:
  - a) 4-week average morning ItchRO(Obs) severity change from baseline of  $\leq$ -1.0 or an average score of  $\leq$ 1.0 AND a normalization or change from baseline in sBA of  $\leq$ -75%, or average sBA level <102  $\mu$ mol/L
  - b) 4-week average morning ItchRO(Obs) severity change from baseline of ≤-1.0 or a score of <1.0
  - c) a normalization or percent change from baseline in sBA of ≤-75%, or average sBA level <102 µmol/L



- Mean change from baseline in average sleep disturbance scores over time (4-week average score at Weeks 6, 10, 14, 18, 22, 26, and average of Weeks 18, 22, and 26), based on sleep-related questions on the PedsQL (parent), Child PedsQL (young child), and Child PedsQL (child and teen) questionnaires, individually
- Proportion of "no" answers for sleep-related questions on the ItchRO(Obs) morning, ItchRO(Obs) evening, and ItchRO(Pt) morning, individually, at the participant level for post-baseline to Week 6, Weeks 7 to 10, Weeks 11 to 14, Weeks 15 to 18, Weeks 19 to 22, Weeks 23 to 26, Week 15 to Week 26, and overall (post-baseline to Week 26)
- Proportion of participants who experience an improvement from baseline in height z-score or weight z-score (i.e., change from baseline >0) at Weeks 2, 4, 6, 10, 14, 18, 22, and 26
- Mean change from baseline in bile acid subspecies to Weeks 10, 18, and 26
- Mean change from baseline in C4, FGF-19, and autotaxin to Weeks 6, 10, 18, and 26 in the PFIC cohort
- Proportion of participants with an elevated liver biochemistry laboratory value at baseline that normalize post-baseline for sBA, ALT, AST and TSB, independently
- Correlation analyses between sBA and pruritus severity

The exploratory objective of evaluating the efficacy of maralixibat vs placebo in the primary cohort on responder rates for various pruritus measures, sBA and biomarkers has been updated to only include responder rates for pruritus severity and total sBA.

In general, analysis on continuous repeated-measures efficacy variables will include a comparison of maralixibat and placebo using the contrast between treatment groups across the last 12 weeks of the study (i.e., Weeks 18, 22, and 26 combined) as described in Section 8.1.

Sensitivity analyses will be performed on the primary efficacy endpoint and the key secondary efficacy endpoint in the primary cohort and PFIC cohort, individually, in the ITT analysis population. The clinical protocol describes sensitivity analysis on the primary and all secondary efficacy endpoints.

Analysis of the primary efficacy endpoint and the key secondary efficacy endpoint (i.e., change from baseline in sBA level) will be performed on the primary cohort in the PP population. The clinical protocol describes analysis in the PP population on all secondary efficacy endpoints.

Treatment-emergent AEs will not be summarized by severity and relationship to study drug.

The clinical protocol references adverse events of special interest; however, the study has no such events.





Total lipids, referenced in the clinical protocol, were not measured. For the following laboratory parameters the sum of cholesterol and triglycerides were used: ratio of alpha tocopherol to the sum of cholesterol and triglycerides, and corrected sodium (see Section 6.1.8).

The clinical protocol states that the number and proportion of subjects with potentially clinically important values for select vital signs, laboratory, and ECG results, individually, will be presented by treatment group. These analyses have been removed from the planned analysis.

Continuous healthcare resource utilization measures will be summarized as the number and percent of subjects and number of occurrences, presented across the entire post-baseline study period (between clinic visits from baseline through Week 27 follow-up), instead of as described in the protocol.

#### 12. References

ASA. (2018) Ethical Guidelines for Statistical Practice. Prepared by the Committee on Professional Ethics, April 2018. http://www.amstat.org/about/ethicalguidelines.cfm

CDC (2000). Centers for Disease Control growth charts – A SAS Program for the 2000 CDC Growth Charts (ages 0 to <20 years)

(www.cdc.gov/nccdphp/dnpao/growthcharts/resources/sas.htm)

Cnaan A., Laird N. M., Slasor P. 1997. Using the general linear mixed model to analyse unbalanced repeated measures and longitudinal data. *Stat Med.*, 16, 2349-2380.

EMA (2010). European Medicines Agency. Guideline on Missing Data in Confirmatory Clinical Trials.

ICH (1998). ICH Harmonised Tripartite Guideline. Statistical Principles for Clinical Trials E9; 1998. https://database.ich.org/sites/default/files/E9 Guideline.pdf

Kenward M. G., Roger J. H. 1997. Small sample inference for fixed effects from restricted maximum likelihood. *Biometrics*, 53, 983-997.

Little R., Rubin D. 1987. Statistical Analysis with Missing Data. New York: John Wiley.

Little R., Yau L. 1996. Intent-to-Treat Analysis for Longitudinal Studies with Drop-Outs, *Biometrics*. 52. 1324-1333.

Mallinckrodt C. H., Clark W. S., David S. R. 2001. Accounting for dropout bias using mixed-effects models. *Journal of Biopharmaceuticals Statistics*, 11, 9-21.

Mallinckrodt C. H., Lane P. W., Schnell D., Peng Y., Mancuso J. P. 2008. Recommendations for the Primary Analysis of Continuous Endpoints in Longitudinal Clinical Trials. *Drug Information Journal*, 42, 303-319.





Mallinckrodt C. H., Roger J., Chuang-Stein C., Molenberghs G., O'Kelly M., Ratitch B., Janssens M., Bunouf P. 2013. Recent Developments in the Prevention and Treatment of Missing Data. *Drug Information Journal*, 48, 68-80.

Molenberghs G., Thijs H., Jansen I., et al. 2004. Analyzing incomplete longitudinal clinical trial data. *Biostatistics*, 5, 445-464.

Molenberghs G., Kenward M. G. 2007. Missing Data in Clinical Studies. New York: Wiley.

PedsQL (2021). The PedsQL Measurement Model for the Pediatric Quality of Life Inventory – Scoring Instructions (www.pedsql.org)

RSS (2014). The Royal Statistical Society: Code of Conduct, 2014. http://www.rss.org.uk/Images/PDF/join-us/RSS-Code-of-Conduct-2014.pdf.

Schafer J. L. 1997. Analysis of Incomplete Multivariate Data. New Yori: Chapman & Hall.

Siddiqui O., Hung H. M., O'Neill R. 2009. MMRM vs. LOCF: a comprehensive comparison based on simulation study and 25 NDA datasets. *Journal of Biopharmaceuticals Statistics*, 19(2), 227-246.

Verbeke G., Molenberghs G. 2000. *Linear Mixed Models for Longitudinal Data*. New York: Springer.

WHO (2000). World Health Organization growth charts – A SAS Program for the WHO Growth Charts (ages 0 to <2 years) (www.cdc.gov/nccdphp/dnpao/growthcharts/resources/sas-who.htm)

### 13. Tables, Listings, and Figures

All listings, tables, and figures will have a header showing the sponsor company name (Mirum Pharmaceuticals, Inc.) and protocol (MRX-502), and a page footer showing the file name and path, and the date/time of program execution along with the database data cut date.

The following reporting conventions will be adopted for the presentation of study data. These conventions will enhance the review process and help to standardize the presentation with common notations.

#### **General Reporting Conventions**

- All tables and data listings will be developed in landscape orientation.
- Specialized text styles, such as bolding, italics, borders, shading, and superscripted and subscripted text will not be used in tables, figures, and data listings unless they add significant value to the table, figure, or data listing.
- Only standard keyboard characters should be used in tables and data listings. Special characters, such as nonprintable control characters, printer-specific characters, or font specific characters, will not be used on a table, figure, or data listing.


- Adverse events with missing MedDRA coding will have their system organ class and/or preferred term presented as "Not Coded" in the tables. The "Not Coded" frequencies will be sorted to the end of the tables. Adverse events that are not coded are not expected.
- Programming notes may be inserted into the shells, these notes will not appear in the final output.

#### **Population Summary Conventions**

- Population sizes may be presented for each classification factor as totals in the column header as (N=xxx), where appropriate.
- All population summaries for categorical variables will include all categories that were planned and for which the participants may have had a response. Percentages corresponding to null categories (cells) will be suppressed; however, counts and percentages of missing values may be needed. Counts of zero will be presented as '0', without the percentage.
- All population summaries for continuous variables will include: n, mean, SD, median, minimum, and maximum. Other summaries (e.g., number missing, geometric mean, median, quartiles, 95% CIs, and coefficient of variation [CV] or % CV) may be used as appropriate. The precision of the maximum and minimum will match the maximum precision in the data. The mean and median will have 1 additional decimal place. The SD will have 2 additional decimal places.
- All percentages are rounded and reported to a single decimal point (xx.x%).

#### 13.1. Planned Table Descriptions

The following are planned summary tables for protocol number MRX-502. The table numbers are place holders only and will be determined when the tables are produced. The efficacy outputs are ordered to account for the hierarchical testing structure as outlined in Section 6.1.3, where possible. For cases where multiple study visits for the same parameter are tested, those visits are consolidated on a single table for ease of review and referencing results. Similarly, for cases where multiple analysis populations or cohort groups are presented, this data will be consolidated on a single table, when practical.

The table shells will be provided under a separate document.

#### 13.1.1. Subject Data

Table 3: Subject Data Summary Tables

| Number | Population | Title |
|---|---|---|
| 14.1.1.1 | All Subjects | Subject Disposition |
| 14.1.1.2 | Safety | Number of Randomized and Completed Subjects by Country |

AD-PR-109.02 Effective date: 17-Aug-2020





| 14.1.1.3 | Safety | Number of Randomized and Completed Subjects by Investigative Site |
|---|---|---|
| 14.1.2 | Safety | Important Protocol Violations/Deviations |
| 14.1.3 | Safety | Demographics and Baseline Characteristics |
| 14.1.4 | Safety | Disease History and Baseline Disease Characteristics |
| 14.1.5 | Safety | Prior Medications/Therapies |
| 14.1.6 | Safety | Study Drug Compliance |

## 13.1.2. Efficacy Data

Table 4: Efficacy Data Summary Tables

| Number | Population | Title |
|---|---|---|
| 14.2.1.x Primary | 14.2.1.x Primary Analysis | |
| 14.2.1.1 | ITT – Primary<br>Cohort | Change from Baseline in ItchRO(Obs) Severity Score Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.1.2 | ITT – Primary<br>Cohort | Change from Baseline in ItchRO(Obs) Severity Score MMRM Model Effects |
| 14.2.2.x Secondar | y Analysis | |
| 14.2.2.1.1 | ITT – PFIC Cohort | Change from Baseline in ItchRO(Obs) Severity Score Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.2.1.2 | ITT – PFIC Cohort | Change from Baseline in ItchRO(Obs) Severity Score MMRM Model Effects |
| 14.2.2.2.1 | ITT | Change from Baseline in Total sBA (µmol/L) Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.2.2.2 | ITT | Change from Baseline in Total sBA (µmol/L) MMRM Model Effects |
| 14.2.2.3 | ITT | Proportion of Responders |
| 14.2.3.x Sensitivit | 14.2.3.x Sensitivity Analysis | |
| 14.2.3.1.1 | ITT | Change from Baseline in Morning ItchRO(Obs) Severity Score – Sibling Sensitivity Analysis Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.3.1.2 | ITT | Change from Baseline in Morning ItchRO(Obs) Severity Score – Sibling Sensitivity Analysis MMRM Model Effects |



| Number | Population | Title |
|---|---|---|
| 14.2.3.2 | ITT | Change from Baseline in Morning ItchRO(Obs) Severity Score –<br>Multiple Imputation Sensitivity Analysis<br>Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.3.3 | ITT | Change from Baseline in Morning ItchRO(Obs) Severity Score to<br>Average of Last 12 Weeks – Tipping Point Sensitivity Analysis |
| 14.2.3.4.1 | ITT | Change from Baseline in Total sBA (µmol/L) – Sibling Sensitivity<br>Analysis<br>Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.3.4.2 | ITT | Change from Baseline in Total sBA (µmol/L) – Sibling Sensitivity Analysis MMRM Model Effects |
| 14.2.3.5 | ITT | Change from Baseline in Total sBA (µmol/L) – Multiple Imputation<br>Sensitivity Analysis<br>Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.3.6 | ITT | Change from Baseline in Total sBA (µmol/L) to Average of Weeks 18, 22, and 26 – Tipping Point Sensitivity Analysis |
| 14.2.4.x Explorate | 14.2.4.x Exploratory Analysis | |
| 14.2.4.1.1 | PP – Primary Cohort | Change from Baseline in Morning ItchRO(Obs) Severity Score Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.1.2 | PP – Primary Cohort | Change from Baseline in Morning ItchRO(Obs) Severity Score<br>MMRM Model Effects |
| 14.2.4.2.1 | PP – Primary Cohort | Change from Baseline in Total sBA (µmol/L) Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.2.2 | PP – Primary Cohort | Change from Baseline in Total sBA (μmol/L) MMRM Model Effects |
| 14.2.4.3.1 | ITT – Primary<br>Cohort | Change from Baseline in Weekly Average Morning ItchRO(Obs) Severity Score Descriptive Statistics by Analysis Week |
| 14.2.4.3.2 | ITT – Primary<br>Cohort | Change from Baseline in Weekly Average Morning ItchRO(Obs) Severity Score by Region Descriptive Statistics by Analysis Week |
| 14.2.4.3.3 | ITT – Primary<br>Cohort | Change from Baseline in Weekly Average Morning ItchRO(Obs) Severity Score by Age at Baseline Descriptive Statistics by Analysis Week |



| Number | Population | Title |
|---|---|---|
| 14.2.4.3.4 | ITT – Primary<br>Cohort | Change from Baseline in Weekly Average Morning ItchRO(Obs)<br>Severity Score by Sex |
| | | Descriptive Statistics by Analysis Week |
| 14.2.4.3.5 | ITT – Primary<br>Cohort | Change from Baseline in Weekly Average Morning ItchRO(Obs) Severity Score by Race Descriptive Statistics by Analysis Week |
| 14.2.4.3.6 | ITT – Primary<br>Cohort | Change from Baseline in Weekly Average Morning ItchRO(Obs) Severity Score by Baseline Median sBA Descriptive Statistics by Analysis Week |
| 14.2.4.3.7 | ITT – Primary<br>Cohort | Change from Baseline in Weekly Average Morning ItchRO(Obs) Severity Score by Baseline UDCA Usage Descriptive Statistics by Analysis Week |
| 14.2.4.3.8 | ITT – Primary<br>Cohort | Change from Baseline in Weekly Average Morning ItchRO(Obs) Severity Score by Baseline Rifampicin Usage Descriptive Statistics by Analysis Week |
| 14.2.4.3.9 | ITT – Primary<br>Cohort | Change from Baseline in Weekly Average Morning ItchRO(Obs) Severity Score by BSEP Type Descriptive Statistics by Analysis Week |
| 14.2.4.4.1 | ITT – Primary<br>Cohort | Change from Baseline in Total sBA (µmol/L) Descriptive Statistics by Analysis Week |
| 14.2.4.4.2 | ITT – Primary<br>Cohort | Change from Baseline in Total sBA (µmol/L) by Region Descriptive Statistics by Analysis Week |
| 14.2.4.4.3 | ITT – Primary<br>Cohort | Change from Baseline in Total sBA (µmol/L) by Age at Baseline<br>Descriptive Statistics by Analysis Week |
| 14.2.4.4.4 | ITT – Primary<br>Cohort | Change from Baseline in Total sBA (µmol/L) by Sex<br>Descriptive Statistics by Analysis Week |
| 14.2.4.4.5 | ITT – Primary<br>Cohort | Change from Baseline in Total sBA (µmol/L) by Race<br>Descriptive Statistics by Analysis Week |
| 14.2.4.4.6 | ITT – Primary<br>Cohort | Change from Baseline in Total sBA (µmol/L) by Baseline Median sBA Descriptive Statistics by Analysis Week |
| 14.2.4.4.7 | ITT – Primary<br>Cohort | Change from Baseline in Total sBA (µmol/L) by Baseline UDCA Usage Descriptive Statistics by Analysis Week |
| 14.2.4.4.8 | ITT – Primary<br>Cohort | Change from Baseline in Total sBA (µmol/L) by Baseline Rifampicin Usage Descriptive Statistics by Analysis Week |



| Number | Population | Title |
|---|---|---|
| 14.2.4.4.9 | ITT – Primary<br>Cohort | Change from Baseline in Total sBA (µmol/L) by BSEP Type<br>Descriptive Statistics by Analysis Week |
| 14.2.4.5.1 | ITT | Change from Baseline in ALT (U/L) Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.5.2 | ITT | Change from Baseline in ALT (U/L) MMRM Model Effects |
| 14.2.4.6.1 | ITT | Change from Baseline in AST (U/L) Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.6.2 | ITT | Change from Baseline in AST (U/L) MMRM Model Effects |
| 14.2.4.7.1 | ITT | Change from Baseline in Total Bilirubin (mg/dL) Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.7.2 | ITT | Change from Baseline in Total Bilirubin (mg/dL) MMRM Model Effects |
| 14.2.4.8.1 | ITT | Change from Baseline in Direct Bilirubin (mg/dL) Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.8.2 | ITT | Change from Baseline in Direct Bilirubin (mg/dL) MMRM Model Effects |
| 14.2.4.9.1 | ITT | Change from Baseline in ALP (U/L) Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.9.2 | ITT | Change from Baseline in ALP (U/L) MMRM Model Effects |
| 14.2.4.10.1 | ITT | Change from Baseline in GGT (U/L) Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.10.2 | ITT | Change from Baseline in GGT (U/L) MMRM Model Effects |
| 14.2.4.11.1 | ITT | Change from Baseline in FIB-4 Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.11.2 | ITT | Change from Baseline in FIG-4 MMRM Model Effects |
| 14.2.4.12.1 | ITT | Change from Baseline in APRI Tabulation of Fitted Summary Statistics from MMRM |



| Number | Population | Title |
|---|---|---|
| 14.2.4.12.2 | ITT | Change from Baseline in APRI<br>MMRM Model Effects |
| 14.2.4.13.1 | ITT | Change from Baseline in PELD Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.13.2 | ITT | Change from Baseline in PELD MMRM Model Effects |
| 14.2.4.14 | ITT | Total sBA Shift from Baseline: Number and Proportion of Subjects |
| 14.2.4.15 | ITT | Number of Days Morning ItchRO(Obs) Severity Score ≤1<br>Over the Last 84 Study Days |
| 14.2.4.16 | ITT | Number and Proportion of Subjects with Morning ItchRO(Obs) Severity Score ≤1 for >50% of Time Period |
| 14.2.4.17.1.1 | ITT – Primary<br>Cohort | Change from Baseline in ItchRO(Obs) Frequency Score Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.17.1.2 | ITT – Primary<br>Cohort | Change from Baseline in ItchRO(Obs) Frequency Score MMRM Model Effects |
| 14.2.4.17.2.1 | ITT – PFIC Cohort | Change from Baseline in ItchRO(Obs) Frequency Score Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.17.2.2 | ITT – PFIC Cohort | Change from Baseline in ItchRO(Obs) Frequency Score MMRM Model Effects |
| 14.2.4.18.1.1 | ITT – Primary<br>Cohort | Change from Baseline in ItchRO(Pt) Severity Score Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.18.1.2 | ITT – Primary<br>Cohort | Change from Baseline in ItchRO(Pt) Severity Score MMRM Model Effects |
| 14.2.4.18.2.1 | ITT – PFIC Cohort | Change from Baseline in ItchRO(Pt) Severity Score Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.18.2.2 | ITT – PFIC Cohort | Change from Baseline in ItchRO(Pt) Severity Score<br>MMRM Model Effects |
| 14.2.4.19.1.1 | ITT – Primary<br>Cohort | Change from Baseline in ItchRO(Pt) Frequency Score Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.19.1.2 | ITT – Primary<br>Cohort | Change from Baseline in ItchRO(Pt) Frequency Score<br>MMRM Model Effects |
| 14.2.4.19.2.1 | ITT – PFIC Cohort | Change from Baseline in ItchRO(Pt) Frequency Score Tabulation of Fitted Summary Statistics from MMRM |



| Number | Population | Title |
|---|---|---|
| 14.2.4.19.2.2 | ITT – PFIC Cohort | Change from Baseline in ItchRO(Pt) Frequency Score MMRM Model Effects |
| 14.2.4.20.1 | ITT | Change from Baseline in Clinician Scratch Scale (CSS) Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.20.2 | ITT | Change from Baseline in Clinician Scratch Scale (CSS) MMRM Model Effects |
| 14.2.4.21.1 | ITT | Change from Baseline in Caregiver Impression of Severity (CIS) Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.21.2 | ITT | Change from Baseline in Caregiver Impression of Severity (CIS) MMRM Model Effects |
| 14.2.4.22.1 | ITT | Change from Baseline in Patient Impression of Severity (PIS) Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.22.2 | ITT | Change from Baseline in Patient Impression of Severity (PIS) MMRM Model Effects |
| 14.2.4.23.1.1 | ITT – Primary<br>Cohort | Change from Baseline in EDQ(Obs) Severity Score Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.23.1.2 | ITT – Primary<br>Cohort | Change from Baseline in EDQ(Obs) Severity Score<br>MMRM Model Effects |
| 14.2.4.23.2.1 | ITT – PFIC Cohort | Change from Baseline in EDQ(Obs) Severity Score Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.23.2.2 | ITT – PFIC Cohort | Change from Baseline in EDQ(Obs) Severity Score<br>MMRM Model Effects |
| 14.2.4.24.1 | ITT | Change from Baseline in Morning EDQ(Obs) Sleep Disturbance Score<br>Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.24.2 | ITT | Change from Baseline in Morning EDQ(Obs) Sleep Disturbance Score<br>MMRM Model Effects |
| 14.2.4.25 | ITT | Number and Proportion of Subjects with Improvement from Baseline in<br>Morning EDQ(Obs) Sleep Disturbance Score |
| 14.2.4.26 | ITT | Number and Proportion of Subjects with Morning EDQ(Obs) Sleep Disturbance Scores ≤2 from Post-Baseline through Week 26 |
| 14.2.4.27.1 | ITT | Change from Baseline in PedsQL Total Scale Score Tabulation of Fitted Summary Statistics from MMRM |



| Number | Population | Title |
|---|---|---|
| 14.2.4.27.2 | ITT | Change from Baseline in PedsQL Total Scale Score MMRM Model Effects |
| 14.2.4.28.1 | ITT | Change from Baseline in Height z-Score Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.28.2 | ITT | Change from Baseline in Height z-Score MMRM Model Effects |
| 14.2.4.29.1 | ITT | Change from Baseline in Weight z-Score Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.29.2 | ITT | Change from Baseline in Weight z-Score MMRM Model Effects |
| 14.2.4.30.1 | ITT | Percent Change from Baseline in Total sBA Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.30.2 | ITT | Percent Change from Baseline in Total sBA MMRM Model Effects |
| 14.2.4.31.1 | ITT | Change from Baseline in 7 Alpha-hydroxy-4-cholesten-3-one (C4), ng/mL Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.31.2 | ITT | Change from Baseline in 7 Alpha-hydroxy-4-cholesten-3-one (C4), ng/mL MMRM Model Effects |
| 14.2.4.32.1 | ITT | Change from Baseline in Fibroblast Growth Factor 19 (pg/mL) Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.32.2 | ITT | Change from Baseline in Fibroblast Growth Factor 19 (pg/mL) MMRM Model Effects |
| 14.2.4.33.1 | ITT | Change from Baseline in Autotaxin (ng/mL) Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.33.2 | ITT | Change from Baseline in Autotaxin (ng/mL) MMRM Model Effects |
| 14.2.4.34.1 | ITT | Change from Baseline in Albumin (g/dL) Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.34.2 | ITT | Change from Baseline in Albumin (g/dL) MMRM Model Effects |
| 14.2.4.35 | ITT | Time to First Liver-Associated Event (Days) |



# 13.1.3. Safety Data

Table 5: Safety Data Summary Tables

| Number | Population | Title |
|---|---|---|
| 14.3.1 Study Drug E | xposure | |
| 14.3.1 | Safety | Maralixibat Exposure |
| 14.3.2 Displays of Ac | lverse Events | |
| 14.3.2.1.1 | Safety | Overall Summary of Treatment-Emergent Adverse Events |
| 14.3.2.1.2 | Safety | Overall Summary of Treatment-Emergent Adverse Events by Age<br>Group |
| 14.3.2.1.3 | Safety | Overall Summary of Treatment-Emergent Adverse Events by Sex |
| 14.3.2.1.4 | Safety | Overall Summary of Treatment-Emergent Adverse Events by Race |
| 14.3.2.2.1 | Safety | Incidence of Treatment-Emergent Adverse Events |
| 14.3.2.2.2 | Safety | Incidence of Treatment-Emergent Adverse Events by Age Group |
| 14.3.2.2.3 | Safety | Incidence of Treatment-Emergent Adverse Events by Sex |
| 14.3.2.2.4 | Safety | Incidence of Treatment-Emergent Adverse Events by Race |
| 14.3.3 Summary of I | Deaths, Other Seri | ous and Significant Adverse Events |
| 14.3.3.1 | Safety | Incidence of Treatment-Emergent Serious Adverse Events |
| 14.3.3.2 | Safety | Incidence of Treatment Related Adverse Events |
| 14.3.3.3 | Safety | Incidence of Treatment Related Adverse Events Leading to Permanent Discontinuation of Study Drug |
| 14.3.3.4.1 | Safety | Incidence of Events of Clinical Interest – Diarrhoea Events |
| 14.3.3.4.2 | Safety | Incidence of Events of Clinical Interest – LSV Deficiency Events |
| 14.3.3.4.3 | Safety | Incidence of Events of Clinical Interest – Elevated Transaminases |
| 14.3.3.4.4 | Safety | Incidence of Events of Clinical Interest – Elevated Bilirubin |
| 14.3.4 Narratives of | 14.3.4 Narratives of Deaths, Other Serious and Certain Other Significant Adverse Events | |
| 14.3.4.1 | Safety | Listing of Serious Adverse Events |
| 14.3.4.2 | Safety | Listing of Adverse Events Leading to Permanent Discontinuation of Study Drug |
| 14.3.4.3 | Safety | Listing of Deaths |



| Number | Population | Title |
|---|---|---|
| 14.3.5 Laboratory Da | ta Summary Tal | bles |
| 14.3.5.1 | Safety | Summary of Safety Laboratory Data: Chemistry |
| 14.3.5.2 | Safety | Summary of Safety Laboratory Data: Hematology |
| 14.3.5.3 | Safety | Summary of Safety Laboratory Data: Lipid Panel |
| 14.3.5.4 | Safety | Summary of Safety Laboratory Data: Lipid Soluble Vitamins (LSV) |
| 14.3.5.5 | Safety | Summary of Safety Laboratory Data: Alpha-Fetoprotein (ng/mL) |
| 14.3.5.6 | Safety | Shift Table for Select Safety Laboratory Tests |
| 14.3.6 Physical Exam | 14.3.6 Physical Examination, Vital Signs, and ECG Safety Data Summary Tables | |
| 14.3.6.1 | Safety | Summary of Subject Height, Weight, and BMI z-Scores |
| 14.3.6.2 | Safety | Summary of Vital Signs |
| 14.3.6.3.1 | Safety | Summary of Electrocardiogram Parameters |
| 14.3.6.3.2 | Safety | Summary of Electrocardiogram Interpretation |
| 14.3.7 Other Safety D | 14.3.7 Other Safety Data Summary Tables | |
| 14.3.7 | Safety | Summary of Concomitant Therapies/Medications |

### 13.1.4. Other Data

Table 6: Other Data Summary Tables

| Number | Population | Title |
|---|---|---|
| 14.4 Other Data Sum | mary Tables | |
| 14.4.1 | Safety | Summary of Healthcare Utilization Measures |
| 14.4.2 | Safety | Summary of Plasma Sample Maralixibat Concentrations (ng/mL) |





#### 13.2. Planned Figure Descriptions

The following are planned summary figures for protocol number MRX-502. The figure numbers are place holders only and will be determined when the figures are produced.

Estimates from the MMRM model (over time) will be graphically displayed for select efficacy variables in the ITT population for the primary and PFIC cohorts, separately. These plots will display the LS Mean ±SE for each treatment group at each analysis visit/time period, as appropriate. Each of the treatment group LS means will be displayed side-by-side, with vertical lines emanating from each LS Mean to represent the standard error. At minimum, these graphical displays will be presented for the change from baseline in morning ItchRO(Obs) severity score and change from baseline in sBA levels, over time. The number of subjects with non-missing change from baseline values, for each treatment group and analysis visit, will be displayed along the horizontal axis at each time point, baseline through Week 26.

Tipping point results, for the sensitivity analysis of the primary efficacy endpoint and the key secondary efficacy endpoint, will be presented in a heatmap. This figure will be generated to display p-values corresponding to all combinations of shifts from the imputed data. For the heatmap figure, each cell will be colored according to the p-value: green for p-values < 0.05; yellow for p-values of 0.05 to < 0.10; orange for p-values of 0.10 to < 0.20; and red for p-values of 0.20 to 1.00.

Additional figures may be added post-hoc to further examine study data.

#### 13.2.1. Efficacy Data

Table 7: Efficacy Data Summary Figures

| Number | Population | Title |
|---|---|---|
| 14.2.1.x Primary | Analysis | |
| 14.2.1.1 | ITT – Primary<br>Cohort | Plot of MMRM LS Mean (± SE) Change from Baseline in Morning ItchRO(Obs) Severity Score Over Time |
| 14.2.2.x Secondary Analysis | | |
| 14.2.2.2.1 | ITT – Primary<br>Cohort | Plot of MMRM LS Mean (± SE) Change from Baseline in Total sBA (μmol/L) Over Time |
| 14.2.3.x Sensitivity Analysis | | |
| 14.2.3.3 | ITT – Primary<br>Cohort | Heatmap Displaying p-values from Tipping Point Analysis on Change from Baseline in Morning ItchRO(Obs) Severity Score to Average of Last 12 Weeks |



| Number | Population | Title |
|---|---|---|
| 14.2.3.6 | ITT – Primary<br>Cohort | Heatmap Displaying p-values from Tipping Point Analysis on Change from Baseline in Total sBA (μmol/L) to Average of Weeks 18, 22, and 26 |

#### 13.3. Planned Listing Descriptions

In general, listings produced will include the participant data collected on associated CRF pages. All listings will be sorted by treatment, PFIC type, and subject ID. For safety data (i.e., study drug exposure, AEs, vital signs, laboratory tests, ECG, physical examination, and plasma maralixibat concentration levels), listings will be presented by treatment received. For all other listings (including efficacy laboratory tests), where applicable, data will be presented by randomized treatment group.

For listings of efficacy variables, change from baseline values will be included, as appropriate.

For adverse event listings, study day relative to the date of first dose of study drug will be provided along with stop and start dates. The dose of study drug at the onset of AEs in the maralixibat treatment group will also be provided. For partial event dates, study day will be derived using an imputed date as described in Section 6.1.9.

Study day relative to the first dose of study drug will also be included on laboratory listings, along with laboratory collection dates, and on study drug exposure listings, along with start and stop dates.

For the concomitant treatment listing, medications that are ongoing at the time of informed consent will be indicated.

Weight, height, and BMI will be presented in the vital signs listing, rather than the physical examination listing.

PedsQL listings will present total scale and summary scores, including PedsQL Total Scale Score, Physical Health Summary Score, Psychosocial Health Summary Score, Multidimensional Fatigue Scale Score, Family Impact Total Scale Score, Parent Functioning Summary Score, and Family Impact Summary Score. Subject listings of PedsQL raw scores for each of the model items will not be included.

Assessments denoted as clinic visit "Week 26/ET" in listings will include assessments performed at the Early Termination visit for participants who withdraw early from the study.





In all listings a blank line will be placed between participants. Within a data listing, if an item appears line after line (e.g., repetition of participant number), then only the first occurrence will be displayed.

The listing shells will be provided under a separate document.

#### 13.4. Standard Layout for all Tables, Listings, and Figures

The following standard layout will be applied to all Tables, Listings, and Figures (TLFs) in support of this study. Note that programming notes may be added if appropriate after each TLF shell.





## Figure 2. Standardized Layout

| Mirum Pharmaceuticals Inc. Protocol: MRX-502 | Page xx of xx<br>Version xxxxx |
|---|---|
| <table, figure="" listing,=""> xx.x.x</table,> | |
| <title figure="" listing="" of="" or="" table="">&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;Study Population and if applicable subgroup Description&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;Body of Table, Listing or Figure&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;a href="#"&gt;&lt;Abbreviations: If applicable&gt;&lt;/a&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;Note: If applicable&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;Footnote 1 &lt;if applicable&gt; Recommendation is to keep footnotes to a minimum Footnote 2 &lt;if applicable&gt; Footnote n &lt;if applicable&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;pre&gt;&lt;pgm path and name&gt; &lt;Executed on &lt;date&gt; at &lt;time&gt; on data from &lt;data cut date&gt;&lt;/pre&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;/tbody&gt;&lt;/table&gt;</title> | |



# **Appendix 1: Listing of Safety and Efficacy Laboratory Analytes**

| SAFETY LABS | | | |
|---|---|---|---|
| <b>Hematology</b> | <b>Clinical Chemistry</b> | Lipid Panel | <u>Urinalysis</u> [1] |
| Erythrocytes (RBC), 10 <sup>6</sup> /µL Hemoglobin, g/dL Hematocrit, % MCV, fL MCH, pg MCHC, g/dL Platelets, 10 <sup>3</sup> /µL Leukocytes (WBC), 10 <sup>3</sup> /µL Differential (% and 10 <sup>3</sup> /µL) • Neutrophils • Eosinophils • Basophils • Lymphocytes • Monocytes | Sodium, mEq/L Potassium, mEq/L Chloride, mEq/L Bicarbonate, mEq/L Protein, g/dL Calcium, mg/dL Phosphate, mg/dL Glucose, mg/dL Lipase, U/L BUN, mg/dL Creatinine, mg/dL Urate, mg/dL Corrected Sodium, mEq/L [3] Amylase, U/L Measured Osmolality, mOsm/kg Calculated Osmolality, mOsm/kg [3] Osmolar Gap, mOsm/kg [3] Anion Gap, mEq/L [3] | Triglycerides, mg/dL Cholesterol, mg/dL LDL-C, mg/dL HDL-C, mg/dL [1] Lipid Soluble Vitamins 25-Hydroxy Vitamin D, ng/mL Vitamin A (retinol), µg/dL Retinol Binding Protein (RBP), mg/dL Alpha Tocopherol, mg/dL INR (surrogate marker for Vitamin K deficiency) Retinol: RBP Molar Ratio, mol/mol [3] Ratio of Alpha Tocopherol to the sum of Cholesterol and Triglycerides, mg/g [3] aPTT, sec (surrogate for LSV) PT, sec (surrogate for LSV) Marker of hepatocellular carcinoma Alpha-Fetoprotein (AFP), ng/mL | pH Specific Gravity Renal Epithelial Cells, /HPF Squamous Epithelial Cells, /HPF Granular Casts, /LPF Hyaline Casts, /LPF RBC Casts, /LPF Erythrocytes, /HPF Leukocytes, /HPF WBC Casts, /LPF Waxy Casts, /LPF Protein * Glucose * Ketones * Bilirubin * Nitrite * Urobilinogen * Leukocyte Esterase * Calcium Oxalate Crystals * Triple Phosphate Crystals * Uric Acid Crystals * Bacteria * Creatinine * Transitional Epithelial Cells * Occult Blood * Yeast Cells * |





#### EFFICACY LABS

#### **Clinical Chemistry**

Total Bilirubin, mg/dL [2] Direct Bilirubin (conjugated), mg/dL [2] ALT, U/L [2] AST, U/L [2] ALP, U/L [2] GGT, U/L [2] Albumin, g/dL [2] APRI [3] FIB-4 [3] PELD [3]

#### **Cholestasis Biomarkers**

Serum Bile Acids, µmol/L [2]
7 alpha-hydroxy-4-cholesten-3-one (C4), ng/mL
Autotaxin, ng/mL
FGF-19, pg/mL [2]
Bile Acid Subspecies, µmol/L
(15 subspecies) [1]

Abbreviations: ALP = alkaline phosphatase; ALT = alanine aminotransferase; aPTT = activated partial thromboplastin time; APRI = AST to platelet ratio index; AST = aspartate aminotransferase; FGF-19 = fibroblast growth factor 19; FIB-4 = fibrosis-4; GGT = gamma-glutamyl transferase; PT = prothrombin time; MCH = mean corpuscular hemoglobin; MCHC = mean corpuscular hemoglobin concentration; MCV = mean corpuscular volume; MELD = model for end-stage liver disease; PELD = pediatric end-stage liver disease; WBC = white blood cell; \* Qualitative urinalysis

[1] Listing only

MELD [3]

- [2] Safety and efficacy lab tests
- [3] Calculated lab parameters (see Sec 6.1.8);





# **Appendix 2: Listing of Lipid Soluble Vitamin Deficiency Events**

The following MedDRA Preferred Terms associated with lipid soluble vitamin (LSV) deficiency events are included as an AECI:

- Vitamin A deficiency
- Vitamin A abnormal
- Vitamin A decreased
- Vitamin D deficiency
- Vitamin D abnormal
- Vitamin D decreased
- Vitamin E deficiency
- Vitamin E decreased
- Vitamin K deficiency
- Vitamin K decreased
- International normalised ratio increased
- International normalised ratio abnormal
- Blood 1,25-dihydroxycholecalciferol decreased
- Blood 25-hydroxycholecalciferol decreased

Sponsor: Mirum Pharmaceuticals Inc. Protocol: Maralixibat-502 (Amendment 4) PCN Number: MIRU8967



| Sponsor | Mirum Pharmaceuticals Inc. |
|---|---|
| Protocol Title: | Randomized Double-blind Placebo-controlled Phase 3 Study to Evaluate the Efficacy and Safety of Maralixibat in the Treatment of Children with Progressive Familial Intrahepatic Cholestasis (PFIC) – MARCH-PFIC |
| Protocol Number: | MRX-502 (Amendment 4) |
| Premier Research PCN: | MIRU8967 |
| Document Author: | Jana Steinmetz |
| Document Version: | Final 1.0 |
| Document Date: | 09Oct2022 |

Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



#### **Table Conventions, Titles, and Shells** 1.

All tables will have a page header showing the sponsor company name (Mirum Pharmaceuticals Inc.) and protocol (MRX-502), and a page footer showing the file name and path, and the date/time of program execution along with the database data cut date.

The following reporting conventions will be adopted for the presentation of study data. These conventions will enhance the review process and help to standardize the presentation with common notations.

#### **General Reporting Conventions**

- All tables will be developed in landscape orientation.
- Abbreviations, general note, specific item footnotes, and source of data (as applicable), in this order, will be presented on each page of a table.
- In general, specialized text styles, such as bolding, italics, borders, shading, and superscripted and subscripted text will not be used in tables unless they add significant value.
- Only standard keyboard characters will be used in the tables. Special characters, such as nonprintable control characters, printer-specific characters, or font specific characters, will not be used.
- Adverse events with missing MedDRA coding will have their system organ class and/or preferred term presented as "Not Coded". The "Not Coded" frequencies will be sorted to the end of the tables. Adverse events that are not coded are not expected.
- Programming notes may be inserted into the shells, these notes will not appear in the final output.

#### **Population Summary Conventions**

- Population sizes may be presented for each cohort, treatment group, subgroup, and classification factor, where appropriate, as totals in the column header as (N=xxx).
- All population summaries for categorical variables will include all categories that were planned and for which the subjects may have had a response. Percentages corresponding to null categories (cells) will be suppressed; however, counts and percentages of missing values may be needed. Counts of zero will be presented as '0', without the percentage.
- In general, population summaries for continuous variables will include: n, mean, SD, SE, median, Q1, Q3, minimum, and maximum. Other summaries (e.g., number missing, geometric mean, 95% CIs, and coefficient of variation [CV] or % CV) may be used as appropriate. The precision of the maximum and minimum will match the maximum precision in the data. The mean, median, Q1, and Q3 will have 1 additional decimal place. The SD will have 2 additional decimal places.
- All percentages are rounded and reported to a single decimal point (xx.x%).

CONFIDENTIAL. 

Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



#### 1.1. **Planned Table Descriptions**

The following are planned summary tables for protocol number MRX-502. The table numbers are place holders only and will be determined when the tables are produced. The efficacy outputs are ordered to account for the hierarchical testing structure as outlined in the SAP, where possible. For cases where multiple subject cohorts or, in the case of ItchRO and EDQ morning, evening, and highest daily scores are presented, data columns are consolidated on a single table, when practical, for ease of review and referencing results.

### 1.1.1. Subject Data

Table 1: Subject Data Summary Tables

| Number | Population | Title |
|---|---|---|
| 14.1.1.1 | All Subjects | Subject Disposition |
| 14.1.1.2 | Safety | Number of Randomized and Completed Subjects by Country |
| 14.1.1.3 | Safety | Number of Randomized and Completed Subjects by<br>Investigative Site |
| 14.1.2 | Safety | Important Protocol Violations/Deviations |
| 14.1.3 | Safety | Demographics and Baseline Characteristics |
| 14.1.4 | Safety | Disease History and Baseline Disease Characteristics |
| 14.1.5 | Safety | Prior Medications/Therapies |
| 14.1.6 | Safety | Study Drug Compliance |

#### 1.1.2. Efficacy Data

Table 2: Efficacy Data Summary Tables

| Number | Population | Title |
|---|---|---|
| 14.2.1.x Primar | 14.2.1.x Primary Analysis | |
| 14.2.1.1 | ITT – Primary<br>Cohort | Change from Baseline in ItchRO(Obs) Severity Score Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.1.2 | ITT – Primary<br>Cohort | Change from Baseline in ItchRO(Obs) Severity Score<br>MMRM Model Effects |
| 14.2.2.x Secondary Analysis | | |
| 14.2.2.1.1 | ITT – PFIC<br>Cohort | Change from Baseline in ItchRO(Obs) Severity Score Tabulation of Fitted Summary Statistics from MMRM |


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4) PCN Number: MIRU8967



| Number | Population | Title |
|---|---|---|
| 14.2.2.1.2 | ITT – PFIC<br>Cohort | Change from Baseline in ItchRO(Obs) Severity Score<br>MMRM Model Effects |
| 14.2.2.2.1 | ITT | Change from Baseline in Total sBA (µmol/L) Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.2.2.2 | ITT | Change from Baseline in Total sBA (µmol/L) MMRM Model Effects |
| 14.2.2.3 | ITT | Proportion of Responders |
| 14.2.3.x Sensitiv | vity Analysis | |
| 14.2.3.1.1 | ITT | Change from Baseline in Morning ItchRO(Obs) Severity Score – Sibling Sensitivity Analysis |
| | | Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.3.1.2 | ITT | Change from Baseline in Morning ItchRO(Obs) Severity Score – Sibling Sensitivity Analysis MMRM Model Effects |
| 14.2.3.2 | ITT | Change from Baseline in Morning ItchRO(Obs) Severity Score – Multiple Imputation Sensitivity Analysis |
| | | Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.3.3 | ITT | Change from Baseline in Morning ItchRO(Obs) Severity Score to Average of Last 12 Weeks – Tipping Point Sensitivity Analysis |
| 14.2.3.4.1 | ITT | Change from Baseline in Total sBA (µmol/L) – Sibling Sensitivity Analysis Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.3.4.2 | ITT | Change from Baseline in Total sBA (µmol/L) – Sibling Sensitivity Analysis MMRM Model Effects |
| 14.2.3.5 | ITT | Change from Baseline in Total sBA (µmol/L) – Multiple Imputation Sensitivity Analysis Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.3.6 | ITT | Change from Baseline in Total sBA (µmol/L) to Average of Weeks 18, 22, and 26 – Tipping Point Sensitivity Analysis |


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4) PCN Number: MIRU8967



| Number | Population | Title |
|---|---|---|
| 14.2.4.x Explor | 14.2.4.x Exploratory Analysis | |
| 14.2.4.1.1 | PP – Primary<br>Cohort | Change from Baseline in Morning ItchRO(Obs) Severity Score Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.1.2 | PP – Primary<br>Cohort | Change from Baseline in Morning ItchRO(Obs) Severity Score<br>MMRM Model Effects |
| 14.2.4.2.1 | PP – Primary<br>Cohort | Change from Baseline in Total sBA (µmol/L) Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.2.2 | PP – Primary<br>Cohort | Change from Baseline in Total sBA (µmol/L) MMRM Model Effects |
| 14.2.4.3.1 | ITT – Primary<br>Cohort | Change from Baseline in Weekly Average Morning ItchRO(Obs) Severity Score Descriptive Statistics by Analysis Week |
| 14.2.4.3.2 | ITT – Primary<br>Cohort | Change from Baseline in Weekly Average Morning ItchRO(Obs) Severity Score by Region Descriptive Statistics by Analysis Week |
| 14.2.4.3.3 | ITT – Primary<br>Cohort | Change from Baseline in Weekly Average Morning ItchRO(Obs) Severity Score by Age at Baseline Descriptive Statistics by Analysis Week |
| 14.2.4.3.4 | ITT – Primary<br>Cohort | Change from Baseline in Weekly Average Morning ItchRO(Obs) Severity Score by Sex Descriptive Statistics by Analysis Week |
| 14.2.4.3.5 | ITT – Primary<br>Cohort | Change from Baseline in Weekly Average Morning ItchRO(Obs) Severity Score by Race Descriptive Statistics by Analysis Week |
| 14.2.4.3.6 | ITT – Primary<br>Cohort | Change from Baseline in Weekly Average Morning ItchRO(Obs) Severity Score by Baseline Median sBA Descriptive Statistics by Analysis Week |
| 14.2.4.3.7 | ITT – Primary<br>Cohort | Change from Baseline in Weekly Average Morning ItchRO(Obs) Severity Score by Baseline UDCA Usage Descriptive Statistics by Analysis Week |


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4) PCN Number: MIRU8967



| Number | Population | Title |
|---|---|---|
| 14.2.4.3.8 | ITT – Primary<br>Cohort | Change from Baseline in Weekly Average Morning ItchRO(Obs) Severity Score by Baseline Rifampicin Usage Descriptive Statistics by Analysis Week |
| 14.2.4.3.9 | ITT – Primary<br>Cohort | Change from Baseline in Weekly Average Morning ItchRO(Obs) Severity Score by BSEP Type Descriptive Statistics by Analysis Week |
| 14.2.4.4.1 | ITT – Primary<br>Cohort | Change from Baseline in Total sBA (µmol/L) Descriptive Statistics by Analysis Week |
| 14.2.4.4.2 | ITT – Primary<br>Cohort | Change from Baseline in Total sBA (µmol/L) by Region Descriptive Statistics by Analysis Week |
| 14.2.4.4.3 | ITT – Primary<br>Cohort | Change from Baseline in Total sBA (µmol/L) by Age at Baseline<br>Descriptive Statistics by Analysis Week |
| 14.2.4.4.4 | ITT – Primary<br>Cohort | Change from Baseline in Total sBA (µmol/L) by Sex<br>Descriptive Statistics by Analysis Week |
| 14.2.4.4.5 | ITT – Primary<br>Cohort | Change from Baseline in Total sBA (µmol/L) by Race<br>Descriptive Statistics by Analysis Week |
| 14.2.4.4.6 | ITT – Primary<br>Cohort | Change from Baseline in Total sBA (µmol/L) by Baseline<br>Median sBA<br>Descriptive Statistics by Analysis Week |
| 14.2.4.4.7 | ITT – Primary<br>Cohort | Change from Baseline in Total sBA (µmol/L) by Baseline UDCA Usage Descriptive Statistics by Analysis Week |
| 14.2.4.4.8 | ITT – Primary<br>Cohort | Change from Baseline in Total sBA (µmol/L) by Baseline<br>Rifampicin Usage<br>Descriptive Statistics by Analysis Week |
| 14.2.4.4.9 | ITT – Primary<br>Cohort | Change from Baseline in Total sBA (µmol/L) by BSEP Type<br>Descriptive Statistics by Analysis Week |
| 14.2.4.5.1 | ITT | Change from Baseline in ALT (U/L) Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.5.2 | ITT | Change from Baseline in ALT (U/L) MMRM Model Effects |


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4) PCN Number: MIRU8967



| Number | Population | Title |
|---|---|---|
| 14.2.4.6.1 | ITT | Change from Baseline in AST (U/L) Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.6.2 | ITT | Change from Baseline in AST (U/L) MMRM Model Effects |
| 14.2.4.7.1 | ITT | Change from Baseline in Total Bilirubin (mg/dL) Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.7.2 | ITT | Change from Baseline in Total Bilirubin (mg/dL) MMRM Model Effects |
| 14.2.4.8.1 | ITT | Change from Baseline in Direct Bilirubin (mg/dL) Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.8.2 | ITT | Change from Baseline in Direct Bilirubin (mg/dL) MMRM Model Effects |
| 14.2.4.9.1 | ITT | Change from Baseline in ALP (U/L) Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.9.2 | ITT | Change from Baseline in ALP (U/L) MMRM Model Effects |
| 14.2.4.10.1 | ITT | Change from Baseline in GGT (U/L) Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.10.2 | ITT | Change from Baseline in GGT (U/L) MMRM Model Effects |
| 14.2.4.11.1 | ITT | Change from Baseline in FIB-4 Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.11.2 | ITT | Change from Baseline in FIB-4 MMRM Model Effects |
| 14.2.4.12.1 | ITT | Change from Baseline in APRI Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.12.2 | ITT | Change from Baseline in APRI<br>MMRM Model Effects |
| 14.2.4.13.1 | ITT | Change from Baseline in PELD Tabulation of Fitted Summary Statistics from MMRM |


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4) PCN Number: MIRU8967



| Number | Population | Title |
|---|---|---|
| 14.2.4.13.2 | ITT | Change from Baseline in PELD MMRM Model Effects |
| 14.2.4.14 | ITT | Total sBA Shift from Baseline: Number and Proportion of Subjects |
| 14.2.4.15 | ITT | Number of Days Morning ItchRO(Obs) Severity Score ≤1<br>Over the Last 84 Study Days |
| 14.2.4.16 | ITT | Number and Proportion of Subjects with Morning ItchRO(Obs) Severity Score ≤1 for >50% of Time Period |
| 14.2.4.17.1.1 | ITT – Primary<br>Cohort | Change from Baseline in ItchRO(Obs) Frequency Score Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.17.1.2 | ITT – Primary<br>Cohort | Change from Baseline in ItchRO(Obs) Frequency Score MMRM Model Effects |
| 14.2.4.17.2.1 | ITT – PFIC<br>Cohort | Change from Baseline in ItchRO(Obs) Frequency Score Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.17.2.2 | ITT – PFIC<br>Cohort | Change from Baseline in ItchRO(Obs) Frequency Score MMRM Model Effects |
| 14.2.4.18.1.1 | ITT – Primary<br>Cohort | Change from Baseline in ItchRO(Pt) Severity Score Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.18.1.2 | ITT – Primary<br>Cohort | Change from Baseline in ItchRO(Pt) Severity Score MMRM Model Effects |
| 14.2.4.18.2.1 | ITT – PFIC<br>Cohort | Change from Baseline in ItchRO(Pt) Severity Score Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.18.2.2 | ITT – PFIC<br>Cohort | Change from Baseline in ItchRO(Pt) Severity Score MMRM Model Effects |
| 14.2.4.19.1.1 | ITT – Primary<br>Cohort | Change from Baseline in ItchRO(Pt) Frequency Score Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.19.1.2 | ITT – Primary<br>Cohort | Change from Baseline in ItchRO(Pt) Frequency Score MMRM Model Effects |
| 14.2.4.19.2.1 | ITT – PFIC<br>Cohort | Change from Baseline in ItchRO(Pt) Frequency Score Tabulation of Fitted Summary Statistics from MMRM |


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4) PCN Number: MIRU8967



| Number | Population | Title |
|---|---|---|
| 14.2.4.19.2.2 | ITT – PFIC<br>Cohort | Change from Baseline in ItchRO(Pt) Frequency Score<br>MMRM Model Effects |
| 14.2.4.20.1 | ITT | Change from Baseline in Clinician Scratch Scale (CSS) Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.20.2 | ITT | Change from Baseline in Clinician Scratch Scale (CSS) MMRM Model Effects |
| 14.2.4.21.1 | ITT | Change from Baseline in Caregiver Impression of Severity (CIS) Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.21.2 | ITT | Change from Baseline in Caregiver Impression of Severity (CIS) MMRM Model Effects |
| 14.2.4.22.1 | ITT | Change from Baseline in Patient Impression of Severity (PIS) Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.22.2 | ITT | Change from Baseline in Patient Impression of Severity (PIS) MMRM Model Effects |
| 14.2.4.23.1.1 | ITT – Primary<br>Cohort | Change from Baseline in EDQ(Obs) Severity Score Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.23.1.2 | ITT – Primary<br>Cohort | Change from Baseline in EDQ(Obs) Severity Score<br>MMRM Model Effects |
| 14.2.4.23.2.1 | ITT – PFIC<br>Cohort | Change from Baseline in EDQ(Obs) Severity Score Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.23.2.2 | ITT – PFIC<br>Cohort | Change from Baseline in EDQ(Obs) Severity Score MMRM Model Effects |
| 14.2.4.24.1 | ITT | Change from Baseline in Morning EDQ(Obs) Sleep Disturbance<br>Score<br>Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.24.2 | ITT | Change from Baseline in Morning EDQ(Obs) Sleep Disturbance<br>Score<br>MMRM Model Effects |
| 14.2.4.25 | ITT | Number and Proportion of Subjects with Improvement from Baseline in Morning EDQ(Obs) Sleep Disturbance Score |


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4) PCN Number: MIRU8967



Number **Population** Title Number and Proportion of Subjects with Morning EDQ(Obs) 14.2.4.26 ITT Sleep Disturbance Scores ≤2 from Post-Baseline through Week 26 Change from Baseline in PedsQL Total Scale Score 14.2.4.27.1 ITT Tabulation of Fitted Summary Statistics from MMRM Change from Baseline in PedsQL Total Scale Score 14.2.4.27.2 ITT MMRM Model Effects Change from Baseline in Height z-Score 14.2.4.28.1 ITT Tabulation of Fitted Summary Statistics from MMRM Change from Baseline in Height z-Score 14.2.4.28.2 ITT MMRM Model Effects Change from Baseline in Weight z-Score 14.2.4.29.1 ITT Tabulation of Fitted Summary Statistics from MMRM Change from Baseline in Weight z-Score 14.2.4.29.2 ITT MMRM Model Effects Percent Change from Baseline in Total sBA 14.2.4.30.1 ITT Tabulation of Fitted Summary Statistics from MMRM Percent Change from Baseline in Total sBA 14.2.4.30.2 ITT MMRM Model Effects Change from Baseline in 7 Alpha-hydroxy-4-cholesten-3-one 14.2.4.31.1 ITT (C4), ng/mLTabulation of Fitted Summary Statistics from MMRM Change from Baseline in 7 Alpha-hydroxy-4-cholesten-3-one (C4), ng/mL14.2.4.31.2 ITT MMRM Model Effects Change from Baseline in Fibroblast Growth Factor 19 (pg/mL) 14.2.4.32.1 ITT Tabulation of Fitted Summary Statistics from MMRM Change from Baseline in Fibroblast Growth Factor 19 (pg/mL) 14.2.4.32.2 ITT MMRM Model Effects Change from Baseline in Autotaxin (ng/mL) 14.2.4.33.1 ITT Tabulation of Fitted Summary Statistics from MMRM


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4) PCN Number: MIRU8967



| Number | Population | Title |
|---|---|---|
| 14.2.4.33.2 | ITT | Change from Baseline in Autotaxin (ng/mL) MMRM Model Effects |
| 14.2.4.34.1 | ITT | Change from Baseline in Albumin (g/dL) Tabulation of Fitted Summary Statistics from MMRM |
| 14.2.4.34.2 | ITT | Change from Baseline in Albumin (g/dL) MMRM Model Effects |
| 14.2.4.35 | ITT | Time to First Liver-Associated Event (Days) |

# 1.1.3. Safety Data

Table 3: Safety Data Summary Tables

| Number | Population | Title |
|---|---|---|
| 14.3.1 Study | 14.3.1 Study Drug Exposure | |
| 14.3.1 | Safety | Maralixibat Exposure |
| 14.3.2 Displa | ys of Adverse | Events |
| 14.3.2.1.1 | Safety | Overall Summary of Treatment-Emergent Adverse Events |
| 14.3.2.1.2 | Safety | Overall Summary of Treatment-Emergent Adverse Events by Age<br>Group |
| 14.3.2.1.3 | Safety | Overall Summary of Treatment-Emergent Adverse Events by Sex |
| 14.3.2.1.4 | Safety | Overall Summary of Treatment-Emergent Adverse Events by Race |
| 14.3.2.2.1 | Safety | Incidence of Treatment-Emergent Adverse Events |
| 14.3.2.2.2 | Safety | Incidence of Treatment-Emergent Adverse Events by Age Group |
| 14.3.2.2.3 | Safety | Incidence of Treatment-Emergent Adverse Events by Sex |
| 14.3.2.2.4 | Safety | Incidence of Treatment-Emergent Adverse Events by Race |
| 14.3.3 Summ | ary of Death | s, Other Serious and Significant Adverse Events |
| 14.3.3.1 | Safety | Incidence of Treatment-Emergent Serious Adverse Events |
| 14.3.3.2 | Safety | Incidence of Treatment Related Adverse Events |
| 14.3.3.3 | Safety | Incidence of Treatment Related Adverse Events Leading to<br>Permanent Discontinuation of Study Drug |
| 14.3.3.4.1 | Safety | Incidence of Events of Clinical Interest – Diarrhoea Events |
| 14.3.3.4.2 | Safety | Incidence of Events of Clinical Interest – LSV Deficiency Events |


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



| Number | Population | Title |
|---|---|---|
| 14.3.3.4.3 | Safety | Incidence of Events of Clinical Interest – Elevated Transaminases |
| 14.3.3.4.4 | Safety | Incidence of Events of Clinical Interest – Elevated Bilirubin |
| 14.3.4 Narra | 14.3.4 Narratives of Deaths, Other Serious and Certain Other Significant Adverse Events | |
| 14.3.4.1 | Safety | Listing of Serious Adverse Events |
| 14.3.4.2 | Safety | Listing of Adverse Events Leading to Permanent Discontinuation of Study Drug |
| 14.3.4.3 | Safety | Listing of Deaths |
| 14.3.5 Labor | atory Data Si | ummary Tables |
| 14.3.5.1 | Safety | Summary of Safety Laboratory Data: Chemistry |
| 14.3.5.2 | Safety | Summary of Safety Laboratory Data: Hematology |
| 14.3.5.3 | Safety | Summary of Safety Laboratory Data: Lipid Panel |
| 14.3.5.4 | Safety | Summary of Safety Laboratory Data: Lipid Soluble Vitamins (LSV) |
| 14.3.5.5 | Safety | Summary of Safety Laboratory Data: Alpha-Fetoprotein (ng/mL) |
| 14.3.5.6 | Safety | Shift Table for Select Safety Laboratory Tests |
| 14.3.6 Physic | al Examinati | on, Vital Signs, and ECG Safety Data Summary Tables |
| 14.3.6.1 | Safety | Summary of Subject Height, Weight, and BMI z-Scores |
| 14.3.6.2 | Safety | Summary of Vital Signs |
| 14.3.6.3.1 | Safety | Summary of Electrocardiogram Parameters |
| 14.3.6.3.2 | Safety | Summary of Electrocardiogram Interpretation |
| 14.3.7 Other | Safety Data S | Summary Tables |
| 14.3.7 | Safety | Summary of Concomitant Therapies/Medications |

### 1.1.4. Other Data

Table 4: Other Data Summary Tables

| Number | Population | Title |
|---|---|---|
| 14.4 Other Data Summary Tables | | |
| 14.4.1 | Safety | Summary of Healthcare Utilization Measures |
| 14.4.2 | Safety | Summary of Plasma Sample Maralixibat Concentrations (ng/mL) |

CONFIDENTIALPage 12 of 99

Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4) PCN Number: MIRU8967



#### **Planned Table Shells** 1.2.


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



#### Table 14.1.1.1 Subject Disposition All Subjects

| Status or | Primary Cohort | | | | PFIC Cohort | | All Subjects | | |
|---|---|---|---|---|---|---|---|---|---|
| | Maralixibat | Placebo | Overall | Maralixibat | Placebo | Overall | Maralixibat | Placebo | Overall |
| Variable/Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | Placebo (N=xx) xx | (N=xx) |
| Screened for Eligibility | | | | | | | | | xx |
| Screen Failure | | | | | | | | | xx |
| Randomized [1] | XX | XX | XX | XX | xx | XX | xx | XX | XX |
| Families with Siblings enrolled | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| Total number of Siblings | XX | xx | XX | XX | XX | XX | xx | XX | xx |
| Safety Population [2] | xx | xx | XX | XX | xx | XX | xx | xx | xx |
| ITT Population [1, 3] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Per-Protocol Population [4] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Completed Study Treatment | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Discontinued Early [1] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Abbreviation: ITT = intent-to-treat; PEBD = partial external biliary diversion

Note: Percentages are based on the number of subjects in the Safety Population. Siblings (within the same family) are assigned in a blinded manner to the same treatment group.

- [1] One subject (Subject 023004) was randomized in error within the IRT system on 14Sep2020, the date of the baseline visit. This subject was not dispensed study drug, and was discontinued from the study due to 'administrative error' on the baseline visit day. On 15Oct2022, this same subject was re-randomized as Subject 023005. This subject is only counted once, as Subject 023005, in the Randomized and ITT Population groups, and not counted in the Discontinued Early group.
- [2] The Safety Population includes all subjects who receive at least 1 dose of study drug.
- [3] The ITT Population includes all randomized subjects.
- [4] The Per-Protocol population includes all subjects in the ITT Population who receive at least 1 dose of study drug and do not have any important protocol violations or deviations that have a potential impact on the efficacy analysis.

Source: Reference Listings xx.x.x, xx.x.x




Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4) PCN Number: MIRU8967



Table 14.1.1.1 (Cont'd) Subject Disposition All Subjects

| | Pr | imary Cohort | | | PFIC Cohort | | All Subjects | | |
|---|---|---|---|---|---|---|---|---|---|
| Status or | Maralixibat | Placebo | Overall | Maralixibat | Placebo | Overall | Maralixibat | Placebo | Overall |
| Variable/Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Reason for Discontinuation | | | | | | | | | |
| Adverse Event | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Death | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Lost to follow-up | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Non-compliance with study drug | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Lack of efficacy | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Physician decision | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Pregnancy | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Liver transplant | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| PEBD surgery | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Protocol violation | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Withdrawal of consent | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Study terminated by sponsor | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Disease Progression | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.1.1.2 Number of Randomized and Completed Subjects by Country Safety Population

| | Pr | Primary Cohort | | | PFIC Cohort | | All Subjects | | |
|---|---|---|---|---|---|---|---|---|---|
| Country | Maralixibat<br>(N=xx) | Placebo<br>(N=xx) | Overall<br>(N=xx) | Maralixibat<br>(N=xx) | Placebo<br>(N=xx) | Overall<br>(N=xx) | Maralixibat<br>(N=xx) | Placebo<br>(N=xx) | Overall<br>(N=xx) |
| xxxxxxxx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| xxxxxxx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| xxxxxx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| xxxxx xxxxxx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| xxxxxxx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Note: Percentages are 100\*n/N.

Source: Reference Listings xx.x.x, xx.x.x


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.1.1.3 Number of Randomized and Completed Subjects by Investigative Site Safety Population

Programming Notes: Repeat Table 14.1.1.2 with Investigative Site and change 1st column header to 'Investigative Site ID'.)




Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.1.2 Important Protocol Violations/Deviations Safety Population

| | Primary Cohort | | | | PFIC Cohort | | All Subjects | | |
|---|---|---|---|---|---|---|---|---|---|
| | Maralixibat | Placebo | Overall | Maralixibat | Placebo | Overall | Maralixibat | Placebo | Overall |
| Category/Type [1] | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Informed consent | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Inclusion | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Exclusion | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Study Drug | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Overdose/misuse | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Prohibited co-medication | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Assessment – efficacy | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Assessment – safety | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Laboratory/endpoint data | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Visit Window | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

etc...

Note: Percentages are 100\*n/N.

[1] Important protocol violations/deviations are grouped based on study specific protocol deviation categories as described in the Protocol Deviation Guidance Plan for the Maralixibat-502 clinical protocol. Subjects were counted only once for each category/type.

Source: Reference Listings xx.x.x, xx.x.x




Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.1.3 **Demographics and Baseline Characteristics** Safety Population

| | Р | rimary Cohort | | | PFIC Cohort | | | All Subjects | |
|---|---|---|---|---|---|---|---|---|---|
| Variable | Maralixibat | Placebo | Overall | Maralixibat | Placebo | Overall | Maralixibat | Placebo | Overall |
| Statistic or Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Age (years) [1] | | | | | | | | | |
| n | XX | xx | XX | XX | XX | XX | XX | xx | XX |
| Mean | xx.x | XX.X | xx.x | xx.x | xx.x | xx.x | xx.x | XX.X | xx.x |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | XX.X | XX.X |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | XX, XX | xx, xx | xx, xx | xx, xx | XX, XX | xx, xx | xx, xx | xx, xx |
| Age Category [1] | | | | | | | | | |
| 1 to <6 years | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 6 to <13 years | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 13 to 18 years | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Sex | | | | | | | | | |
| Male | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Female | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Abbreviations: SD = standard deviation; SE = standard error of the mean; Q1 = 25th percentile; Q3 = 75th percentile Note: Percentages are 100\*n/N.

[2] Height, weight, and BMI z-scores are based on a subject's sex and age at the baseline visit. The World Health Organization (WHO) grouth charts were used to derive z-scores for subjects less than 24 months old and the Center for Disease Control (CDC) grouth charts were used to derive z-scores for subjects equal to or greater than 24 months old. Source: Reference Listings xx.x.x, xx.x.x

Programming Note: If a particular category (e.g., race, ethnicity) is not reported, add a category for "Not reported". Subjects reporting more than 1 race will be counted in a "More than one race" category for purpose of tabulating summary statistics for race.


<sup>[1]</sup> Age at baseline visit.


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4) PCN Number: MIRU8967



# Table 14.1.3 (Cont'd) Demographics and Baseline Characteristics Safety Population

| | Pi | rimary Cohort | | | PFIC Cohort | | | All Subjects | |
|---|---|---|---|---|---|---|---|---|---|
| Variable | Maralixibat | Placebo | Overall | Maralixibat | Placebo | Overall | Maralixibat | Placebo | Overall |
| Statistic or Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Race | | | | | | | | | |
| American Indian or Alaska Native | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Asian | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Black or African American | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Native Hawaiian or Other Pacific Islander | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| White | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| More than one race | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Not Reported | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Ethnicity | | | | | | | | | |
| Hispanic or Latino | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Not Hispanic or Latino | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Not Reported | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Region | | | | | | | | | |
| Asia | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Europe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Middle East | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| North America | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| South and Central America | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |




Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4) PCN Number: MIRU8967 premier research

# Table 14.1.3 (Cont'd) Demographics and Baseline Characteristics Safety Population

| | Р | rimary Cohort | | | PFIC Cohort | | | All Subjects | |
|---|---|---|---|---|---|---|---|---|---|
| Variable | Maralixibat | Placebo | Overall | Maralixibat | Placebo | Overall | Maralixibat | Placebo | Overall |
| Statistic or Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Height (cm) | | | | | | | | | |
| n | XX | xx | xx | XX | xx | XX | XX | xx | xx |
| Mean | XX.X | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | XX.X | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | XX.X, XX.X | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Height z-score [2] | | | | | | | | | |
| n | XX | xx | xx | xx | xx | xx | xx | xx | xx |
| Mean | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX | xx, xx |
| Weight (kg) | | | | | | | | | |
| n | XX | xx | xx | xx | xx | xx | XX | xx | xx |
| Mean | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | XX.X | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Weight z-score [2] | | | | | | | | | |
| n | XX | xx | xx | xx | xx | XX | XX | xx | xx |
| Mean | XX.X | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | XX.X | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | XX.X, XX.X | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |




Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4) PCN Number: MIRU8967 premier research

# Table 14.1.3 (Cont'd) Demographics and Baseline Characteristics Safety Population

| | Р | rimary Cohort | | | PFIC Cohort | | | All Subjects | |
|---|---|---|---|---|---|---|---|---|---|
| Variable | Maralixibat | Placebo | Overall | Maralixibat | Placebo | Overall | Maralixibat | Placebo | Overall |
| Statistic or Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| BMI (kg/m2) | | | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX | XX | xx |
| Mean | XX.X | xx.x | xx.x | xx.x | xx.x | xx.x | XX.X | xx.x | xx.x |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | XX.X | xx.x | xx.x | xx.x | xx.x | xx.x | XX.X | xx.x | xx.x |
| Q1, Q3 | XX.X, XX.X | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | XX.X, XX.X | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| BMI z-score [2] | | | | | | | | | |
| n | XX | xx | XX | XX | XX | XX | XX | XX | xx |
| Mean | XX.X | xx.x | xx.x | xx.x | xx.x | xx.x | XX.X | xx.x | xx.x |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | XX.X | xx.x | xx.x | xx.x | xx.x | xx.x | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |




Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



## Table 14.1.4 Disease History and Baseline Disease Characteristics Safety Population

| | Pi | rimary Cohort | | | PFIC Cohort | | | All Subjects | |
|---|---|---|---|---|---|---|---|---|---|
| Variable | Maralixibat | Placebo | Overall | Maralixibat | Placebo | Overall | Maralixibat | Placebo | Overall |
| Statistic or Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Analysis PFIC Type [1] | | | | | | | | | |
| nt-PFIC2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| nt-PFIC2-IsBA | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| nt-PFIC2-surg | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| t-PFIC2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| PFIC1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| PFIC1-surg | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| PFIC3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| PFIC4 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| PFIC4-surg | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| PFIC6 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| nt-PFIC2-het | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| PFIC1-het | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No-variant-found | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Abbreviations: SD = standard deviation; SE = standard error of the mean; Q1 =  $25^{th}$  percentile; Q3 =  $75^{th}$  percentile; UDCA = ursodeoxycholic acid Note: Percentages are 100\*n/N, unless otherwise noted. Subjects with PFIC1 through PFIC6 all have the biallelic disease.

Only applicable for PFIC2 subjects, with exception of one nt-PFIC2 subject (015002) with heterozygosis ABCB11 mutation; N/A for all other subjects.

- [3] One subject (015002) had heterozygous ABCB11 mutation, and another (021006) had heterozygous ATP8B1 mutation.
- [4] Partial dates were imputed based on the SAP.
- [5] For the number and percent of subjects below and above the median baseline sBA level, the median is calculated separately for the Primary Cohort, PFIC Cohort, and All Subjects.
- [6] PELD score is calculated for children <12 years of age at the baseline visit; MELD score is calculated for children 12 years or older at the baseline visit.

Source: Reference Listings xx.x.x, xx.x.x


<sup>[1]</sup> nt-PFIC2 = non-truncated PFIC2 (primary cohort); nt-PFIC2-ISBA = non-truncated PFIC2 with low or fluctuating serum bile acids; nt-PFIC2-surg = non-truncated PFIC2 with a history of surgery; t-PFIC2 = truncated PFIC2; PFIC1-surg = PFIC1 with a history of surgery; PFIC4-surg = PFIC4 with a history of surgery; nt-PFIC2-het = non-truncated PFIC2 with heterozygosis; PFIC1-het = PFIC1 with heterozygosis; No-variant-found = No established variant linked to PFIC disease

<sup>[2]</sup> nt-PFIC2 = partial loss of BSEP function; t-PFIC2 = complete loss of BSEP function



Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



# Table 14.1.4 (Cont'd) Disease History and Baseline Disease Characteristics Safety Population

| | Pi | rimary Cohort | | | PFIC Cohort | | | All Subjects | |
|---|---|---|---|---|---|---|---|---|---|
| Variable | Maralixibat | Placebo | Overall | Maralixibat | Placebo | Overall | Maralixibat | Placebo | Overall |
| Statistic or Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=93) |
| Analysis PFIC Type (genotype) | | | | | | | | | |
| PFIC2 (ABCB11) [2] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| nt-PFIC2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| BSEP1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| BSEP2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| t-PFIC2 (BSEP3) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| PFIC1 (ATP8B1) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| PFIC3 (ABCB4) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| PFIC4 (TJP2) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| PFIC6 (MYO5B) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Heterozygous variant [3] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No-variant-found | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Liver masses detected at baseline | | | | | | | | | |
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |




Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4) PCN Number: MIRU8967 premier

# Table 14.1.4 (Cont'd) Disease History and Baseline Disease Characteristics Safety Population

| | P | rimary Cohort | | | PFIC Cohort | | | All Subjects | |
|---|---|---|---|---|---|---|---|---|---|
| Variable | Maralixibat | Placebo | Overall | Maralixibat | Placebo | Overall | Maralixibat | Placebo | Overall |
| Statistic or Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Time Since Original Diagnosis of | PFIC (months) [4] | | | | | | | | |
| n | XX | xx | xx | XX | xx | XX | XX | xx | xx |
| Mean | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | XX.X | xx.x |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xxx | xx, xxx | xx, xxx | xx, xxx | xx, xxx | xx, xxx | xx, xxx | xx, xxx | xx, xxx |
| Baseline UDCA Usage | | | | | | | | | |
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Baseline Rifampicin Usage | | | | | | | | | |
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Clinical Scratch Scale (CSS) Score | · | | | | | | | | |
| n | XX | xx | xx | Xx | xx | xx | XX | xx | xx |
| Mean | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| 0 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 4 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |




Protocol: MRX-502 (Amendment 4)

Sponsor: Mirum Pharmaceuticals Inc. PCN Number: MIRU8967

## Table 14.1.4 (Cont'd) Disease History and Baseline Disease Characteristics Safety Population

| | P | rimary Cohort | | | PFIC Cohort | | | All Subjects | |
|---|---|---|---|---|---|---|---|---|---|
| Variable | Maralixibat | Placebo | Overall | Maralixibat | Placebo | Overall | Maralixibat | Placebo | Overall |
| Statistic or Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Patient Impression of Severity (PIS) | | | | | | | | | |
| n | xx | xx | xx | XX | xx | XX | xx | XX | xx |
| Mean | XX.X | xx.x | XX.X | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| 0 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 4 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Caregiver Impression of Severity (CIS) | | | | | | | | | |
| n | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| Mean | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| 0 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 4 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |




Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



## Table 14.1.4 (Cont'd) Disease History and Baseline Disease Characteristics Safety Population

| | Р | rimary Cohort | | | PFIC Cohort | | | All Subjects | |
|---|---|---|---|---|---|---|---|---|---|
| Variable | Maralixibat | Placebo | Overall | Maralixibat | Placebo | Overall | Maralixibat | Placebo | Overall |
| Statistic or Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| ItchRO (Obs) 4-wk Morning Avg Severity Score | | | | | | | | | |
| n | xx | xx | xx | xx | xx | xx | xx | XX | xx |
| Mean | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | XX.X | xx.x | xx.x |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | XX.X | xx.x | XX.X |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| ItchRO (Pt) 4-wk Morning Avg Severity Score | | | | | | | | | |
| n | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| Mean | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| ItchRO (Obs) 4-wk Evening Avg Severity Score | | | | | | | | | |
| n | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| Mean | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | XX.X | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| ItchRO (Pt) 4-wk Evening Avg Severity Score | | | | | | | | | |
| n | xx | xx | xx | xx | xx | xx | xx | XX | xx |
| Mean | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |




Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



# Table 14.1.4 (Cont'd) Disease History and Baseline Disease Characteristics Safety Population

| | P | rimary Cohort | | | PFIC Cohort | | | All Subjects | |
|---|---|---|---|---|---|---|---|---|---|
| Variable | Maralixibat | Placebo | Overall | Maralixibat | Placebo | Overall | Maralixibat | Placebo | Overall |
| Statistic or Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| ItchRO (Obs) 4-wk Highest Daily Avg Severity Sco | ore | | | | | | | | |
| n | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| Mean | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX | xx, xx |
| ItchRO (Pt) 4-week Highest Daily Avg Severity | | | | | | | | | |
| Score | | | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | xx.x | xx.x | xx.x | xx.x | xx.x | XX.X | xx.x | xx.x |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | XX.X | xx.x | xx.x | xx.x | xx.x | xx.x | XX.X | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX |
| Total Serum Bile Acid (umol/L) [5] | | | | | | | | | |
| n | xx | xx | xx | xx | xx | XX | XX | XX | xx |
| Mean | XX.X | xx.x | XX.X | xx.x | xx.x | xx.x | XX.X | xx.x | xx.x |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | XX.X | xx.x | XX.X | xx.x | xx.x | xx.x | XX.X | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX | xx, xx | xx, xx |
| < Median | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| ≥ Median | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |




Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



## Table 14.1.4 (Cont'd) Disease History and Baseline Disease Characteristics Safety Population

| | Pri | mary Cohort | | | PFIC Cohort | | All Subjects | | |
|---|---|---|---|---|---|---|---|---|---|
| Variable | Maralixibat | Placebo | Overall | Maralixibat | Placebo | Overall | Maralixibat | Placebo | Overall |
| Statistic or Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |

### Repeat summary statistics for the following:

ItchRO (Obs & Pt) 4-wk avg frequency scores (6 variables); same order as for severity score

Alkaline Phosphate (U/L)

Aspartate Aminotransferase (U/L)

Alanine Aminotransferase (U/L)

Total Bilirubin (mg/dL)

Direct Bilirubin (mg/dL)

Fibroblast Growth Factor 19 (FGF-19) (ng/mL)

Autotaxin (ng/mL)

7 alpha-hydroxyl-4-cholesten-3-one (C4) (ng/mL)

25-Hydroxyvitamin D (ng/mL)

Alpha Tocopherol (mg/dL)

Prothrombin Intl. Normalized Ratio

Vitamin A (μg/dL)

GGT

Albumin (g/dL)

APRI

FIB-4

PELD [6] MELD [6]

> 



Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



## Table 14.1.5 Prior Medications/Therapies Safety Population

| | Pr | rimary Cohort | | | PFIC Cohort | | | All Subjects | |
|---|---|---|---|---|---|---|---|---|---|
| ATC | Maralixibat | Placebo | Overall | Maralixibat | Placebo | Overall | Maralixibat | Placebo | Overall |
| Preferred Term [1] | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Number of Subjects Taking any Prior Medications | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| ACT 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Term 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Term 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| ACT 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Term 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Term 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

etc...

Note: Percentages are 100\*n/N.

[1] Medications were coded using World Health Organization Drug Dictionary (WHO-DD Enhanced version September 2019) ATC level 2 and Chemical Substance (generic name). Subjects were counted only once for each Anatomical Therapeutic Chemical (ATC) or Preferred Term. Medications that started prior to the first dose of study drug will be considered a prior treatment, whether or not they were stopped prior to the first dose of study drug. If a treatment started prior to the first dose of study drug and continues after the first dose of study drug, it was considered both prior and concomitant.

Source: Reference Listings xx.x.x, xx.x.x




Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



### Table 14.1.6 Study Drug Compliance Safety Population

| | Р | rimary Cohort | | | PFIC Cohort | | | All Subjects | |
|---|---|---|---|---|---|---|---|---|---|
| Variable | Maralixibat | Placebo | Overall | Maralixibat | Placebo | Overall | Maralixibat | Placebo | Overall |
| Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Compliance (%) | | | | | | | | | |
| n | XX | xx | xx | xx | xx | XX | XX | xx | xx |
| Mean | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx |
| SD (SE) | x.xxx (x.xxx) | x.xxx (x.xxx) | x.xxx (x.xxx) | x.xxx (x.xxx) | x.xxx (x.xxx) | x.xxx (x.xxx) | x.xxx (x.xxx) | x.xxx (x.xxx) | x.xxx (x.xxx) |
| Median | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | XX.X, XX.X | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| <80% | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 80-<90% | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 90-100% | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Abbreviations: SD = standard deviation; SE = standard error of the mean; Q1 = 25th percentile; Q3 = 75th percentile

Note: Compliance (%) = 100\* (Treatment duration in days - Number of days both morning and evening doses were missed) / Treatment duration in days), where Treatment duration (days) = Date of last dose of study drug – Date of first dose of study drug + 1 day. For subjects that are missing the date of last dose of study drug, the last known contact date is used to calculate treatment duration.

Source: Reference Listings xx.x.x, xx.x.x




Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



## Table 14.2.1.1 Change from Baseline in ItchRO(Obs) Severity Score Tabulation of Fitted Summary Statistics from MMRM ITT Population – Primary Cohort

| Post-Baseline | Morning Score | | Evening | Score | Highest Da | ily Score |
|---|---|---|---|---|---|---|
| Analysis Visit Time Period<br>Statistic [1] | Maralixibat<br>(N=xx) | Placebo<br>(N=xx) | Maralixibat<br>(N=xx) | Placebo<br>(N=xx) | Maralixibat<br>(N=xx) | Placebo<br>(N=xx) |
| Weeks 1-6 | | | | | | |
| LS Mean (SE) | x.xx (x.xxx) | x.xx (x.xxx) | x.xx (x.xxx) | x.xx (x.xxx) | x.xx (x.xxx) | x.xx (x.xxx) |
| (95% CI for LS Mean) | (x.xx, x.xx) | (x.xx, x.xx) | (x.xx, x.xx) | (x.xx, x.xx) | (x.xx, x.xx) | (x.xx, x.xx) |
| p-value (CFB LS Mean = 0) | x.xxxx | x.xxxx | x.xxxx | x.xxxx | x.xxxx | X.XXXX |
| LS Mean Change from Placebo (SE) | x.xx (x.xxx) | | x.xx (x.xxx) | | x.xx (x.xxx) | |
| (95% CI for LS Mean Change from Placebo) | (x.xx, x.xx) | | (x.xx, x.xx) | | (x.xx, x.xx) | |
| p-value (Maralixibat LS Mean = Placebo LS Mean) | x.xxxx | | x.xxxx | | x.xxxx | |

(Continue for Time Periods: Weeks 7-10, Weeks 11-14, Weeks 15-18, Weeks 19-22, Weeks 23-26, and Weeks 15-26 [2])

Abbreviations: LS = Least-squares; SE = standard error of the mean; CFB = change from baseline; CI = confidence interval

[1] Estimates are from a mixed model for repeated measures (MMRM) with change from baseline as the dependent variable and fixed categorical effects of treatment group, time period and treatment-by-time period interaction as well as the continuous fixed covariates of average baseline score and baseline score-by-time period interaction.

[2] Average of time periods Weeks 15-18, 19-22, and 23-26 obtained from the MMRM as an equally weighted average of the 3 individual visit-specific estimates.

Source: Reference Listings xx.x.x, xx.x.x

Programming Note: There is enough space to fit 2 time periods per page (based on output from t\_mmrm.sas used on the 304 IA\_NDA analysis).


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



# Table 14.2.1.2 Change from Baseline in ItchRO(Obs) Severity Score MMRM Model Effects ITT Population – Primary Cohort

| | Overall p-value [1] | | |
|---|---|---|---|
| MMRM Model Effect | Morning Score | Evening Score | Highest Daily Score |
| Treatment Group | x.xxxx | x.xxxx | x.xxxx |
| Time Period | x.xxxx | x.xxxx | x.xxxx |
| Treatment Group x Time Period Interaction | x.xxxx | x.xxxx | x.xxxx |
| Baseline (Covariate) | x.xxxx | x.xxxx | x.xxxx |
| Baseline (Covariate) x Time Period Interaction | x.xxxx | x.xxxx | x.xxxx |

[1] p-value for testing the statistical significance of each effect in the repeated measures model. Change from baseline were analyzed using a restricted maximum likelihood (REML)-based repeated-measures approach. An unstructured covariance structure was used to model the within-subject errors. The Kenward-Roger approximation was used to estimate denominator degrees of freedom and adjust standard errors.

Source: Reference Listings xxxxxxx, xxxxxx


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.2.2.1.1
Change from Baseline in ItchRO(Obs) Severity Score
Tabulation of Fitted Summary Statistics from MMRM
ITT Population – PFIC Cohort

### Programming Notes: Repeat Table 14.2.1.1; change footnote [1] to:

[1] Estimates are from a mixed model for repeated measures (MMRM) with change from baseline as the dependent variable and fixed categorical effects of treatment group, time period and treatment-by-time period interaction as well as the continuous fixed covariates of average baseline score, baseline score-by-time period interaction, and PFIC type.

Table 14.2.2.1.2
Change from Baseline in ItchRO(Obs) Severity Score
MMRM Model Effects
ITT Population – PFIC Cohort

Programming Notes: Repeat Table 14.2.1.2, but add a data row as the last row: "PFIC Type (Covariate)" and add in the p-values from the model


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



# $\label{eq:Table 14.2.2.2.1} Table 14.2.2.2.1 \\ Change from Baseline in Total sBA ($\mu$mol/L) \\ Tabulation of Fitted Summary Statistics from MMRM \\ ITT Population$

| | Primary | / Cohort | PFIC Col | nort |
|---|---|---|---|---|
| Analysis Visit | Maralixibat | Placebo | Maralixibat | Placebo |
| Statistic [1] | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Week 2 | | | | |
| LS Mean (SE) | x.xx (x.xxx) | x.xx (x.xxx) | x.xx (x.xxx) | x.xx (x.xxx) |
| (95% CI for LS Mean) | (x.xx, x.xx) | (x.xx, x.xx) | (x.xx, x.xx) | (x.xx, x.xx) |
| p-value (CFB LS Mean = 0) | x.xxxx | x.xxxx | x.xxxx | x.xxxx |
| LS Mean Change from Placebo (SE) | x.xx (x.xxx) | | x.xx (x.xxx) | |
| (95% CI for LS Mean Change from Placebo) | (x.xx, x.xx) | | (x.xx, x.xx) | |
| p-value (Maralixibat LS Mean = Placebo LS Mean) | x.xxxx | | x.xxxx | |

(Continue for analysis visits: Week 6, Week 10, Week 14, Week 18, Week 22, Week 26, and Weeks 18-26 [2])

Abbreviations: LS = Least-squares; SE = standard error of the mean; CFB = change from baseline; CI = confidence interval

[1] Estimates are from a mixed model for repeated measures (MMRM) with change from baseline as the dependent variable and fixed categorical effects of treatment group, analysis visit and treatment-by-visit interaction as well as the continuous fixed covariates of baseline score and baseline score-by-visit interaction. For the PFIC Cohort, PFIC Type is included in the model as an additional covariate.

[2] Average of Weeks 18, 22, and 26 obtained from the MMRM as an equally weighted average of the 3 individual visit-specific estimates. Source: Reference Listings xx.x.x, xx.x.x

Programming Note: There is enough space to fit 2 time periods per page (based on output from t\_mmrm.sas used on the 304 IA\_NDA analysis).


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



### Table 14.2.2.2.2 Change from Baseline in Total sBA (µmol/L) MMRM Model Effects ITT Population

| | Overall p-value [1] | |
|---|---|---|
| MMRM Model Effect | Primary Cohort | PFIC Cohort |
| Treatment Group | x.xxxx | <0.0001 |
| Time Point (Analysis Visit) | x.xxxx | x.xxxx |
| Treatment Group x Time Point Interaction | x.xxxx | x.xxxx |
| Baseline (Covariate) | x.xxxx | x.xxxx |
| Baseline (Covariate) x Time Point Interaction | x.xxxx | x.xxxx |
| PFIC Type (Covariate) [2] | NA | x.xxxx |

[1] p-value for testing the statistical significance of each effect in the repeated measures model. Change from baseline were analyzed using a restricted maximum likelihood (REML)-based repeated-measures approach. An unstructured covariance structure was used to model the within-subject errors. The Kenward-Roger approximation was used to estimate denominator degrees of freedom and adjust standard errors.

[2] For the PFIC Cohort, PFIC Type is included in the MMRM model as an additional covariate.

Source: Reference Listings xxxxxxxx, xxxxxxx


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



## Table 14.2.2.3 Proportion of Responders ITT Population

| | Primary | Primary Cohort | | Cohort |
|---|---|---|---|---|
| Responder Type | Maralixibat | Placebo | Maralixibat | Placebo |
| Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| ItchRO Responders [1] | | | | |
| Responder | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Non-Responder | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| p-value vs. Placebo [3] | x.xxxx | | x.xxxx | |
| sBA Responders [2] | | | | |
| Responder | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Non-Responder | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| p-value vs. Placebo [3] | x.xxxx | | x.xxxx | |

Note: Percentages are 100\*n/N.

[1] ItchRO responders are defined as a subject having a 4-week average morning ItchRO(Obs) severity change from baseline of ≤-1.0 OR an average severity score of ≤1.0. For the purpose of determining response, the average severity score from the three 4-week periods (Weeks 15-18, 19-22, and 23-26) are used. A subject is defined as an ItchRO non-responder if the 4-week average baseline score is missing OR all three 4-week average (post-baseline) scores are missing.

[2] sBA responders are defined as a subject having an average sBA level of <102 µmol/L (applies only if baseline sBA level was ≥102 µmol/L), OR a ≤-75% average percent change from baseline. For the purpose of determining response, the average sBA value from Weeks 18, 22, and 26 values are used. A subject is defined as an sBA non-responder if the baseline sBA value is missing OR sBA values are missing at all 3 time points (i.e., Weeks 18, 22, and 26).

[3] p-values comparing maralixibat to placebo treatment groups are calculated using a Barnard's exact test.

Source: Reference Listings xx.x.x, xx.x.x


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



#### Table 14.2.3.1.1

Change from Baseline in Morning ItchRO(Obs) Severity Score – Sibling Sensitivity Analysis
Tabulation of Fitted Summary Statistics from MMRM
ITT Population

#### Programming Notes: Repeat Table 14.2.2.2.1; add following Note, and change footnotes [1] and [2] to:

Note: The data from all enrolled subjects (including the 2 pairs of siblings) are used for primary efficacy analysis. The data for only 1 sibling is used for the sensitivity analysis. The choice of sibling is made at random before the database lock, as described in the SAP.

- [1] Estimates are from a mixed model for repeated measures (MMRM) with change from baseline as the dependent variable and fixed categorical effects of treatment group, time period and treatment-by-time period interaction as well as the continuous fixed covariates of average baseline score, and baseline score-by-time period interaction. For the PFIC Cohort, PFIC Type is included in the model as an additional covariate
- [2] Average of time periods Weeks 15-18, 19-22, and 23-26 obtained from the MMRM as an equally weighted average of the 3 individual visit-specific estimates.

Table 14.2.3.1.2

Change from Baseline in Morning ItchRO(Obs) Severity Score – Sibling Sensitivity Analysis

MMRM Model Effects

ITT Population

Programming Notes: Repeat Table 14.2.2.2.2; change 'Time Point (Analysis Visit)' in 2<sup>nd</sup> data row to 'Time Period', and 'Time Period' in data rows 3 and 5 to 'Time Period'

Table 14.2.3.2

Change from Baseline in Morning ItchRO(Obs) Severity Score – Multiple Imputation Sensitivity Analysis
Tabulation of Fitted Summary Statistics from MMRM
ITT Population

#### Programming Notes: Repeat Table 14.2.2.2.1; add following Note, and change footnotes [1] and [2] (same as 14.2.3.1.1) to:

Note: Multiple imputation is based on a standard Missing at Random (MAR) imputation approach. The MAR imputation model imputes missing values using a regression-based multiple imputation model.

- [1] Estimates are from a mixed model for repeated measures (MMRM) with change from baseline as the dependent variable and fixed categorical effects of treatment group, time period and treatment-by-time period interaction as well as the continuous fixed covariates of average baseline score, and baseline score-by-time period interaction. For the PFIC Cohort, PFIC Type is included in the model as an additional covariate.
- [2] Average of time periods Weeks 15-18, 19-22, and 23-26 obtained from the MMRM as an equally weighted average of the 3 individual visit-specific estimates.


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



# Table 14.2.3.3 Change from Baseline in Morning ItchRO(Obs) Severity Score to Average of Last 12 Weeks – Tipping Point Sensitivity Analysis Tabulation of Fitted Summary Statistics from MMRM ITT Population

| | | Primary Cohort | | PFIC Cohort | |
|---|---|---|---|---|---|
| Shift Parameters for | | Maralixibat | Placebo | Maralixibat | Placebo |
| Maralixibat, Placebo | Statistic [1] | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| x.xx, x.xx | LS Mean (SE) | x.xx (x.xxx) | x.xx (x.xxx) | x.xx (x.xxx) | x.xx (x.xxx |
| | (95% CI for LS Mean) | (x.xx, x.xx) | (x.xx, x.xx) | (x.xx, x.xx) | (x.xx, x.xx |
| | p-value (CFB LS Mean = 0) | x.xxxx | x.xxxx | x.xxxx | x.xxxx |
| | LS Mean Change from Placebo (SE) | x.xx (x.xxx) | | x.xx (x.xxx) | |
| | (95% CI for LS Mean Change from Placebo) | (x.xx, x.xx) | | (x.xx, x.xx) | |
| | p-value (Maralixibat LS Mean = Placebo LS Mean) | x.xxxx | | x.xxxx | |

#### (Continue for other shift parameters)

Abbreviations: LS = Least-squares; SE = standard error of the mean; CFB = change from baseline; CI = confidence interval Note: Average of time periods Weeks 15-18, 19-22, and 23-26 obtained from the MMRM as an equally weighted average of the 3 individual visit-specific estimates.

[1] Estimates are from a mixed model for repeated measures (MMRM) with change from baseline as the dependent variable and fixed categorical effects of treatment group, time period and treatment-by-time period interaction as well as the continuous fixed covariates of average baseline score and baseline score-by-time period interaction. For the PFIC Cohort, PFIC Type is included in the model as an additional covariate.

Source: Reference Listings xx.x.x, xx.x.x


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



# Table 14.2.3.4.1 Change from Baseline in Total sBA (µmol/L) – Sibling Sensitivity Analysis Tabulation of Fitted Summary Statistics from MMRM ITT Population

#### Programming Notes: Repeat Table 14.2.2.2.1; add Note:

Note: The data from all enrolled subjects (including the 2 pairs of siblings) are used for primary efficacy analysis. The data for only 1 sibling is used for the sensitivity analysis. The choice of sibling is made at random before the database lock, as described in the SAP.

Table 14.2.3.4.2
Change from Baseline in Total sBA (µmol/L) – Sibling Sensitivity Analysis
MMRM Model Effects
ITT Population

Programming Notes: Repeat Table 14.2.2.2.2

 $Table\ 14.2.3.5$  Change from Baseline in Total sBA (µmol/L) – Multiple Imputation Sensitivity Analysis Tabulation of Fitted Summary Statistics from MMRM ITT Population

#### Programming Notes: Repeat Table 14.2.2.2.1; add Note:

Note: Multiple imputation is based on a standard Missing at Random (MAR) imputation approach. The MAR imputation model imputes missing values using a regression-based multiple imputation model.

Table 14.2.3.5.2
Change from Baseline in Total sBA (µmol/L) – Multiple Imputation Sensitivity Analysis
MMRM Model Effects
ITT Population

Programming Notes: Repeat Table 14.2.2.2.2


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



#### Table 14.2.3.6

Change from Baseline in Total sBA (µmol/L) to Average of Weeks 18, 22, and 26 – Tipping Point Sensitivity Analysis
Tabulation of Fitted Summary Statistics from MMRM
ITT Population

### Programming Notes: Repeat Table 14.2.3.3; change Note and footnote to:

Note: Average of Weeks 18, 22, and 26 obtained from the MMRM as an equally weighted average of the 3 individual visit-specific estimates. [1] Estimates are from a mixed model for repeated measures (MMRM) with change from baseline as the dependent variable and fixed categorical effects of treatment group, analysis visit and treatment-by-visit interaction as well as the continuous fixed covariates of baseline score and baseline score-by-visit interaction. For the PFIC Cohort, PFIC Type is included in the model as an additional covariate.


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



# Table 14.2.4.1.1 Change from Baseline in Morning ItchRO(Obs) Severity Score Tabulation of Fitted Summary Statistics from MMRM Per Protocol Population – Primary Cohort

| Analysis Visit Time Period | Maralixibat | Placebo |
|---|---|---|
| Statistic [1] | (N=xx) | (N=xx) |
| Weeks 1-6 | | |
| LS Mean (SE) | x.xx (x.xxx) | x.xx (x.xxx) |
| (95% CI for LS Mean) | (x.xx, x.xx) | (x.xx, x.xx) |
| p-value (CFB LS Mean = 0) | x.xxxx | X.XXXX |
| LS Mean Change from Placebo (SE) | x.xx (x.xxx) | |
| (95% CI for LS Mean Change from Placebo) | (x.xx, x.xx) | |
| p-value (Maralixibat LS Mean = Placebo LS Mean) | X.XXXX | |

(Continue for Time Periods: Weeks 7-10, Weeks 11-14, Weeks 15-18, Weeks 19-22, Weeks 23-26, and Weeks 15-26 [2])

Abbreviations: LS = Least-squares; SE = standard error of the mean; CFB = change from baseline; CI = confidence interval

[1] Estimates are from a mixed model for repeated measures (MMRM) with change from baseline as the dependent variable and fixed categorical effects of treatment group, time period and treatment-by-time period interaction as well as the continuous fixed covariates of average baseline score and baseline score-by-time period interaction.

[2] Average of time periods Weeks 15-18, 19-22, and 23-26 obtained from the MMRM as an equally weighted average of the 3 individual visit-specific estimates.

Source: Reference Listings xx.x.x, xx.x.x


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



# Table 14.2.4.1.2 Change from Baseline in Morning ItchRO(Obs) Severity Score MMRM Model Effects Per Protocol Population – Primary Cohort

| | Overall |
|------------------------------------------------|-------------|
| MMRM Model Effect | p-value [1] |
| Treatment Group | x.xxxx |
| Time Period | x.xxxx |
| Treatment Group x Time Period Interaction | x.xxxx |
| Baseline (Covariate) | x.xxxx |
| Baseline (Covariate) x Time Period Interaction | x.xxxx |

[1] p-value for testing the statistical significance of each effect in the repeated measures model. Change from baseline were analyzed using a restricted maximum likelihood (REML)-based repeated-measures approach. An unstructured covariance structure was used to model the within-subject errors. The Kenward-Roger approximation was used to estimate denominator degrees of freedom and adjust standard errors.

Source: Reference Listings xxxxxxx, xxxxxx


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



# Table 14.2.4.2.1 Change from Baseline in Total sBA (μmol/L) Tabulation of Fitted Summary Statistics from MMRM Per Protocol Population – Primary Cohort

| Analysis Visit<br>Statistic [1] | Maralixibat<br>(N=xx) | Placebo<br>(N=xx) |
|---|---|---|
| Week 2 | | |
| LS Mean (SE) | x.xx (x.xxx) | x.xx (x.xxx) |
| (95% CI for LS Mean) | (x.xx, x.xx) | (x.xx, x.xx) |
| p-value (CFB LS Mean = 0) | x.xxxx | x.xxxx |
| LS Mean Change from Placebo (SE) | x.xx (x.xxx) | |
| (95% CI for LS Mean Change from Placebo) | (x.xx, x.xx) | |
| p-value (Maralixibat LS Mean = Placebo LS Mean) | x.xxxx | |

(Continue for analysis visits: Week 6, Week 10, Week 14, Week 18, Week 22, Week 26, and Weeks 18-26 [2])

Abbreviations: LS = Least-squares; SE = standard error of the mean; CFB = change from baseline; CI = confidence interval [1] Estimates are from a mixed model for repeated measures (MMRM) with change from baseline as the dependent variable and fixed categorical effects of treatment group, analysis visit and treatment-by-visit interaction as well as the continuous fixed covariates of baseline score and baseline score-by-visit interaction.

[2] Average of Weeks 18, 22, and 26 obtained from the MMRM as an equally weighted average of the 3 individual visit-specific estimates.

Source: Reference Listings xx.x.x, xx.x.x


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



## Table 14.2.4.2.2 Change from Baseline in Total sBA (μmol/L) MMRM Model Effects Per Protocol Population – Primary Cohort

| | Overall |
|-----------------------------------------------|-------------|
| MMRM Model Effect | p-value [1] |
| Treatment Group | x.xxxx |
| Time Point (Analysis Visit) | x.xxxx |
| Treatment Group x Time Point Interaction | x.xxxx |
| Baseline (Covariate) | x.xxxx |
| Baseline (Covariate) x Time Point Interaction | x.xxxx |

[1] p-value for testing the statistical significance of each effect in the repeated measures model. Change from baseline were analyzed using a restricted maximum likelihood (REML)-based repeated-measures approach. An unstructured covariance structure was used to model the within-subject errors. The Kenward-Roger approximation was used to estimate denominator degrees of freedom and adjust standard errors.

Source: Reference Listings xxxxxxx, xxxxxx


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.2.4.3.1
Change from Baseline in Weekly Average Morning ItchRO(Obs) Severity Score
Descriptive Statistics by Analysis Week
ITT Population – Primary Cohort

| Analysis Visit | Maralixibat | Placebo |
|----------------|---------------|---------------|
| Statistic | (N=xx) | (N=xx) |
| Week 1 | | |
| n | xx | xx |
| Mean | xx.x | xx.x |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx |
| Week 2 | | |
| n | xx | XX |
| Mean | xx.x | xx.x |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx |

(Continue for analysis visits: Week 3, 4, . . . , 26)

Abbreviations: SD = standard deviation; SE = standard error of the mean;

Q1 = 25<sup>th</sup> percentile; Q3 = 75<sup>th</sup> percentile

Note: Baseline morning ltchRO(Obs) severity score is the average of 4-weekly (7-day) average scores in the period consisting of the 28 days immediately

before the date of first dose of study drug. Source: Reference Listings xx.x.x, xx.x.x


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.2.4.3.2

Change from Baseline in Weekly Average Morning ItchRO(Obs) Severity Score by Region

Descriptive Statistics by Analysis Week

ITT Population – Primary Cohort

| | E | urope | Mido | dle East | North . | America | South and C | entral America |
|---|---|---|---|---|---|---|---|---|
| Analysis Visit | Maralixibat | Placebo | Maralixibat | Placebo | Maralixibat | Placebo | Maralixibat | Placebo |
| Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Week 1 | | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX | xx |
| Mean | XX.X | XX.X | XX.X | XX.X | xx.x | xx.x | xx.x | xx.x |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Week 2 | | | | | | | | |
| n | XX | Xx | XX | XX | XX | XX | XX | xx |
| Mean | XX.X | xx.x | XX.X | XX.X | xx.x | xx.x | xx.x | xx.x |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | xx.x | XX.X | XX.X | XX.X | xx.x | xx.x | XX.X | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |

(Continue for analysis visits: Week 3, 4, . . . , 26)

Abbreviations: SD = standard deviation; SE = standard error of the mean; Q1 = 25th percentile; Q3 = 75th percentile

Note: There are no Primary Cohort subjects in Asia. Baseline morning ItchRO(Obs) severity score is the average of 4-weekly (7-day) average scores in the period consisting of the 28 days immediately before the date of first dose of study drug.

Source: Reference Listings xx.x.x, xx.x.x


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.2.4.3.3

Change from Baseline in Weekly Average Morning ItchRO(Obs) Severity Score by Age at Baseline

Descriptive Statistics by Analysis Week

ITT Population – Primary Cohort

| | 1 to < | 6 Years | 6 to <1 | .3 Years | 13 to | 18 Years |
|---|---|---|---|---|---|---|
| Analysis Visit | Maralixibat | Placebo | Maralixibat | Placebo | Maralixibat | Placebo |
| Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Week 1 | | | | | | |
| n | XX | XX | XX | xx | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | xx.x |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | XX.X | XX.X | xx.x | XX.X | XX.X | xx.x |
| Q1, Q3 | XX.X, XX.X | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | XX.X, XX.X | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Week 2 | | | | | | |
| n | XX | xx | XX | xx | xx | xx |
| Mean | XX.X | XX.X | xx.x | XX.X | XX.X | xx.x |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | XX.X | XX.X | xx.x | XX.X | XX.X | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |

(Continue for analysis visits: Week 3, 4, . . . , 26)

Abbreviations: SD = standard deviation; SE = standard error of the mean; Q1 = 25th percentile; Q3 = 75th percentile

Note: Age groups based in full years. Baseline morning ItchRO(Obs) severity score is the average of 4-weekly (7-day) average scores in the period consisting of the 28 days immediately before the date of first dose of study drug.

Source: Reference Listings xx.x.x, xx.x.x


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.2.4.3.4

Change from Baseline in Weekly Average Morning ItchRO(Obs) Severity Score by Sex
Descriptive Statistics by Analysis Week

ITT Population – Primary Cohort

| | | Male | Female | |
|---|---|---|---|---|
| Analysis Visit | Maralixibat | Placebo | Maralixibat | Placebo |
| Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Week 1 | | | | |
| n | XX | XX | XX | xx |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx |
| Week 2 | | | | |
| n | XX | XX | XX | xx |
| Mean | XX.X | XX.X | XX.X | xx.x |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | XX.X | XX.X | xx.x | xx.x |
| Q1, Q3 | XX.X, XX.X | xx.x, xx.x | XX.X, XX.X | xx.x, xx.x |
| Min, Max | XX, XX | XX, XX | xx, xx | xx, xx |

(Continue for analysis visits: Week 3, 4, . . . , 26)

Abbreviations: SD = standard deviation; SE = standard error of the mean; Q1 = 25<sup>th</sup> percentile; Q3 = 75<sup>th</sup> percentile Note: Baseline morning ItchRO(Obs) severity score is the average of 4-weekly (7-day) average scores in the period consisting of the 28 days immediately before the date of first dose of study drug.

Source: Reference Listings xx.x.x, xx.x.x


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



#### Table 14.2.4.3.5

Change from Baseline in Weekly Average Morning ItchRO(Obs) Severity Score by Race
Descriptive Statistics by Analysis Week
ITT Population – Primary Cohort

Programming Notes: Repeat Table 14.2.4.3.2, replacing the 4 Regions with the 4 Races: White, Black or African American, American Indian or Alaska Native, and More than One Race; change 1<sup>st</sup> sentence in Note to "There is 1 Primary Cohort subject (038002) that did not report their race. No Primary Cohort subjects reported as Asian."

#### Table 14.2.4.3.6

Change from Baseline in Weekly Average Morning ItchRO(Obs) Severity Score by Baseline Median sBA

Descriptive Statistics by Analysis Week

ITT Population – Primary Cohort

Programming Notes: Repeat Table 14.2.4.3.4, replacing the 2 Sexes with the 2 baseline sBA categories: < Baseline Median sBA; ≥ Baseline Median sBA; add the following as the 1<sup>st</sup> few sentences to the Note: "Three subjects (002003, 028003, and 031002), all in the Primary Cohort, are missing baseline sBA samples. Only subjects in the Primary Cohort are used to calculate the baseline median sBA level."

#### Table 14.2.4.3.7

Change from Baseline in Weekly Average Morning ItchRO(Obs) Severity Score by Baseline UDCA Usage
Descriptive Statistics by Analysis Week
ITT Population – Primary Cohort

Programming Notes: Repeat Table 14.2.4.3.4, replacing the 2 Sexes with the 2 baseline UDCA usage categories: Baseline UDCA Usage, No Baseline UDCA Usage; add abbreviation for UDCA: "UDCA = ursodeoxycholic acid" with other abbreviations; add the following as the 1st sentence to the Note:

"A subject reporting the use of UDCA, based on ATC Class Level 5 (chemical substance), with a start date on or prior to the first dose of study drug and either be ongoing or have a stop date on or after the first dose of study drug would be considered as using UDCA at baseline."


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.2.4.3.8

Change from Baseline in Weekly Average Morning ItchRO(Obs) Severity Score by Baseline Rifampicin Usage

Descriptive Statistics by Analysis Week

ITT Population – Primary Cohort

Programming Notes: Repeat Table 14.2.4.3.4, replacing the 2 Sexes with the 2 baseline Rifampicin usage categories: Baseline Rifampicin Usage, No Baseline Rifampicin Usage; add the following as the 1<sup>st</sup> sentence to the Note:

"A subject reporting the use of Rifampicin, based on ATC Class Level 5 (chemical substance), with a start date on or prior to the first dose of study drug and either be ongoing or have a stop date on or after the first dose of study drug would be considered as using Rifampicin at baseline."

Table 14.2.4.3.9

Change from Baseline in Weekly Average Morning ItchRO(Obs) Severity Score by BSEP Type

Descriptive Statistics by Analysis Week

ITT Population – Primary Cohort

Programming Notes: Repeat Table 14.2.4.3.4, replacing the 2 Sexes with the 2 BSEP types: BSEP 1. BSEP 2


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.2.4.4.1 Change from Baseline in Total sBA (μmol/L) Descriptive Statistics by Analysis Week ITT Population – Primary Cohort

| Analysis Visit | Maralixibat | Placebo |
|----------------|---------------|---------------|
| Statistic | (N=xx) | (N=xx) |
| Week 2 | | |
| n | xx | xx |
| Mean | xx.x | xx.x |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | xx.x | XX.X |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx |
| Week 6 | | |
| N | xx | XX |
| Mean | xx.x | XX.X |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | xx.x | XX.X |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | XX, XX |

(Continue for analysis visits: Week 10, Week 14, Week 18, Week 22, and Week 26)

Abbreviations: SD = standard deviation; SE = standard error of the mean;

Q1 = 25<sup>th</sup> percentile; Q3 = 75<sup>th</sup> percentile Source: Reference Listings xx.x.x, xx.x.x


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



## Table 14.2.4.4.2 Change from Baseline in Total sBA (μmol/L) by Region Descriptive Statistics by Analysis Week ITT Population – Primary Cohort

| | E | urope | Mido | lle East | North . | America | South and C | entral America |
|---|---|---|---|---|---|---|---|---|
| Analysis Visit | Maralixibat | Placebo | Maralixibat | Placebo | Maralixibat | Placebo | Maralixibat | Placebo |
| Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Week 2 | | | | | | | | |
| n | XX | XX | XX | xx | XX | xx | XX | xx |
| Mean | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X | xx.x | XX.X |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | xx.x | xx.x | XX.X | XX.X | xx.x | XX.X | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | XX.X, XX.X | XX.X, XX.X | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Week 6 | | | | | | | | |
| n | XX | Xx | XX | xx | XX | xx | XX | xx |
| Mean | xx.x | xx.x | xx.x | XX.X | xx.x | XX.X | xx.x | xx.x |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | xx.x | xx.x | XX.X | XX.X | xx.x | XX.X | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |

(Continue for analysis visits: Week 10, Week 14, Week 18, Week 22, and Week 26)

Abbreviations: SD = standard deviation; SE = standard error of the mean; Q1 = 25<sup>th</sup> percentile; Q3 = 75<sup>th</sup> percentile

Note: There are no Primary Cohort subjects in Asia.

Source: Reference Listings xx.x.x, xx.x.x

**Programming Notes:** Add 'NE = not estimable' to abbreviations where applicable


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.2.4.4.3
Change from Baseline in Total sBA (µmol/L) by Age at Baseline
Descriptive Statistics by Analysis Week
ITT Population – Primary Cohort

| | 1 to < | <6 Years | 6 to <1 | L3 Years | 13 to | 18 Years |
|---|---|---|---|---|---|---|
| Analysis Visit | Maralixibat | Placebo | Maralixibat | Placebo | Maralixibat | Placebo |
| Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Week 2 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | xx.x |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | xx.x |
| Q1, Q3 | XX.X, XX.X | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Week 6 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | xx.x | xx.x | XX.X | xx.x |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | XX.X | XX.X | xx.x | xx.x | XX.X | xx.x |
| Q1, Q3 | XX.X, XX.X | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | XX.X, XX.X | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |

(Continue for analysis visits: Week 10, Week 14, Week 18, Week 22, and Week 26)

Abbreviations: SD = standard deviation; SE = standard error of the mean; Q1 = 25th percentile; Q3 = 75th percentile

Note: Age groups based in full years. Source: Reference Listings xx.x.x, xx.x.x


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.2.4.4.4
Change from Baseline in Total sBA (μmol/L) by Sex
Descriptive Statistics by Analysis Week
ITT Population – Primary Cohort

| | | Male | Female | |
|---|---|---|---|---|
| Analysis Visit | Maralixibat | Placebo | Maralixibat | Placebo |
| Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Week 2 | | | | |
| n | XX | XX | XX | xx |
| Mean | XX.X | XX.X | XX.X | xx.x |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | XX.X | XX.X | XX.X | xx.x |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx |
| Week 6 | | | | |
| n | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | xx.x |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | xx.x | XX.X | XX.X | xx.x |
| Q1, Q3 | XX.X, XX.X | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx |

(Continue for analysis visits: Week 10, Week 14, Week 18, Week 22, and Week 26)

Abbreviations: SD = standard deviation; SE = standard error of the mean; Q1 = 25<sup>th</sup> percentile; Q3 = 75<sup>th</sup> percentile Source: Reference Listings xx.x.x, xx.x.x


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.2.4.4.5
Change from Baseline in Total sBA (μmol/L) by Race
Descriptive Statistics by Analysis Week
ITT Population – Primary Cohort

Programming Notes: Repeat Table 14.2.4.4.2, replacing the 4 Regions with the 4 Races: White, Black or African American, American Indian or Alaska Native, and More than One Race; change 1<sup>st</sup> sentence in Note to "There is 1 Primary Cohort subject (038002) that did not report their race. No Primary Cohort subjects reported as Asian."

Table 14.2.4.4.6
Change from Baseline in Total sBA (µmol/L) by Baseline Median sBA
Descriptive Statistics by Analysis Week
ITT Population – Primary Cohort

Programming Notes: Repeat Table 14.2.4.4.4, replacing the 2 Sexes with the 2 baseline sBA categories: < Baseline Median sBA; ≥ Baseline Median sBA; add the following as the 1<sup>st</sup> few sentences to the Note: "Three subjects (002003, 028003, and 031002), all in the Primary Cohort, are missing baseline sBA samples. Only subjects in the Primary Cohort are used to calculate the baseline median sBA level."

Table 14.2.4.4.7
Change from Baseline in Total sBA (μmol/L) by Baseline UDCA Usage
Descriptive Statistics by Analysis Week
ITT Population – Primary Cohort

Programming Notes: Repeat Table 14.2.4.4.4, replacing the 2 Sexes with the 2 baseline UDCA usage categories: Baseline UDCA Usage, No Baseline UDCA Usage; add abbreviation for UDCA: "UDCA = ursodeoxycholic acid" with other abbreviations; add the following as the 1st sentence to the Note:
"A subject reporting the use of UDCA, based on ATC Class Level 5 (chemical substance), with a start date on or prior to the first dose of study drug and either be ongoing or have a stop date on or after the first dose of study drug would be considered as using UDCA at baseline."


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.2.4.4.8

Change from Baseline in Total sBA (µmol/L) by Baseline Rifampicin Usage
Descriptive Statistics by Analysis Week

ITT Population – Primary Cohort

Programming Notes: Repeat Table 14.2.4.4.4, replacing the 2 Sexes with the 2 baseline Rifampicin usage categories: Baseline Rifampicin Usage, No Baseline Rifampicin Usage; add the following as the 1st sentence to the Note:

"A subject reporting the use of Rifampicin, based on ATC Class Level 5 (chemical substance), with a start date on or prior to the first dose of study drug and either be ongoing or have a stop date on or after the first dose of study drug would be considered as using Rifampicin at baseline."

Table 14.2.4.4.9
Change from Baseline in Total sBA (μmol/L) by BSEP Type
Descriptive Statistics by Analysis Week
ITT Population – Primary Cohort

Programming Notes: Repeat Table 14.2.4.4.4, replacing the 2 Sexes with the 2 BSEP types: BSEP 1. BSEP 2


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.2.4.5.1
Change from Baseline in ALT (U/L)
Tabulation of Fitted Summary Statistics from MMRM
ITT Population

Programming Notes: Repeat Table 14.2.2.2.1

Table 14.2.4.5.2
Change from Baseline in ALT (U/L)
MMRM Model Effects
ITT Population

Programming Notes: Repeat Table 14.2.2.2.2

Table 14.2.4.6.1
Change from Baseline in AST (U/L)
Tabulation of Fitted Summary Statistics from MMRM
ITT Population

Programming Notes: Repeat Table 14.2.2.2.1

Table 14.2.4.6.2 Change from Baseline in AST (U/L) MMRM Model Effects ITT Population

Programming Notes: Repeat Table 14.2.2.2.2


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.2.4.7.1 Change from Baseline in Total Bilirubin (mg/dL Tabulation of Fitted Summary Statistics from MMRM **ITT Population** 

Programming Notes: Repeat Table 14.2.2.2.1

Table 14.2.4.7.2 Change from Baseline in Total Bilirubin (mg/dL) MMRM Model Effects **ITT Population** 

Programming Notes: Repeat Table 14.2.2.2.2

Table 14.2.4.8.1 Change from Baseline in Direct Bilirubin (mg/dL) Tabulation of Fitted Summary Statistics from MMRM **ITT Population** 

Programming Notes: Repeat Table 14.2.2.2.1

Table 14.2.4.8.2 Change from Baseline in Direct Bilirubin (mg/dL) MMRM Model Effects **ITT Population** 

Programming Notes: Repeat Table 14.2.2.2.2


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.2.4.9.1
Change from Baseline in ALP (U/L)
Tabulation of Fitted Summary Statistics from MMRM
ITT Population

Programming Notes: Repeat Table 14.2.2.2.1

Table 14.2.4.9.2
Change from Baseline in ALP (U/L)
MMRM Model Effects
ITT Population

Programming Notes: Repeat Table 14.2.2.2.2

Table 14.2.4.10.1 Change from Baseline in GGT (U/L) Tabulation of Fitted Summary Statistics from MMRM ITT Population

Programming Notes: Repeat Table 14.2.2.2.1

Table 14.2.4.10.2 Change from Baseline in GGT (U/L) MMRM Model Effects ITT Population

Programming Notes: Repeat Table 14.2.2.2.2


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.2.4.11.1
Change from Baseline in FIB-4
Tabulation of Fitted Summary Statistics from MMRM
ITT Population

Programming Notes: Repeat Table 14.2.2.2.1; add to Abbreviations: 'FIB-4 = fibrosis-4'; add Note: Note: FIB-4 is based on a subject's age in years at the time of sample collection.

Table 14.2.4.11.2 Change from Baseline in FIB-4 MMRM Model Effects ITT Population

Programming Notes: Repeat Table 14.2.2.2.2

Table 14.2.4.12.1
Change from Baseline in APRI
Tabulation of Fitted Summary Statistics from MMRM
ITT Population

Programming Notes: Repeat Table 14.2.2.2.1; add to Abbreviations: 'APRI = AST to platelet ratio index'

Table 14.2.4.12.2 Change from Baseline in APRI MMRM Model Effects ITT Population

Programming Notes: Repeat Table 14.2.2.2.2


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.2.4.13.1
Change from Baseline in PELD
Tabulation of Fitted Summary Statistics from MMRM
ITT Population

Programming Notes: Repeat Table 14.2.2.2.1; add to Abbreviations: 'PELD = pediatric end-stage liver disease'; add Note:

Note: PELD score is calculated for children under 12 years of age at the baseline visit.

Table 14.2.4.13.2
Change from Baseline in PELD
MMRM Model Effects
ITT Population

Programming Notes: Repeat Table 14.2.2.2.2


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.2.4.14

Total sBA Shift from Baseline: Number and Proportion of Subjects

ITT Population

| | Prima | ry Cohort | PFIC ( | Cohort | All Subjects | |
|---|---|---|---|---|---|---|
| Analysis Visit | Maralixibat | Placebo | Maralixibat | Placebo | Maralixibat | Placebo |
| % Decrease from Baseline | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Week 2 | nn | nn | nn | nn | nn | nn |
| >75% (large decrease) | xx (xx.x%) | x xx (xx.x%) | x xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 0 to 75% (decrease) | xx (xx.x%) | x xx (xx.x%) | x xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| <0% (any increase) | xx (xx.x%) | x xx (xx.x%) | x xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| p-value vs Placebo [1] | x.xxxx | | x.xxxx | | x.xxxx | |
| Week 6 | nn | nn | nn | nn | nn | nn |
| >75% (large decrease) | xx (xx.x%) | x xx (xx.x%) | x xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 0 to 75% (decrease) | xx (xx.x%) | x xx (xx.x%) | x xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| <0% (any increase) | xx (xx.x%) | x xx (xx.x%) | x xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| p-value vs Placebo [1] | x.xxxx | | x.xxxx | | x.xxxx | |
| Week 10 | nn | nn | nn | nn | nn | nn |
| >75% (large decrease) | xx (xx.x%) | x xx (xx.x%) | x xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 0 to 75% (decrease) | xx (xx.x%) | x xx (xx.x%) | x xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| <0% (any increase) | xx (xx.x%) | x xx (xx.x%) | x xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| p-value vs Placebo [1] | x.xxxx | | x.xxxx | | x.xxxx | |

(Continue for analysis visits: Week 14, Week 18, Week 22, and Week 26)

Note: Percentages are 100\*n/Number of subjects with non-missing change from baseline in total sBA values at each visit.

[1] p-value is calculated using a Cochran-Mantel-Haenszel (CMH) test.

Source: Reference Listing xx.x.x

Programming Note: nn is # of subjects with non-missing CFB in total sBA data. For these ordinal non-binary outcomes, the CMH test is used to take the ordinal nature of the variable into account.


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



# Table 14.2.4.15 Number of Days Morning ItchRO(Obs) Severity Score ≤1 Over the Last 84 Study Days ITT Population

| | Prim | ary Cohort | PFIC Cohort | |
|---|---|---|---|---|
| | Maralixibat | Placebo | Maralixibat | Placebo |
| Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Mean | xx.x | xx.x | xx.x | xx.x |
| (95% CI for Mean) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | xx.x | XX.X | XX.X | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | XX.X, XX.X | xx.x, xx.x |
| Min, Max | XX, XX | xx, xx | xx, xx | xx, xx |
| Mean Change from Placebo | xx.x | | xx.x | |
| (95% CI for Mean Change from Placebo) | (xx.x, xx.x) | | (xx.x, xx.x) | |
| p-value (Maralixibat Mean = Placebo Mean [1] | x.xxxx | | x.xxxx | |

Abbreviations: SD = standard deviation; SE = standard error of the mean; Q1 = 25<sup>th</sup> percentile; Q3 = 75<sup>th</sup> percentile; CI = confidence interval

Note: ItchRO scores have a range from 0 to 4, with the higher score indicating increasing itch severity. Missing data during the 84-day period is treated using the most conservative approach (i.e., severity score >1).

[1] Student's 2 sample mean t-test, assuming unequal variances, is used to test for treatment differences. Satterthwaite's method for computing standard error of the mean of the difference is used.

Source: Reference Listings xx.x.x, xx.x.x


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.2.4.16

Number and Proportion of Subjects with Morning ItchRO(Obs) Severity Score ≤1 for >50% of Time Period ITT Population

| Post-Baseline | Primary | Cohort | PFIC ( | Cohort |
|---|---|---|---|---|
| Analysis Visit Time Period Category | Maralixibat<br>(N=xx) | Placebo<br>(N=xx) | Maralixibat<br>(N=xx) | Placebo<br>(N=xx) |
| Weeks 1-6<br>p-value vs. Placebo [1] | xx (xx.x%)<br>x.xxxx | xx (xx.x%) | xx (xx.x%)<br>x.xxxx | xx (xx.x%) |
| Weeks 7-10<br>p-value vs. Placebo [1] | xx (xx.x%)<br>x.xxxx | xx (xx.x%) | xx (xx.x%)<br>x.xxxx | xx (xx.x%) |
| Weeks 11-14<br>p-value vs. Placebo [1] | xx (xx.x%)<br>x.xxxx | xx (xx.x%) | xx (xx.x%)<br>x.xxxx | xx (xx.x%) |
| Weeks 15-18<br>p-value vs. Placebo [1] | xx (xx.x%)<br>x.xxxx | xx (xx.x%) | xx (xx.x%)<br>x.xxxx | xx (xx.x%) |
| Weeks 19-22<br>p-value vs. Placebo [1] | xx (xx.x%)<br>x.xxxx | xx (xx.x%) | xx (xx.x%)<br>x.xxxx | xx (xx.x%) |

(Continue for Time Periods: Weeks 23-26, and Weeks 15-26)

Note: Percentages are 100\*n/N. Days with missing data are <u>not</u> considered to have met the  $\le 1$  criteria for that day. In computing the % of time the score is  $\le 1$  within each time period for each subject, the denominator of the proportion includes all days within the specified time period (i.e., days with missing and non-missing data), while the numerator only includes those days that the score is 0 or 1.

 $[1] \ p\text{-values comparing maralixibat to placebo treatment groups are calculated using a Barnard's exact test.}$ 

Source: Reference Listings xx.x.x, xx.x.x


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.2.4.17.1.1
Change from Baseline in ItchRO(Obs) Frequency Score
Tabulation of Fitted Summary Statistics from MMRM
ITT Population – Primary Cohort

Programming Notes: Repeat Table 14.2.1.1

Programming Notes: Repeat Table 14.2.1.2

Table 14.2.4.17.2.1
Change from Baseline in ItchRO(Obs) Frequency Score
Tabulation of Fitted Summary Statistics from MMRM
ITT Population – PFIC Cohort

#### Programming Notes: Repeat Table 14.2.1.1; change footnote [1] to:

[1] Estimates are from a mixed model for repeated measures (MMRM) with change from baseline as the dependent variable and fixed categorical effects of treatment group, time period and treatment-by-time period interaction as well as the continuous fixed covariates of average baseline score, baseline score-by-time period interaction, and PFIC type.

Programming Notes: Repeat Table 14.2.1.2, but add a data row as the last row: "PFIC Type (Covariate)" and add in the p-values from the model


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.2.4.18.1.1
Change from Baseline in ItchRO(Pt) Severity Score
Tabulation of Fitted Summary Statistics from MMRM
ITT Population – Primary Cohort

Programming Notes: Repeat Table 14.2.1.1

Table 14.2.4.18.1.2
Change from Baseline in ItchRO(Pt) Severity Score
MMRM Model Effects
ITT Population – Primary Cohort

Programming Notes: Repeat Table 14.2.1.2

Table 14.2.4.18.2.1 Change from Baseline in ItchRO(Pt) Severity Score Tabulation of Fitted Summary Statistics from MMRM ITT Population – PFIC Cohort

#### Programming Notes: Repeat Table 14.2.1.1; change footnote [1] to:

[1] Estimates are from a mixed model for repeated measures (MMRM) with change from baseline as the dependent variable and fixed categorical effects of treatment group, time period and treatment-by-time period interaction as well as the continuous fixed covariates of average baseline score, baseline score-by-time period interaction, and PFIC type.

Table 14.2.4.18.2.2
Change from Baseline in ItchRO(Pt) Severity Score
MMRM Model Effects
ITT Population – PFIC Cohort

Programming Notes: Repeat Table 14.2.1.2, but add a data row as the last row: "PFIC Type (Covariate)" and add in the p-values from the model


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.2.4.19.1.1
Change from Baseline in ItchRO(Pt) Frequency Score
Tabulation of Fitted Summary Statistics from MMRM
ITT Population – Primary Cohort

Programming Notes: Repeat Table 14.2.1.1

Programming Notes: Repeat Table 14.2.1.2

Table 14.2.4.19.2.1
Change from Baseline in ItchRO(Pt) Frequency Score
Tabulation of Fitted Summary Statistics from MMRM
ITT Population – PFIC Cohort

#### Programming Notes: Repeat Table 14.2.1.1; change footnote [1] to:

[1] Estimates are from a mixed model for repeated measures (MMRM) with change from baseline as the dependent variable and fixed categorical effects of treatment group, time period and treatment-by-time period interaction as well as the continuous fixed covariates of average baseline score, baseline score-by-time period interaction, and PFIC type.

Table 14.2.4.19.2.2
Change from Baseline in ItchRO(Pt) Frequency Score
MMRM Model Effects
ITT Population – PFIC Cohort

Programming Notes: Repeat Table 14.2.1.2, but add a data row as the last row: "PFIC Type (Covariate)" and add in the p-values from the model


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



#### Table 14.2.4.20.1

Change from Baseline in Clinician Scratch Scale (CSS) Tabulation of Fitted Summary Statistics from MMRM ITT Population

#### Programming Notes: Repeat Table 14.2.2.2.1, adding Week 4; add Note:

Note: The CSS provides an assessment of itch severity. The clinician's assessment of the subject's pruritus will focus on scratching and visible damage to the skin as a result of scratching as observed by the physician. The CSS uses a 5-point scale, in which 0 designates no evidence of scratching and 4 designates cutaneous mutilation with bleeding, hemorrhage and scarring.

Table 14.2.4.20.2 Change from Baseline in Clinician Scratch Scale (CSS) MMRM Model Effects ITT Population

Programming Notes: Repeat Table 14.2.2.2.2

Table 14.2.4.21.1

Change from Baseline in Caregiver Impression of Severity (CIS)
Tabulation of Fitted Summary Statistics from MMRM
ITT Population

#### Programming Notes: Repeat Table 14.2.2.2.1, replacing Week 2 with Week 4; add Note:

Note: The CIS is designed to assess the caregiver's perception of itch severity of their child, using a 5-point scale, in which 0 designates no itch and 4 designates very severe itch. The questionnaire is administered with a recall period of 1 week.

Table 14.2.4.21.2
Change from Baseline in Caregiver Impression of Severity (CIS)
MMRM Model Effects
ITT Population

Programming Notes: Repeat Table 14.2.2.2.2


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



# Table 14.2.4.22.1 Change from Baseline in Patient Impression of Severity (PIS) Tabulation of Fitted Summary Statistics from MMRM ITT Population

### Programming Notes: Repeat Table 14.2.2.2.1, replacing Week 2 with Week 4; add Note:

Note: Subjects aged ≥9 years self-complete the PIS questionnaire. The PIS is designed to assess the subject's perception of their itch severity using a 5-point scale, in which 0 designates not feeling itchy at all and 4 designates feeling very, very itchy. The questionnaire is administered with a recall period of 1 week.

Table 14.2.4.22.2
Change from Baseline in Patient Impression of Severity (PIS)
MMRM Model Effects
ITT Population

Programming Notes: Repeat Table 14.2.2.2.2


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



#### For next 6 EDQ(Obs) tables, add 'Abbreviations: EDQ(Obs) = Exploratory Diary Questionnaire (Observer)'

Table 14.2.4.23.1.1
Change from Baseline in EDQ(Obs) Severity Score
Tabulation of Fitted Summary Statistics from MMRM
ITT Population – Primary Cohort

Programming Notes: Repeat Table 14.2.1.1; add following Note:

Note: Caregivers for all subjects aged <9 years complete the EDQ(Obs) instrument.

Table 14.2.4.23.1.2
Change from Baseline in EDQ(Obs) Severity Score
MMRM Model Effects
ITT Population – Primary Cohort

Programming Notes: Repeat Table 14.2.1.2

Table 14.2.4.23.2.1
Change from Baseline in EDQ(Obs) Severity Score
Tabulation of Fitted Summary Statistics from MMRM
ITT Population – PFIC Cohort

#### Programming Notes: Repeat Table 14.2.1.1; add Note and change footnote [1] to:

Note: Caregivers for all subjects aged <9 years complete the EDQ(Obs) instrument.

[1] Estimates are from a mixed model for repeated measures (MMRM) with change from baseline as the dependent variable and fixed categorical effects of treatment group, time period and treatment-by-time period interaction as well as the continuous fixed covariates of average baseline score, baseline score-by-time period interaction, and PFIC type.


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.2.4.23.2.2
Change from Baseline in EDQ(Obs) Severity Score
MMRM Model Effects
ITT Population – PFIC Cohort

Programming Notes: Repeat Table 14.2.1.2, but add a data row as the last row: "PFIC Type (Covariate)" and add in the p-values from the model

Table 14.2.4.24.1
Change from Baseline in Morning EDQ(Obs) Sleep Disturbance Score
Tabulation of Fitted Summary Statistics from MMRM
ITT Population

Programming Notes: Repeat Table 14.2.2.2.1, except use time periods as in Table 14.2.1.1, including updating 1st column header; add Note and update footnotes [1] and [2] to:

Note: Caregivers for all subjects aged <9 years complete the EDQ(Obs) instrument. Sleep disturbance is scored in the morning using a 5-point scale, in which 1 designates because of itch my child never had trouble staying asleep and 5 designates because of itch my child almost always has trouble staying asleep.

- [1] Estimates are from a mixed model for repeated measures (MMRM) with change from baseline as the dependent variable and fixed categorical effects of treatment group, time period and treatment-by-time period interaction as well as the continuous fixed covariates of average baseline score, and baseline score-by-time period interaction. For the PFIC Cohort, PFIC Type is included in the model as an additional covariate.
- [2] Average of time periods Weeks 15-18, 19-22, and 23-26 obtained from the MMRM as an equally weighted average of the 3 individual visit-specific estimates.

Table 14.2.4.24.2
Change from Baseline in Morning EDQ(Obs) Sleep Disturbance Score
MMRM Model Effects
ITT Population

Programming Notes: Repeat Table 14.2.2.2.2; change 'Time Point (Analysis Visit)' in 2<sup>nd</sup> data row to 'Time Period', and 'Time Period' in data rows 3 and 5 to 'Time Period'


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.2.4.25

Number and Proportion of Subjects with Improvement from Baseline in Morning EDQ(Obs) Sleep Disturbance Score
ITT Population

| Post-Baseline | Primary | Cohort | PFIC C | Cohort |
|---|---|---|---|---|
| Analysis Visit Time Period<br>Category | Maralixibat<br>(N=xx) | Placebo<br>(N=xx) | Maralixibat<br>(N=xx) | Placebo<br>(N=xx) |
| Weeks 1-6<br>p-value vs. Placebo [1] | xx (xx.x%)<br>x.xxxx | xx (xx.x%) | xx (xx.x%)<br>x.xxxx | xx (xx.x%) |
| Weeks 7-10<br>p-value vs. Placebo [1] | xx (xx.x%)<br>x.xxxx | xx (xx.x%) | xx (xx.x%)<br>x.xxxx | xx (xx.x%) |
| Weeks 11-14<br>p-value vs. Placebo [1] | xx (xx.x%)<br>x.xxxx | xx (xx.x%) | xx (xx.x%)<br>x.xxxx | xx (xx.x%) |
| Weeks 15-18<br>p-value vs. Placebo [1] | xx (xx.x%)<br>x.xxxx | xx (xx.x%) | xx (xx.x%)<br>x.xxxx | xx (xx.x%) |
| Weeks 19-22<br>p-value vs. Placebo [1] | xx (xx.x%)<br>x.xxxx | xx (xx.x%) | xx (xx.x%)<br>x.xxxx | xx (xx.x%) |

(Continue for Time Period: Weeks 23-26)

Abbreviations: EDQ(Obs) = Exploratory Diary Questionnaire (Observer)

Note: Percentages are 100\*n/N. Caregivers for all subjects aged <9 years complete the EDQ(Obs) instrument. Sleep disturbance is scored in the morning using a 5-point scale, in which 1 designates because of itch my child never had trouble staying asleep and 5 designates because of itch my child almost always has trouble staying asleep. Improvement is defined as a change from baseline <0, using 4- or 6-week (for the first time period) average scores. A subject is defined as having no improvement (i.e., non-responder) for an analysis visit time period if the 4-week average baseline score is missing OR the average sleep score at the analysis visit is missing.

[1] p-values comparing maralixibat to placebo treatment groups are calculated using a Barnard's exact test.

Source: Reference Listings xx.x.x, xx.x.x


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.2.4.26

Number and Proportion of Subjects with Morning EDQ(Obs) Sleep Disturbance Scores ≤2 from Post-Baseline through Week 26 ITT Population

| Post-Baseline | Primary | Cohort | PFIC Cohort | |
|---|---|---|---|---|
| Analysis Visit Time Period Category | Maralixibat<br>(N=xx) | Placebo<br>(N=xx) | Maralixibat<br>(N=xx) | Placebo<br>(N=xx) |
| Weeks 1-26<br>p-value vs. Placebo [1] | xx (xx.x%)<br>x.xxxx | xx (xx.x%) | xx (xx.x%)<br>x.xxxx | xx (xx.x%) |

Abbreviations: EDQ(Obs) = Exploratory Diary Questionnaire (Observer)

Note: Percentages are 100\*n/N. Caregivers for all subjects aged <9 years complete the EDQ(Obs) instrument. Sleep disturbance is scored in the morning using a 5-point scale, in which 1 designates because of itch my child never had trouble staying asleep and 5 designates because of itch my child almost always has trouble staying asleep. Missing scores are treated as a non-responder (i.e., score >2).

[1] p-values comparing maralixibat to placebo treatment groups are calculated using a Barnard's exact test.

Source: Reference Listings xx.x.x, xx.x.x


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.2.4.27.1
Change from Baseline in PedsQL Total Scale Score
Tabulation of Fitted Summary Statistics from MMRM
ITT Population

Programming Notes: Repeat Table 14.2.2.2.1, removing Week 2 and adding Week 4; add Abbreviations and Note:

Abbreviations: PedsQL = Pediatric Quality of Life Inventory

Note: PedsQL individual item scores (0-4 scale) are reverse-scored and linearly transformed to a 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0), so that higher scores indicate better HRQoL (less negative impact). If >50% of the items in the scale are missing, the scale score is not computed.

Table 14.2.4.27.2
Change from Baseline in PedsQL Total Scale Score
MMRM Model Effects
ITT Population

Programming Notes: Repeat Table 14.2.2.2.2; add Abbreviations:

Abbreviations: PedsQL = Pediatric Quality of Life Inventory


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



# Table 14.2.4.28.1 Change from Baseline in Height z-Score Tabulation of Fitted Summary Statistics from MMRM ITT Population

#### Programming Notes: Repeat Table 14.2.2.2.1, adding Week 4; add Note:

Note: z-scores are based on a subject's sex and age at each analysis visit. For subjects less than 24 months of age, the World Health Organization (WHO) growth charts are used to derive z-scores. For subjects at least 24 months of age, the Center for Disease Control (CDC) growth charts are used to derive z-scores.

Table 14.2.4.28.2
Change from Baseline in Height z-Score
MMRM Model Effects
ITT Population

Programming Notes: Repeat Table 14.2.2.2.2

Table 14.2.4.29.1
Change from Baseline in Weight z-Score
Tabulation of Fitted Summary Statistics from MMRM
ITT Population

#### Programming Notes: Repeat Table 14.2.2.2.1, adding Week 4; add Note:

Note: z-scores are based on a subject's sex and age at each analysis visit. For subjects less than 24 months of age, the World Health Organization (WHO) growth charts are used to derive z-scores. For subjects at least 24 months of age, the Center for Disease Control (CDC) growth charts are used to derive z-scores.

Table 14.2.4.29.2
Change from Baseline in Weight z-Score
MMRM Model Effects
ITT Population

Programming Notes: Repeat Table 14.2.2.2.2


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



# Table 14.2.4.30.1 Percent Change from Baseline in Total sBA Tabulation of Fitted Summary Statistics from MMRM ITT Population

Programming Notes: Repeat Table 14.2.2.2.1, changing 'CFB' to '% CFB' in 1st column

Table 14.2.4.30.2
Percent Change from Baseline in Total sBA
MMRM Model Effects
ITT Population

Programming Notes: Repeat Table 14.2.2.2.2

Table 14.2.4.31.1
Change from Baseline in 7 Alpha-hydroxy-4-cholesten-3-one (C4), ng/mL
Tabulation of Fitted Summary Statistics from MMRM
ITT Population

Programming Notes: Repeat Table 14.2.2.2.1, removing Weeks 2, 14, and 22; change footnote [2] to:

[2] Average of Weeks 18 and 26 obtained from the MMRM as an equally weighted average of the 2 individual visit-specific estimates.

Table 14.2.4.31.2
Change from Baseline in 7 Alpha-hydroxy-4-cholesten-3-one (C4), ng/mL
MMRM Model Effects
ITT Population

Programming Notes: Repeat Table 14.2.2.2.2


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.2.4.32.1
Change from Baseline in Fibroblast Growth Factor 19 (pg/mL)
Tabulation of Fitted Summary Statistics from MMRM
ITT Population

Programming Notes: Repeat Table 14.2.2.2.1, removing Weeks 2, 14, and 22; add 'Note: For analysis, one-half of the lower limit of quantitation (LLOQ=10.0 pg/mL) is used for values reported as <LLOQ.'; and change footnote [2] to:

[2] Average of Weeks 18 and 26 obtained from the MMRM as an equally weighted average of the 2 individual visit-specific estimates.

Table 14.2.4.32.2
Change from Baseline in Fibroblast Growth Factor 19 (pg/mL)
MMRM Model Effects
ITT Population

Programming Notes: Repeat Table 14.2.2.2.2

Table 14.2.4.33.1
Change from Baseline in Autotaxin (ng/mL)
Tabulation of Fitted Summary Statistics from MMRM
ITT Population

Programming Notes: Repeat Table 14.2.2.2.1, removing Weeks 2, 14, and 22; change footnote [2] to:

[2] Average of Weeks 18 and 26 obtained from the MMRM as an equally weighted average of the 2 individual visit-specific estimates.

Table 14.2.4.33.2 Change from Baseline in Autotaxin (ng/mL) MMRM Model Effects ITT Population

Programming Notes: Repeat Table 14.2.2.2.2


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.2.4.34.1 Change from Baseline in Albumin (g/dL) Tabulation of Fitted Summary Statistics from MMRM **ITT Population** 

Programming Notes: Repeat Table 14.2.2.2.1

Table 14.2.4.34.2 Change from Baseline in Albumin (g/dL) MMRM Model Effects ITT Population

Programming Notes: Repeat Table 14.2.2.2.2


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.2.4.35
Time to First Liver-Associated Event (Days)
ITT Population

| | Primary | Cohort | PFIC Cohort | |
|---|---|---|---|---|
| Kaplan-Meier | Maralixibat | Placebo | Maralixibat | Placebo<br>(N=xx) |
| Estimates [1] | (N=xx) | (N=xx) | (N=xx) | |
| Number of Events (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Number Censored (%) [2] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 25 <sup>th</sup> Percentile | xx.x | xx.x | XX.X | xx.x |
| 95% CI for 25 <sup>th</sup> Percentile) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| Median | xx.x | xx.x | xx.x | xx.x |
| 95% CI for Median) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| 75 <sup>th</sup> Percentile | xx.x | xx.x | xx.x | xx.x |
| (95% CI for 75 <sup>th</sup> Percentile) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| p-value [3] | x.xxxx | | x.xxxx | |
| p-value [4] | x.xxxx | | x.xxxx | |

Abbreviations: CI = confidence interval

Note: Liver-associated events include partial external biliary diversion (PEBD) surgery, listing for liver transplantation, liver decompensation (i.e., hepatic encephalopathy, variceal bleeding, ascites, and spontaneous bacterial peritonitis) events, hepatocellular carcinoma (HCC), and death.

- [1] Estimates calculated using Kaplan-Meier product-limit survival curve methodology. Missing estimates are due to insufficient events.
- [2] If a subject does not report a liver-associated event, then the time to first liver-associated event is censored at the last contact date.
- [3] p-value from a log-rank test, comparing maralixibat versus placebo.
- [4] p-value from a Wilcoxon test, comparing maralixibat versus placebo.

Source: Reference Listing xx.x.x


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.3.1 Maralixibat Exposure Safety Population

| Variable | Primary Cohort | PFIC Cohort | All Subjects |
|---|---|---|---|
| Statistic | (N=xx) | (N=xx) | (N=xx) |
| Average Daily Dose (μg/kg/day) | | | |
| n | xx | xx | XX |
| Mean | xx.x | xx.x | XX.X |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | xx.x | xx.x | XX.X |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx |
| Total Dose (μg/kg) | | | |
| n | xx | xx | XX |
| Mean | xx.x | xx.x | xx.x |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | xx.x | xx.x | XX.X |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx |
| Treatment Duration (days) | | | |
| n | xx | xx | XX |
| Mean | xx.x | xx.x | xx.x |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | xx.x | xx.x | XX.X |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx |

[ Continue for: Treatment Exposure (days) ]

Abbreviations: SD = standard deviation; SE = standard error of the mean; Q1 = 25<sup>th</sup> percentile; Q3 = 75<sup>th</sup> percentile Note: Only subjects exposed to Maralixibat are included. Treatment duration (days) = Date of last dose of study drug – Date of first dose of study drug + 1 day. For subjects that are missing the date of last dose of study drug, the last known contact date is used to calculate treatment duration. Treatment exposure (days) = Treatment duration in days – Number of days both morning and evening doses were missed. Source: Reference Listings xx.x.x, xx.x.x


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.3.2.1.1

Overall Summary of Treatment-Emergent Adverse Events
Safety Population

| | Primary | Cohort | PFIC C | ohort | All Subjects | |
|---|---|---|---|---|---|---|
| Subjects with at Least One Treatment-Emergent: | Maralixibat<br>(N=xx) | Placebo<br>(N=xx) | Maralixibat<br>(N=xx) | Placebo<br>(N=xx) | Maralixibat<br>(N=xx) | Placebo<br>(N=xx) |
| Adverse Event | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Adverse Event Categorized as Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Adverse Event Related to Study Drug | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Adverse Event Categorized as Severe and Related to Study Drug | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Serious Adverse Event | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Serious Adverse Event Related to Study Drug | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Adverse Event Leading to Permanent Study Drug Discontinuation | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| Adverse Event Leading to Death | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |

Note: Percentages are 100\*n/N. AEs are coded using MedDRA Version 22.1. Subjects who reported more than one adverse event (AE) within each category were only counted once. A treatment-emergent AE (TEAE) is defined as an AE that starts or deteriorates on or after the first dose of study drug and no later than 7 days following the last dose of study drug (for subjects not participating in the extension study) or reported through the Week 26/EOT visit (for subjects participating in the extension study). For subjects with > 7 days of study drug interruption/withdrawal, the definition of a TEAE considers both the date of the last dose prior to drug interruption and the actual last dose.

Source: Reference Listing xx.x.x




Sponsor: Mirum Pharmaceuticals Inc.

Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



### Table 14.3.2.1.2 Overall Summary of Treatment-Emergent Adverse Events by Age Group Safety Population

Age Group: 1 to <6 years

| | Primary | Cohort | PFIC C | ohort | All Sul | ojects |
|---|---|---|---|---|---|---|
| | Maralixibat | Placebo | Maralixibat | Placebo | Maralixibat | Placebo |
| Subjects with at Least One Treatment-Emergent: | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Adverse Event | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Adverse Event Categorized as Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Adverse Event Related to Study Drug | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Adverse Event Categorized as Severe and Related to Study Drug | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| Serious Adverse Event | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| Serious Adverse Event Related to Study Drug | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| Adverse Event Leading to Permanent Study Drug Discontinuation | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| Adverse Event Leading to Death | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |

Note: Percentages are 100\*n/N. AEs are coded using MedDRA Version 22.1. Subjects who reported more than one adverse event (AE) within each category were only counted once. A treatment-emergent AE (TEAE) is defined as an AE that starts or deteriorates on or after the first dose of study drug and no later than 7 days following the last dose of study drug (for subjects not participating in the extension study) or reported through the Week 26/EOT visit (for subjects participating in the extension study). For subjects with > 7 days of study drug interruption/withdrawal, the definition of a TEAE considers both the date of the last dose prior to drug interruption and the actual last dose.

Source: Reference Listing xx.x.x

Programming Note: Repeat table for the other 2 age groups: '6 to <13 years' and '13 to 18 years'; N should be the total # of subjects in each age group, cohort, and treatment group


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



## Table 14.3.2.1.3 Overall Summary of Treatment-Emergent Adverse Events by Sex Safety Population

Programming Note: Same shell as Table 14.3.2.1.2, replacing 'Age Group: xxxxx' at top of table with 'Sex: xxxx', repeating table for each sex (Male, Female))

Table 14.3.2.1.4

Overall Summary of Treatment-Emergent Adverse Events by Race
Safety Population

Programming Note: Same shell as Table 14.3.2.1.2, replacing 'Age Group: xxxxx' at top of table with 'Race: xxxx', repeating table for each race (American Indian or Alaska Native, Asian, Black or African American, White, More than one race, and Not Reported)


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



## Table 14.3.2.2.1 Incidence of Treatment-Emergent Adverse Events Safety Population

| | Primary | Cohort | PFIC ( | Cohort | All Subjects | |
|---|---|---|---|---|---|---|
| System Organ Class<br>Preferred Term | Maralixibat<br>(N=xx) | | | Placebo<br>(N=xx) | Maralixibat<br>(N=xx) | Placebo<br>(N=xx) |
| Number of Subjects with at Least One TEAE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| System Organ Class #1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Term #1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Term #2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Term #3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| System Organ Class #2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Term #1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Term #2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Term #3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

•••

Note: Percentages are 100\*n/N. AEs are coded using MedDRA Version 22.1. At each level of summarization (System Organ Class and Preferred Term), subjects who reported more than one adverse event (AE) were only counted once.

Source: Reference Listing xx.x.x

Programming Note: SOC and PT are sorted alphabetically by SOC and descending frequency of PT within each SOC


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



## Table 14.3.2.2.2 Incidence of Treatment-Emergent Adverse Events by Age Group Safety Population

Age Group: 1 to <6 years

| | Primary | Cohort | PFIC C | Cohort | All Subjects | |
|---|---|---|---|---|---|---|
| System Organ Class<br>Preferred Term | Maralixibat<br>(N=xx) | Placebo<br>(N=xx) | Maralixibat<br>(N=xx) | Placebo<br>(N=xx) | Maralixibat<br>(N=xx) | Placebo<br>(N=xx) |
| Number (%) of Subjects with at Least One TEAE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| System Organ Class #1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Term #1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Term #2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Term #3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| System Organ Class #2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Term #1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Term #2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Term #3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

...

Note: Percentages are 100\*n/N. AEs are coded using MedDRA Version 22.1. At each level of summarization (System Organ Class and Preferred Term), subjects who reported more than one adverse event (AE) were only counted once.

Source: Reference Listing xx.x.x

Programming Note: Repeat table for the other 2 age groups: '6 to <13 years' and '13 to 18 years'. N should be the total # of subjects in each age group, cohort, and treatment group.

SOC and PT are sorted alphabetically by SOC and descending frequency of PT within each SOC.


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



## Table 14.3.2.2.3 Incidence of Treatment-Emergent Adverse Events by Sex Safety Population

Programming Note: Same shell as Table 14.3.2.2.2, replacing 'Age Group: xxxxx' at top of table with 'Sex: xxxx', repeating table for each sex (Male, Female)

Table 14.3.2.2.4
Incidence of Treatment-Emergent Adverse Events by Race
Safety Population

Programming Note: Same shell as Table 14.3.2.2.2, replacing 'Age Group: xxxxx' at top of table with 'Race: xxxx', repeating table for each race (American Indian or Alaska Native, Asian, Black or African American, White, More than one race, and Not Reported)

Table 14.3.3.1
Incidence of Treatment-Emergent Serious Adverse Events
Safety Population

Programming Note: Same shell as Table 14.3.2.2.1

Table 14.3.3.2 Incidence of Treatment Related Adverse Events Safety Population

Programming Note: Same shell as Table 14.3.2.2.1

Table 14.3.3.3
Incidence of Treatment Related Adverse Events Leading to Permanent Discontinuation of Study Drug
Safety Population

Programming Note: Same shell as Table 14.3.2.2.1


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.3.3.4.1 Incidence of Events of Clinical Interest - Diarrhoea Events Safety Population

Programming Note: Same shell as 14.3.2.2.1, adding at end of Note: "Refer to SAP Sec. 6.1.9 for the preferred terms included in the definition of each event of clinical interest."

> Table 14.3.3.4.2 Incidence of Events of Clinical Interest – LSV Deficiency Events Safety Population

Programming Note: Same shell as 14.3.2.2.1, adding at end of Note: "Refer to SAP Sec. 6.1.9 for the preferred terms included in the definition of each event of clinical interest."

> Table 14.3.3.4.3 Incidence of Events of Clinical Interest – Elevated Transaminases Safety Population

Programming Note: Same shell as 14.3.2.2.1, adding at end of Note: "Refer to SAP Sec. 6.1.9 for the preferred terms included in the definition of each event of clinical interest."

> Table 14.3.3.4.4 Incidence of Events of Clinical Interest – Elevated Bilirubin Safety Population

Programming Note: Same shell as 14.3.2.2.1, adding at end of Note: "Refer to SAP Sec. 6.1.9 for the preferred terms included in the definition of each event of clinical interest."




Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



### Table 14.3.4.1 Listing of Serious Adverse Events Safety Population

| Subject<br>ID | Cohort<br>[1] | Treatment<br>Received<br>[2] | System Organ Class/<br>Preferred Term/<br>Verbatim Term | TEAE? | Start Date<br>(Study Day) [3] | End Date<br>(Study Day) [3] | Event<br>Duration<br>(days) | Severity/<br>Relationship to<br>Study Drug | Outcome/<br>Study Drug<br>Action Taken | Serious?/Life<br>Threatening? | Treatment<br>Required |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXXXX | Primary | 600 | xxxxxxxxxx xxxxx xxxxx/<br>xxxxxxxxxxxxxxx | Yes | DDMMMYYYY<br>(xx) | DDMMMYYYY<br>(xx) | xx | Moderate/<br>Not Related | xxxxxxxx/<br>xxxx xxx xxxxxxx | Yes/<br>No | None |
| xxxxxx | PFIC | Placebo | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | No | DDMMMYYYY<br>(xx) | DDMMMYYYY<br>(xx) | xx | Severe/<br>Related | xxxxxxxx/<br>xxxx xxx xxxxxxx | Yes/<br>No | xxxx; xxxxx |

Note: AEs are coded using MedDRA Version 22.1. In determining treatment-emergent AEs (TEAEs) and study day, partial dates were imputed based on the SAP.

[3] Study Day is calculated relative to the date of the first dose of study drug.

Source: Reference Listing xx.x.x

**Programming Note:** Sort AEs (within subject) by start date and then by end date; events that are ongoing would be listed after those with end dates (for those events with the same start date). For Treatment Required column, concatenate treatment required (e.g., Medication; Hospitalization). If "Other" is answered, concatenate the specify (e.g., Medication; Other: change settings in hearing aid). If subject was never dosed, Study Day will be reported as "NT".


<sup>[1]</sup> Subject cohorts include Primary, PFIC, or Other. Subjects in the Primary Cohort, that are all a subset of the PFIC Cohort, are presented as 'Primary'.

<sup>[2]</sup> Treatment received at the start of the event, including dose (reported in units of µg/kg/day) for subjects on maralixibat. For AEs that started within 7 days after the last dose of study drug, the last treatment received is listed. For AEs that started >7 days after the last dose of study drug, treatment received is blank. NT = Not Treated (for AEs that started prior to 1st dose of study drug)

Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.3.4.2
Listing of Adverse Events Leading to Permanent Discontinuation of Study Drug
Safety Population

Programming Note: Same shell as Table 14.3.4.1

Table 14.3.4.3 Listing of Deaths Safety Population

Programming Note: Same shell as Table 14.3.4.1


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



### Table 14.3.5.1 Summary of Safety Laboratory Data: Chemistry Safety Population

< Lab Test (units) >

| | Primary Cohort | | | | PFIC Cohort | | | |
|---|---|---|---|---|---|---|---|---|
| Analysis Visit Statistic | Maralixibat (N=xx) | | Placebo (N=xx) | | Maralixibat (N=xx) | | Placebo (N=xx) | |
| | Obs | CFB | Obs | CFB | Obs | CFB | Obs | CFB |
| Baseline | х | | X | | x | | x | |
| n | xx | | xx | | xx | | xx | |
| Mean | xx.x | | xx.x | | xx.x | | xx.x | |
| (95% CI for Mean) | (xx.x, xx.x) | | (xx.x, xx.x) | | (xx.x, xx.x) | | (xx.x, xx.x) | |
| SD (SE) | xx.xx (xx.xx) | | xx.xx (xx.xx) | | xx.xx (xx.xx) | | xx.xx (xx.xx) | |
| Median | xx.x | | xx.x | | xx.x | | xx.x | |
| Q1, Q3 | xx.x, xx.x | | xx.x, xx.x | | xx.x, xx.x | | xx.x, xx | |
| Min, Max | xx, xx | | xx, xx | | xx, xx | | xx, xx | |
| Week 2 | x | Х | Х | x | x | x | x | Χ |
| N | xx | xx | xx | xx | xx | xx | XX | Xx |
| Mean | xx.x | xx.x | xx.x | xx.x | xx.x | XX.X | xx.x | xx.x |
| (95% CI for Mean) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x | XX.X | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |

(Continue for each planned analysis visit: Week 6, Week 10, Week 14, Week 18, Week 22, and Week 26)

Abbreviations: Obs = observed values; CFB = change from baseline; CI = confidence interval; SD = standard deviation; SE = standard error of the mean; Q1 = 25<sup>th</sup> percentile; Q3 = 75<sup>th</sup> percentile

Note: For analysis, one-half of the lower limit of quantitation (LLOQ) is used for values reported as <LLOQ.

- [1] Anion Gap (mEq/L) = sodium (mEq/L) chloride (mEq/L) bicarbonate (mEq/L)
- [2] Corrected Sodium (mEq/L) = sodium (mEq/L) +  $[0.002 \times triglycerides (mg/dL)]$
- [3] Calculated Osmolality (mOsm/kg) = [2 x (sodium (mEq/L) + potassium (mEq/L))] + [glucose (mg/dL) / 18] + [BUN (mg/dL) / 2.8]
- [4] Osmolar Gap (mOsm/kg) = measured osmolality (mOsm/kg) calculated osmolality (mOsm/kg)

SOURCE: Listing x.x.x.x

Programming Note: Repeat for each test in lab panel, left justified at top of table (as listed in SAP Appendix 1, under SAFETY LABS), noting footnotes required for derived labs; Min and Max values for the following derived labs should be rounded, for presentation purposes, as follows: Anion Gap [1] (1 decimal), Corrected Sodium [2] (integer), Calculated Osmolality [3] (integer), and Osmolar Gap [4] (integer)


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



### Table 14.3.5.2 Summary of Safety Laboratory Data: Hematology Safety Population

Programming Note: Same shell as Table 14.3.5.1, replacing footnotes with:

Abbreviations: Obs = observed values; CFB = change from baseline; CI = confidence interval; SD = standard deviation; SE = standard error of the mean; Q1 = 25<sup>th</sup>

percentile; Q3 = 75<sup>th</sup> percentile

Note: For analysis, one-half of the lower limit of quantitation (LLOQ) is used for values reported as <LLOQ.

SOURCE: Listing x.x.x.x

Programming Note (cont'd): Repeat for each test in lab panel, left justified at top of table (as listed in SAP Appendix 1, under SAFETY LABS)

Table 14.3.5.3

Summary of Safety Laboratory Data: Lipid Panel
Safety Population

Programming Note: Same shell as Table 14.3.5.1, replacing footnotes with:

Abbreviations: Obs = observed values; CFB = change from baseline; CI = confidence interval; SD = standard deviation; SE = standard error of the mean; Q1 = 25<sup>th</sup> percentile; Q3 = 75<sup>th</sup> percentile

Note: For analysis, one-half of the lower limit of quantitation (LLOQ) is used for values reported as <LLOQ.

SOURCE: Listing x.x.x.x

Programming Note (cont'd): Repeat for each test in lab panel, left justified at top of table (as listed in SAP Appendix 1, under SAFETY LABS, except for HDL-C which will only be presented in a subject listing)


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



### Table 14.3.5.4 Summary of Safety Laboratory Data: Lipid Soluble Vitamins (LSV) Safety Population

Programming Note: Same shell as Table 14.3.5.1, removing Week 2 except for INR, PT, and aPTT, and replacing footnotes with:

Abbreviations: Obs = observed values; CFB = change from baseline; CI = confidence interval; SD = standard deviation; SE = standard error of the mean; Q1 = 25<sup>th</sup> percentile; Q3 = 75<sup>th</sup> percentile

Note: For analysis, one-half of the lower limit of quantitation (LLOQ) is used for values reported as <LLOQ. For concentrations reported as above the upper limit of quantitation (ULOQ), the ULOQ is used as the analysis value.

[1] Ratio of Alpha Tocopherol to the sum of Cholesterol and Triglycerides (mg/g) = 1000 x alpha tocopherol (mg/dL) / [cholesterol (mg/dL) + triglycerides (mg/dL)]

[2] Retinol:RBP Molar Ratio (mol/mol) = 0.0734 x retinol (µg/dL) / RBP (mg/dL)

SOURCE: Listing x.x.x.x

Programming Note (cont'd): Repeat for each test in lab panel, left justified at top of table (as listed in SAP Appendix 1, under SAFETY LABS), noting footnotes required for derived labs; Min and Max values for the 2 derived labs should be rounded, for presentation purposes, to 2 decimal places

Table 14.3.5.5

Summary of Safety Laboratory Data: Alpha-Fetoprotein (ng/mL)

Safety Population

Programming Note: Same shell as Table 14.3.5.1 except remove 'Lab Test: xxxx' before table; only present Baseline, Week 10, and Week 26, and replace footnotes with:

Abbreviations: Obs = observed values; CFB = change from baseline; CI = confidence interval; SD = standard deviation; SE = standard error of the mean; Q1 = 25<sup>th</sup>

percentile; Q3 = 75<sup>th</sup> percentile

Note: For analysis, one-half of the lower limit of quantitation (LLOQ) is used for values reported as <LLOQ.

SOURCE: Listing x.x.x.x




Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4) PCN Number: MIRU8967 **premier** 

Table 14.3.5.6
Shift Table for Select Safety Laboratory Tests
Safety Population

| Lab Test (Unit)/ | | | | | Base | line | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Analysis Visit | | Mara | alixibat (N=xx) | | | Placebo (N=xx) | | | | |
| Post-Baseline | Below | Within | Above | Missing | Total | Below | Within | Above | Missing | Total |
| 25-Hydroxyvitamin D (ng/mL)<br>Week 6 | | | | | | | | | | |
| Below | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Within | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Above | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Total | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| (Continue for Weeks 10, 1 | 4, 18, 22, and 20 | 6) | | | | | | | | |
| Alpha Tocopherol (mg/dL) | | | | | | | | | | |
| Week 6 | | | | | | | | | | |
| Below | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Within | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| Above | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| Missing | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| Total | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |

(Continue for following lab tests: Prothrombin Intl. Normalized Ratio, and Vitamin A (µg/dL)

Note: For analysis, one-half of the lower limit of quantitation (LLOQ) is used for values reported as <LLOQ. For concentrations reported as above the upper limit of quantitation (ULOQ), the ULOQ is used as the analysis value.

Source: Reference Listing xx.x.x

Note to programmer: Repeat for 'PFIC Cohort'; start new page for each cohort and each lab test


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



## Table 14.3.6.1 Summary of Subject Height, Weight, and BMI z-Scores Safety Population

Programming Note: Same shell as Table 14.3.5.1 except change 'Lab Test: xxxx' to '<parameter> where parameter includes: Height z-score, Weight z-score, and BMI z-score; add Week 4, and replace footnotes with:

Abbreviations: Obs = observed values; CFB = change from baseline; CI = confidence interval; SD = standard deviation; SE = standard error of the mean; Q1 = 25<sup>th</sup> percentile; Q3 = 75<sup>th</sup> percentile

Note: z-scores are derived using a subject's age and sex. For subjects less than 24 months of age, WHO growth charts are used to derive z-scores. For subjects at least 24 months of age, CDC growth charts are used to derive z-scores.

SOURCE: Listing x.x.x.x

Table 14.3.6.2 Summary of Vital Signs Safety Population

Programming Note: Same shell as Table 14.3.5.1 except change 'Lab Test: xxxx' to '<parameter> where parameter includes: Systolic BP (mmHg), Diastolic BP (mmHg), Heart Rate (bpm), Respiratory Rate (breaths/min), and Body Temperature (°C); add Week 4, and replace footnotes with:

Abbreviations: Obs = observed values; CFB = change from baseline; CI = confidence interval; SD = standard deviation; SE = standard error of the mean; Q1 = 25<sup>th</sup>

percentile; Q3 = 75<sup>th</sup> percentile

SOURCE: Listing x.x.x.x

Table 14.3.6.3.1 Summary of Electrocardiogram Parameters Safety Population

Programming Note: Same shell as Table 14.3.5.1 except change 'Lab Test: xxxx' to '<parameter> where parameter includes: PR Interval (msec), QRS Duration (msec), QTcB Interval (msec), and QTcF Interval (msec); only include Baseline, Week 10, and Week 26, and replace footnotes with:

Abbreviations: Obs = observed values; CFB = change from baseline; CI = confidence interval; SD = standard deviation; SE = standard error of the mean; Q1 = 25<sup>th</sup> percentile; Q3 = 75<sup>th</sup> percentile; QTcB = QT interval corrected using Bazett's formula; QTcF = QT Interval corrected using Fridericia's formula SOURCE: Listing x.x.x.x


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.3.6.3.2
Summary of Electrocardiogram Interpretation
Safety Population

| | Primary | Cohort | PFIC ( | Cohort |
|----------------|-------------|------------|-------------|------------|
| Analysis Visit | Maralixibat | Placebo | Maralixibat | Placebo |
| Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Baseline | nn | nn | nn | nn |
| Abnormal – CS | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Abnormal – NCS | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Week 10 | nn | nn | nn | nn |
| Abnormal – CS | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Abnormal – NCS | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Week 26 | nn | nn | nn | nn |
| Abnormal – CS | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Abnormal – NCS | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Abbreviations: CS = Clinically Significant; NCS = Not Clinically Significant

Note: Percentages are 100\*n/Number of subjects with ECG interpretation data at each visit.

Source: Reference Listing xx.x.x

Programming Note: nn is # of subjects with non-missing ECG data




Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



## Table 14.3.7 Concomitant Medications/Therapies Safety Population

Programming Notes: Repeat Table 14.1.5 except for changing 'Prior' in 1st data row to 'Concomitant', and footnotes as below

Note: Percentages are 100\*n/N.

[1] Medications were coded using World Health Organization Drug Dictionary (WHO-DD Enhanced version September 2019) ATC level 2 and Chemical Substance (generic name). Subjects were counted only once for each Anatomical Therapeutic Chemical (ATC) or Preferred Term. Any treatments continuing or starting after the first dose of study drug will be considered concomitant. If a treatment started prior to the first dose of study drug and continues after the first dose of study drug, it was considered both prior and concomitant.

Source: Reference Listings xx.x.x, xx.x.x


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.4.1 Summary of Healthcare Utilization Measures Safety Population

| | Primary | Cohort | PFIC Co | ohort | All Sub | jects |
|---|---|---|---|---|---|---|
| Healthcare Utilization Measure<br>Statistic | Maralixibat<br>(N=xx) | Placebo<br>(N=xx) | Maralixibat<br>(N=xx) | Placebo<br>(N=xx) | Maralixibat<br>(N=xx) | Placebo<br>(N=xx) |
| Number of ER Visits [1] | | | | | | |
| Number and % of Subjects | xx (x.x%) | xx (x.x%) | xx (x.x%) | xx (x.x%) | xx (x.x%) | xx (x.x%) |
| Number of Occurrences | xx | xx | xx | xx | xx | xx |
| Number of PFIC-Related Hospitalizations [1] | | | | | | |
| Number and % of Subjects | xx (x.x%) | xx (x.x%) | xx (x.x%) | xx (x.x%) | xx (x.x%) | xx (x.x%) |
| Number of Occurrences | xx | xx | xx | xx | xx | xx |
| Length of Stay for Hospitalizations (days) [2] | | | | | | |
| Mean (SD) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) |
| Median | x.x | x.x | x.x | x.x | x.x | x.x |
| Min, Max | x, x | x, x | x, x | x, x | x, x | x, x |
| Number of Days Caregiver Missed Work Due to | | | | | | |
| Healthcare Resource Utilization Events [2] | | | | | | |
| Mean (SD) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) | x.x (x.xx) |
| Median | x.x | x.x | x.x | x.x | x.x | x.x |
| Min, Max | x, x | x, x | x, x | x, x | x, x | x, x |

Abbreviations: PFIC = progressive familial intrahepatic cholestasis; ER = emergency room; SD = standard deviation

Note: Percentages are 100\*n/N. Data are presented across the entire post-baseline study period, between clinic visits from baseline through Week 27 Follow-up. [1] Subjects that visit the Emergency Room and the visit results in the subject being admitted to the hospital will be counted in both the Number of Hospitalizations and the Number of ER Visits.

[2] For those subjects reporting PFIC-related hospitalizations, summary statistics on the number of days are presented.

Source: Reference Listing xx.x.x


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967



Table 14.4.2
Summary of Plasma Sample Maralixibat Concentrations (ng/mL)
Safety Population

| Analysis Visit | Primary | y Cohort | PFIC C | Cohort | All Sul | bjects |
|---|---|---|---|---|---|---|
| Sample Time Point | Maralixibat | Placebo | Maralixibat | Placebo | Maralixibat | Placebo |
| Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Week 10 | | | | | | |
| Pre-Dose | | | | | | |
| n | XX | XX | XX | XX | XX | xx |
| Mean | XX.X | xx.x | XX.X | XX.X | XX.X | xx.x |
| (95% CI for Mean) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| CV (%) | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Median | xx.x | xx.x | xx.x | XX.X | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Geometric Mean | xx.x | xx.x | xx.x | xx.x | xx.x | XX.X |
| Post-Dose | | | | | | |
| n | XX | XX | XX | XX | XX | xx |
| Mean | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| (95% CI for Mean) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| SD (SE) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| CV (%) | XX.X | xx.x | XX.X | XX.X | XX.X | xx.x |
| Median | XX.X | xx.x | XX.X | XX.X | XX.X | xx.x |
| Q1, Q3 | XX.X, XX.X | xx.x, xx.x | XX.X, XX.X | xx.x, xx.x | XX.X, XX.X | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Geometric Mean | XX.X | xx.x | xx.x | xx.x | XX.X | xx.x |

(Repeat for Analysis Visits: Week 14 and Week 26)

Abbreviations: CI = confidence interval; SD = standard deviation; SE = standard error of the mean; CV = coefficient of variation Note: The lower limit of quantitation (LLOQ) is 0.250 ng/mL. For any concentration reported below this limit, a zero value is used in the calculation of summary statistics. Post-dose samples were drawn approximately 2.5 hours after the morning dose.

Source: Reference Listing xx.x.x


Listing Shells Sponsor: Mirum Pharmaceuticals Inc. Protocol: Maralixibat-502 (Amendment 4) PCN Number: MIRU8967



| Sponsor | Mirum Pharmaceuticals Inc. |
|---|---|
| Protocol Title: | Randomized Double-blind Placebo-controlled Phase 3 Study to Evaluate the Efficacy and Safety of Maralixibat in the Treatment of Children with Progressive Familial Intrahepatic Cholestasis (PFIC) – MARCH-PFIC |
| Protocol Number: | MRX-502 (Amendment 4) |
| Premier Research PCN: | MIRU8967 |
| Document Author: | Taryn Robertson |
| Document Version: | Final 1.0 |
| Document Date: | 13Oct2022 |

PROGRAMMING NOTE FOR <u>ALL</u> LISTINGS (EXCEPT LISTING 16.2.2.1): Sort by Treatment (Maralixibat or Placebo), then PFIC Type (ordered according to the list below), then Subject ID (and Study Day, when applicable), placing Treatment in sub-title.

Present and sort by PFIC Type in the following order:

nt-PFIC2
PFIC3
PFIC4
PFIC6
nt-PFIC2-het
nt-PFIC2-IsBA
nt-PFIC2-surg
t-PFIC2
PFIC1-het
PFIC1-surg

No-variant-found

Analysis Visit is presented in addition to Clinic Visit for all data that is available in a single ADaM dataset (ie, not for subject profile listings which merge data from across multiple ADaM datasets).

| Listing 16.1.1 | Subject Profile: Select Labs and Itch/Scratch Scores |
|---|---|
| Listing 16.1.2 | Subject Profile: Pediatric Quality of Life Inventory – Total Scale and Summary Scores |
| Listing 16.1.3 | Subject Profile: Efficacy and Safety Labs (Serum Bile Acid, Lipids, Lipid Soluble Vitamins, and Coagulation) |
| Listing 16.1.4 | Subject Profile: Sodium and Lipid Soluble Vitamin Level Abnormalities |
| Listing 16.2.1 | Analysis Populations and Siblings |
| Listing 16.2.2.1 | Subject Disposition: Screen Failure Subjects Enrolled in Study |
| Listing 16.2.2.2 | Subject Disposition and Completion: Intent-to-Treat Population |
| Listing 16.2.3.1 | Randomized Subjects by Randomized Cohort and Phenotype |
| Listing 16.2.3.2 | Subjects Where Randomized Cohort Conflicts with PFIC Type |
| Listing 16.3.1 | Inclusion and Exclusion Criteria |
| Listing 16.3.2 | Important Protocol Deviations |
| Listing 16.4.1 | Demographics and Baseline Information |
| Listing 16.4.2 | Long-Term Follow-Up Informed Consent and Disease Progression |
| Listing 16.4.3 | Informed Consent |
| Listing 16.4.4 | Medical History |
| Listing 16.4.5 | Prior and Concomitant Medications/Therapies |
| Listing 16.5.1 | Liver Imaging |
| Listing 16.5.2 | Liver-Associated Events |
| Listing 16.5.3 | Liver Transplant List |
| Listing 16.6.1 | Study Drug Supplied and Compliance |
| Listing 16.6.2 | Study Drug Exposure |
| Listing 16.6.3 | Study Drug Accountability |
| Listing 16.7.1 | Total Serum Bile Acid |


Listing Shells Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4) PCN Number: MIRU8967

| Listin = 4.6.7.2 | Commun Dilla Antid College and a |
|---|---|
| Listing 16.7.2 | Serum Bile Acid Subspecies |
| Listing 16.7.3 | Clinician Scratch Score |
| Listing 16.7.4 | Itch Reported Outcomes (Subject and Caregiver) Average Morning and Evening Scores |
| Listing 16.7.5 | Exploratory Diary Questionnaire (Subject and Caregiver) Average Morning and Evening Scores |
| Listing 16.7.6.1 | PIC and CIC |
| Listing 16.7.6.2 | PIS and CIS |
| Listing 16.7.7 | Efficacy Laboratory Tests |
| Listing 16.7.8 | Height, Weight, and BMI z-Score |
| Listing 16.7.9 | Sleep Disturbance |
| Listing 16.8.1 | Adverse Events |
| Listing 16.8.2.1 | Adverse Events of Clinical Interest: Diarrhoea Events |
| Listing 16.8.2.2 | Adverse Events of Clinical Interest: Lipid Soluble Vitamin Deficiency Events |
| Listing 16.8.2.3 | Adverse Events of Clinical Interest: Elevated Transaminases Events |
| Listing 16.8.2.4 | Adverse Events of Clinical Interest: Elevated Bilirubin Events |
| Listing 16.8.3 | Treatment Related Adverse Events |
| Listing 16.8.4.1 | Serious Adverse Events |
| Listing 16.8.4.2 | Serious Related Adverse Events |
| Listing 16.8.5 | Adverse Events Leading to Study Drug Discontinuation |
| Listing 16.8.6 | Severe Adverse Events |
| Listing 16.8.7 | Adverse Events Resulting in Death |
| Listing 16.9.1 | Vital Signs |
| Listing 16.9.2 | Physical Examination |
| Listing 16.9.3 | 12-Lead Safety ECG |
| Listing 16.10.1 | Clinical Laboratory Tests: Clinical Chemistry |
| Listing 16.10.2 | Clinical Laboratory Tests: Hematology |
| Listing 16.10.3 | Clinical Laboratory Tests: Urinalysis |
| Listing 16.10.4 | Clinical Laboratory Tests: Lipid Soluble Vitamins |
| Listing 16.10.5 | Clinical Laboratory Tests: Lipid Panel |
| Listing 16.10.6 | Clinical Laboratory Tests: Hepatocellular Carcinoma Marker - Alpha-Fetoprotein (AFP) |
| Listing 16.10.7 | Clinical Laboratory Tests: Timing of Sample Collection and Last Meal |
| Listing 16.10.8 | Microbiology Tests |
| Listing 16.10.9 | Pregnancy Tests |
| Listing 16.10.10 | Plasma Sample Maralixibat Concentrations |
| Listing 16.11 | Telephone Contact Log |
| Listing 16.12 | Visit Dates and Type |
| Listing 16.13 | Healthcare Utilization |
| Listing 16.14 | COVID-19 Impact |

CONFIDENTIALPage 3 of 51

Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

## Listing 16.1.1 Subject Profile: Select Labs and Itch/Scratch Scores Safety Population

Treatment: <Maralixibat or Placebo>

| | | | | | | | | | | | | | | | | | PedsQL | Itc | hRO |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Age [1]/ | | Study | MRX | | | | Biliru | bin | | | PELD/ | | | CIC/ | | Parent | Morn | ing Avg. |
| PFIC | Sex/ | Analysis | Day | PFIC | sBA [4] | ALT | AST | (mg/ | dL) | C4 | ATX | MELD | | | PIC | | Total | Severity | Score [7] |
| Туре | Subject Country | Visit | [2] | Rcvd [3] | (umol/L) | (U/L) | (U/L) | Direct | Total | (ng/mL) | (ng/mL) | [5] | APRI | FIB-4 | [6] | CSS | Score | Obs [8] | Pt [9] |
| xxxxxx | xxxxxx x/x/xxx | Baseline<br>Week 2<br>Week 4 | -x<br>xx<br>xx | NT<br>300<br>600 | xx.x<br>xx.x b | xx<br>xx | xx<br>xx | x.x<br>x.x | x.x<br>x.x | xx.x<br>xx.x | xxxx<br>xxxx | xx<br>xx | x.x<br>x.x | xxx<br>xxx | x/x | x<br>x | xx.x<br>xx.x | x.xx w<br>[8] | x.xx<br>[8] |

#### Continue for all analysis visits

Abbreviations: sBA = serum Bile Acid; ALT = Alanine Aminotransferase; AST = Aspartate Aminotransferase; C4 = 7 alpha-hydroxy-4- cholesten-3-one (C4); ATX = Autotaxin; PELD = pediatric end-stage liver disease; MELD = model for end-stage liver disease; APRI = AST to platelet ratio index; FIB-4 = fibrosis-4; CIC = Caregiver Impression of Change; PIC = Patient Impression of Change; CSS = Clinician Scratch Scale; PedsQL = Pediatric Quality of Life; ItchRO = Itch Reported Outcome; ARG = Argentina; AUT = Austria; BEL = Belgium; BRA = Brazil; CAN = Canada; COL = Columbia; DEU = Germany; FRA = France; GBR = United Kingdom; ITA = Italy; LBN = Lebanon; MEX = Mexico; POL = Poland; SGP = Singapore; TUR = Turkey; USA = United States; Obs = Observer; Pt = Patient

- [1] Age (years) at Baseline.
- [2] Study Day is calculated relative to the date of the first dose of study drug.
- [3] Treatment received (MRX µg/kg BID) on the date of the assessment/sample collection or last MRX BID dose received if dose was missed or administered as QD. NT = not treated (pre-dose or Placebo dose)
- [4] 'b' indicates ≥ 75% reduction from baseline (ie, CFB ≤ -75%) OR sBA < 102 umol/L.
- [5] PELD is calculated for children < 12 years of age at the baseline visit; MELD is calculated for children ≥ 12 years of age at baseline.
- [6] PIC is completed by subjects who are at least 9 years of age.
- [7] ItchRO weekly scores calculated relative to first dose of study drug. For each post-baseline analysis visit, average score is calculated for the following periods: Week 1-6 (42 days), Weeks 7-10, 11-14, 15-18, 19-22, and 23-26. Average ItchRO score at baseline is calculated averaging the 4-weekly average scores before the first dose of study drug.
- [8] 'w' indicates average ItchRO score change from baseline  $\leq$  -1.0.
- [9] ItchRO self-report is completed by subjects who are at least 9 years of age.

Programming Note: Use data from ADaM.ADLB, ADQS. Use raw values; for example, <0.10, not analysis value.


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

## Listing 16.1.2 Subject Profile: Pediatric Quality of Life Inventory – Total Scale and Summary Scores Safety Population

Treatment: <Maralixibat or Placebo>

| PFIC | Age [1]/<br>Sex/ | Analysis | Study | Total<br>Sco | Scale<br>ore | Physical<br>Summar | | Psychosoc<br>Summai | | Multidim<br>Fatigue Sc | | Family<br>Impact<br>Total Scale | Parent<br>Functioning<br>Summary | Family<br>Impact<br>Summary |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Type | Subject Country | Visit | Day [2] | Parent | Child | Parent | Child | Parent | Child | Parent | Child | Score | Score | Score |
| xxxxxx | xxxxxx x/x/xxx | Baseline | -x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xxx.x |
| | | Week 4 | XX | xx.x | xx.x | XX.X | xx.x | XX.X | xx.x | xx.x | XX.X | xx.x | xx.x | xx.x |
| | | Week 6 | xx | xx.x | xx.x | XX.X | xx.x | xx.x | XX.X | xx.x | xx.x | xx.x | xx.x | xx.x |
| | | Week 10 | XX | xx.x | xx.x | XX.X | xx.x | XX.X | xx.x | xx.x | XX.X | xx.x | xx.x | xx.x |
| | | Week 14 | XX | xx.x | xx.x | XX.X | xx.x | XX.X | XX.X | xx.x | xx.x | xx.x | xx.x | xx.x |
| | | Week 18 | XX | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | XX.X | xx.x | xx.x | XX.X | xx.x |

(Continue for all analysis visits)

Abbreviations: ARG = Argentina; AUT = Austria; BEL = Belgium; BRA = Brazil; CAN = Canada; COL = Columbia; DEU = Germany; FRA = France; GBR = United Kingdom; ITA = Italy; LBN = Lebanon; MEX = Mexico; POL = Poland; SGP = Singapore; TUR = Turkey; USA = United States

Note: Pediatric Quality of Life (PedsQL) self-report is measured in subjects who are 5 to 18 years of age. Individual item scores (0-4 scale) are reverse-scored and linearly transformed to a 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0), so that higher scores indicate better HRQoL (less negative impact). Total scale and summary scores are computed as the average score. If more than 50% of the items in the scale are missing, the scale score is not computed. For scoring each total scale and summary score, refer to SAP.

- [1] Age (years) at Screening. The age-based questionnaires are based on age at screening.
- [2] Study Day is calculated relative to the date of the first dose of study drug.

**Programming Note:** Use data from ADaM.ADQS.


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

Listing 16.1.3

Subject Profile: Efficacy and Safety Labs (Serum Bile Acid, Lipids, Lipid Vitamins, and Coagulation)

Safety Population

Treatment: <Maralixibat or Placebo>

| | | Age [1]/ | | Study | | | Lipi | ds | | Lip | id Solub | le Vitami | ins | Coa | gulatio | n |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PFIC | | Sex/ | Analysis | Day | sBA [3] | CHOL | LDL | HDL | TG | VITD | VITA | VITE | RBP | aPTT | PT | |
| Туре | Subject | Country | Visit | [2] | (umol/L) | (mg/dL) | (mg/dL) | (mg/dL) | (mg/dL) | (ng/mL) | (μg/dL) | (mg/dL) | (mg/dL) | (sec) | (sec) | INR |
| xxxxx | xxxxx | x/x/xxx | Baseline | -x | xx.x | xxx | xxx | xx | xxx | xx.x | xx.x | x.xx | xx.xx | xx.x | xx.x | x.x |
| | | | Week 2 | xx | xx.x b | XXX | XXX | XX | XXX | xx.x | XX.X | x.xx | XX.XX | xx.x | xx.x | x.x |
| | | | Week 6 | xx | XX.X | XXX | XXX | XX | XXX | xx.x | XX.X | x.xx | XX.XX | xx.x | xx.x | x.x |
| | | | Week 10 | xx | XX.X | XXX | xxx | XX | XXX | xx.x | xx.x | x.xx | xx.xx | xx.x | xx.x | x.x |
| | | | Week 14 | xx | XX.X | XXX | xxx | XX | XXX | xx.x | xx.x | x.xx | xx.xx | xx.x | xx.x | x.x |
| | | ( | Continue for | all anal | lysis visits) | | | | | | | | | | | |

Abbreviations: sBA = Serum Bile Acid; CHOL = Cholesterol; LDL = LDL Cholesterol; HDL = HDL Cholesterol; TG = Triglycerides; VITD = 25-Hydroxyvitamin D; VITA = Vitamin A; VITE = Alpha Tocopherol; RBP = Retinol Binding Protein; aPTT = Activated Partial Thromboplastin Time; PT = Prothrombin Time; INR = International Normalized Ratio; ARG = Argentina; AUT = Austria; BEL = Belgium; BRA = Brazil; CAN = Canada; COL = Columbia; DEU = Germany; FRA = France; GBR = United Kingdom; ITA = Italy; LBN = Lebanon; MEX = Mexico; POL = Poland; SGP = Singapore; TUR = Turkey; USA = United States

- [1] Age (years) at Baseline.
- [2] Study Day is calculated relative to the date of the first dose of study drug.
- [3] 'b' indicates  $\geq$  75% reduction (ie, CFB  $\leq$  -75%) OR sBA < 102 umol/L.

Programming Note: Use data from ADaM.ADLB. Responder indicator needs to be added for sBA (see footnote 4). Add abbreviations to 'Note:' as needed for missing labs


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

## Listing 16.1.4 Subject Profile: Sodium and Lipid Soluble Vitamin Levels Safety Population

Treatment: <Maralixibat or Placebo>

| PFIC<br>Type | Subject | Age [1]/<br>Sex/<br>Country | Analysis<br>Visit | Study<br>Day [2] | VITD<br>(ng/ml) | VITA<br>(ug/dL) | VITE<br>(mg/dL) | Alpha<br>Tocopherol/<br>CHOL + TG<br>Ratio (mg/g)<br>[3] | RBP<br>(mg/dL) | Retinol:<br>RBP Molar<br>Ratio<br>(mol/mol) [4] | International<br>Normalized<br>Ratio | Sodium<br>(mEq/L) | Corrected<br>Sodium<br>(mEq/L)<br>[5] |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxxx | xxxxx | x/M/xxx | Baseline<br>Week 2<br>Week 4 | -x<br>xx<br>xxx | XX.X<br>XX.X<br>XX.X | xx.x<br>xx.x<br>xx.x | x.xx<br>x.xx<br>x.xx | x.xx<br>x.xx<br>x.xx | x.xx<br>x.xx<br>x.xx | x.xx<br>x.xx<br>x.xx | x.x<br>x.x<br>x.x | xxx<br>xxx<br>xxx | xxx<br>xxx<br>xxx |

#### (Continue for all analysis visits)

Abbreviations: ARG = Argentina; AUT = Austria; BEL = Belgium; BRA = Brazil; CAN = Canada; COL = Columbia; DEU = Germany; FRA = France; GBR = United Kingdom; ITA = Italy; LBN = Lebanon; MEX = Mexico; POL = Poland; SGP = Singapore; TUR = Turkey; USA = United States; VITD = 25-Hydroxyvitamin D; VITA = Vitamin A; VITE = Alpha Tocopherol; CHOL = Cholesterol; TG = Triglycerides; RBP = Retinol Binding Protein

- [1] Age (years) at Baseline.
- [2] Study Day is calculated relative to the date of the first dose of study drug.
- [3] Ratio (mg/g) = 1000 x alpha tocopherol (mg/dL) / [ cholesterol (mg/dL) + triglycerides (mg/dL)]. For alpha tocopherol concentrations reported as below the minimum quantitation limit (ie, 0.1 mg/dL), half of the minimum quantitation limit is used as the analysis value.
- [4] Molar Ratio (mol/mol) = 0.0734 x retinol (ug/dL) / RBP (mg/dL)
- [5] Corrected Sodium (mEq/L) = sodium (mEq/L) + [0.002 x triglycerides (mg/dL)]

**Programming Note:** Use data from ADaM.ADLB.


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

### Listing 16.2.1 Analysis Populations and Siblings All Subjects

Treatment: <Maralixibat or Placebo>

| PFIC | | Sibling in | Analy | | |
|--------|---------|------------|--------|-----|--------------|
| Туре | Subject | Study? [1] | Safety | ITT | Per-Protocol |
| xxxxxx | XXXXXX | | Yes | Yes | Yes |
| | XXXXXX | Yes | Yes | Yes | Yes |
| | XXXXXX | Yes | Yes | Yes | No |
| xxxxxx | xxxxxx | | Yes | Yes | No |

Abbreviation: ITT = Intent-to-Treat

Note: Safety population consists of all subjects who received at least 1 dose of study drug. ITT population consists of all randomized subjects. Per-protocol population consists of all subjects in the ITT population who receive at least 1 dose of study drug and do not have any important protocol violations or deviations that have a potential impact on the efficacy analysis.

[1] Siblings are assigned in a blinded manner to the same treatment arm. Each sibling is considered for the Safety, ITT, and Per-Protocol populations. One sibling within a family is considered for a sensitivity analysis on the primary and key secondary efficacy endpoints for the primary and PFIC cohorts in the ITT Population. The choice of sibling to use in the sensitivity analysis is made at random, unless only 1 sibling is evaluable in the specific cohort and ITT Population and the other sibling is not. In this case, the evaluable sibling will be used in sensitivity analyses.

**Programming Note:** Use data from ADaM.ADSL


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4) PCN Number: MIRU8967

### Listing 16.2.2.1 **Subject Disposition** Screen Failure Subjects Enrolled in Study

| Subject | Protocol<br>Criteria Version | Date<br>Screened | Screen Failure Reason |
|---|---|---|---|
| XXXXXX | Amendment 2 – 22NOV2019 | DDMMMYYYY | EXCLO8: XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| XXXXXX | xxxxxxxxxx | DDMMMYYYY | INCL02: XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| XXXXXX | xxxxxxxxxxx | DDMMMYYYY | OTHER: XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| XXXXXX | xxxxxxxxxxx | DDMMMYYYY | XXXXXX: XXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |

**Programming Note:** Only include subjects that were screen failures but were enrolled in the study, regardless of if the Sponsor granted a waiver. Use data from CRF.IE, CRF.SFR and CRF.STATFRM. For Screen Failure Reason, use CRF.IE.IENUM | | ': ' | | CRF.IE.IEREAS. If CRF.SFR.SFREAS = OTHER then Reason = CRF.SFR.SFREAS||': '||CRF.SFR.SFREASOT.

CONFIDENTIALPage 9 of 51

Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

### Listing 16.2.2.2 Subject Disposition and Completion Intent-to-Treat Population

Treatment: <Maralixibat or Placebo>

| | | | | | Date of | Specify | Enroll | | Tol. | | | Date of |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | Discon- | Reason for | in | Max | Min. | | Date of | Last Contact |
| PFIC | | Date | Date | | tinuation/ | Discontinuation | MRX | Dose | Dose?/ | Date of | Last Dose | (Study Day) |
| Type | Subject | Screened | Enrolled | Status | Completion | from Study | 503? | [1] | LTFU? | First Dose | (Study Day) | [2] |
| xxxxx | xxxxxx | DDMMMYYYY | DDMMMYYYY | Comp | DDMMMYYYY | | Yes | 600 | Yes/<br>Yes | DDMMMYYYY | DDMMMYYYY<br>(xx) | DDMMMYYYY<br>(xx) |
| | xxxxxx | DDMMMYYYY | DDMMMYYYY | Disc | DDMMMYYYY | xxxxxxxxxxx | No | 300 | Yes/<br>No | DDMMMYYYY | DDMMMYYYY<br>(xx) | DDMMMYYYY<br>(xx) |
| XXXX | xxxxxx | DDMMMYYYY | DDMMMYYYY | Disc | DDMMMYYYY | | No | 450 | Yes/<br>No | DDMMMYYYY | DDMMMYYYY<br>(xx) | DDMMMYYYY<br>(xx) |

Abbreviations: Comp = Completed; Disc = Discontinued; Max = Maximum; Tol. Min. Dose? = Did Subject Tolerate Minimum Drug Dose?; LTFU = Willing to provide Informed Consent and Assent as applicable for Long-Term Follow-Up Period?

Note: Study Day is calculated relative to the date of the first dose of study drug.

- [1] Maximum dose presented in units of µg/kg/day.
- [2] Completed only if subject is lost to follow-up.

**Programming Note:** If subject discontinues the study prematurely for Reason=AE, Physician Decision, Protocol Violation, Withdrawal of Consent, or Other, then Reason for d/c is DS.DSTERM concatenated with DS.DSREASSP (e.g., Other: Family Emergency). If DS.DSTERM = Death then Reason for d/c is DS.DSTERM concatenated with DS.DSDEATH. If subject discontinues the study due to Lost to follow-up then Reason=Lost to follow-up concatenated with the DS.DSLFCOMT field (e.g., Lost to follow-up: xxxxxxxxxxxxxxxxxxxx). Date of First Dose pulled from CRF.SDFD. Use data from CRF.DS, SDFD and STATFRM.


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

## Listing 16.2.3.1 Randomized Subjects by Randomized Cohort and Phenotype Intent-to-Treat Population

Treatment: <Maralixibat or Placebo>

| | | | | From [ | Dummy | Rand F | ile | | ype From<br>nent Log | An | alysis | | | Mutatio | า 1 | | Mutatio | n 2 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Random<br>ized<br>Phenotype | Mutation<br>e in Gene | | Treatment<br>Start Date | Rand.<br>Date | Rand.<br>Num. | Trtmt | Strata | At<br>Screen<br>ing | At<br>Random<br>ization | BSEP<br>Pheno. | PFIC<br>Type | BSEP<br>Pheno. | . cDNA | Protein | BSEP Zy | g. cDNA | Protein | BSEP Z | Other<br>g. Mutation |
| PFIC2 -<br>Primary<br>Cohort | ABCB11 | xxxxxx | DDMMYYYY | DDMMYYYY | XXXX | MRX | PFIC2 | PFIC2 -<br>Primary<br>Cohort | PFIC2 -<br>Primary<br>Cohort | BSEP 2 | nt-PFIC2 | nt | xxxxxxx | xxxxxxxx | BSEP2 HE | T xxxxxxx<br>xx | xxxxxxx<br>xx | k BSEP2 H | ĒΤ |
| | | xxxxxx | DDMMYYYY | DDMMYYYY | xxxx | MRX | PFIC2 | PFIC2 -<br>Supplem<br>ental<br>Cohort | PFIC2 -<br>Primary<br>Cohort | BSEP 2 | nt-PFIC2 | nt | xxxxxxx | XXXXXXXX<br>XXXXXXXX<br>XXXXXXXX<br>XX | | T xxxxxxxx<br>xxxxxxxx<br>xx | | k BSEP2 H | ΞT |
| | xxxxx | xxxxxx | DDMMYYYY | DDMMYYYY | xxxx | MRX | PFIC2 | PFIC2 -<br>Primary<br>Cohort | PFIC2 -<br>Primary<br>Cohort | | No-<br>variant-<br>found | NA | | | NA HO | M | | Н | DΜ |

Abbreviations: Rand = Randomization; Trtmt = Treatment; BSEP = bile salt excretion pump; Pheno = Phenotype; cDNA = complementary DNA; Zyg = Zygocity; t = truncated; nt = not truncated; HET = Heterozygous; HOM = Homozygous; NA = not applicable

Note: Sample is used to provide a full characterization and documentation of the mutation type in support of the diagnosis of PFIC. Mutation in Gene data is collected at Screening visit.

**Programming Note:** Use data from CRF.RAND, ADSL, CRF.CPGR.


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

## Listing 16.2.3.2 Subjects Where Randomized Cohort Conflicts with PFIC Type Intent-to-Treat Population

Treatment: <Maralixibat or Placebo>

| | | | | From [ | Dummy l | Rand F | ile | | ype From<br>nent Log | An | alysis | | | Mutatio | n 1 | | Mutatio | n 2 | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Random<br>ized<br>Phenotype | Mutation<br>in Gene | Subject | Treatment<br>Start Date | Rand.<br>Date | Rand.<br>Num. | Trtmt | Strata | At<br>Screen<br>ing | At<br>Random<br>ization | BSEP<br>Pheno. | PFIC<br>Type | BSEP<br>Pheno. | cDNA | Protein | BSEP Zyg. | cDNA | Protein | BSEP : | Zyg. | Other<br>Mutation |
| PFIC2 -<br>Primary<br>Cohort | ABCB11 | xxxxxx | DDMMYYYY | DDMMYYYY | xxxx | MRX | PFIC2 | PFIC2 -<br>Primary<br>Cohort | PFIC2 -<br>Primary<br>Cohort | BSEP 2 | nt-PFIC2 | nt | xxxxxxx | xxxxxxx | BSEP2 HET | xxxxxxxx | xxxxxxxx | BSEP2 | HET | |
| | | xxxxxx | DDMMYYYY | DDMMYYYY | xxxx | MRX | PFIC2 | PFIC2 -<br>Supplem<br>ental<br>Cohort | | BSEP 2 | nt-PFIC2 | nt | xxxxxxx | XXXXXXXX<br>XXXXXXXX<br>XXXXXXXX | | XXXXXXXX<br>XXXXXXXX<br>XX | xxxxxxx | BSEP2 | HET | |
| | xxxxx | xxxxxx | DDMMYYYY | DDMMYYYY | xxxx | MRX | PFIC2 | PFIC2 -<br>Primary<br>Cohort | PFIC2 -<br>Primary<br>Cohort | | No-<br>variant-<br>found | NA | | | NA HOM | | | ŀ | НОМ | |

Abbreviations: Rand = Randomization; Trtmt = Treatment; BSEP = bile salt excretion pump; Pheno = Phenotype; cDNA = complementary DNA; Zyg = Zygocity; t = truncated; nt = not truncated; HET = Heterozygous; HOM = Homozygous; NA = not applicable

Note: Sample is used to provide a full characterization and documentation of the mutation type in support of the diagnosis of PFIC. Mutation in Gene data is collected at Screening visit.

**Programming Note:** Use data from CRF.RAND, ADSL, CRF.CPGR.


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

### Listing 16.3.1 Inclusion and Exclusion Criteria All Subjects

Treatment: <Maralixibat or Placebo>

| | | Meet All | | Reason | |
|---|---|---|---|---|---|
| | Protocol | Eligibility | Criteria | Eligibility | |
| Subject | Criteria Version | Criteria? | Not Met | Criteria Not Met | |
| XXXXXX | Original – 14MAR2019 | No | Excl04 | xxxxxxxxxxxxx | |
| XXXXXX | Amendment 1 – 29APR2019 | No | Excl04 | xxxxxxxxxxxx | |
| XXXXXX | Amendment 2 – 22NOV1029 | Yes | | | |
| XXXXXX | Amendment 3 – 16JUN2020 | Yes | | | |
| | xxxxxx<br>xxxxxx | Subject Criteria Version XXXXXXX Original – 14MAR2019 XXXXXXX Amendment 1 – 29APR2019 XXXXXXX Amendment 2 – 22NOV1029 | Protocol Eligibility Criteria Version Criteria? XXXXXXX Original – 14MAR2019 No XXXXXXX Amendment 1 – 29APR2019 No XXXXXXX Amendment 2 – 22NOV1029 Yes | Protocol Eligibility Criteria Subject Criteria Version Criteria? Not Met XXXXXXX Original – 14MAR2019 No Excl04 XXXXXXX Amendment 1 – 29APR2019 No Excl04 XXXXXXX Amendment 2 – 22NOV1029 Yes | Protocol Eligibility Criteria Eligibility Subject Criteria Version Criteria? Not Met Criteria Not Met XXXXXXX Original – 14MAR2019 No Excl04 xxxxxxxxxxxxxx XXXXXXX Amendment 1 – 29APR2019 No Excl04 xxxxxxxxxxxxxx XXXXXXX Amendment 2 – 22NOV1029 Yes |

**Programming Note:** Use CRF.IE.IEPVER for Protocol Criteria Version. See IEVER\_ format in the eCRF document for proper decoding. Use data from CRF.IE.


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

### Listing 16.3.2 Important Protocol Deviations Intent-to-Treat Population

Treatment: <Maralixibat or Placebo>

| | | Event | Event Report | Excl<br>from | | | | | Sponsor | |
|---|---|---|---|---|---|---|---|---|---|---|
| PFIC | | Date | Date | PP | | | Action | | Prior | Date |
| Type | Subject | (Study Day) [1] | (Study Day) [1] | Pop? | Event Type | Description | Taken | Comments | Approval? | Approved |
| xxxxx | XXXXXX | DDMMMYYYY<br>(xx) | DDMMMYYYY<br>(xx) | Υ | Study/Protocol Procedure | xxxxxxxxxxxxx xxxxxx | xxxx xxxxxxxx | xxxxxx | Yes | DDMMMYYYY |
| | | DDMMMYYYY | DDMMMYYYY | | Dosing Error (specify) | XXXXXXXXXXXXXXXXXXXXXXXXX | xxxxxxxxx | xxxxxxx xxxxx | No | |
| | | (xx)<br>DDMMMYYYY<br>(xx) | (xx)<br>DDMMMYYYY<br>(xx) | | Dosing Error (specify) | xxxxxxxxxxxxxxx xxxxx | xxxxxxxx | xxxx | No | |
| | | DDMMMYYYY<br>(xx) | DDMMMYYYY<br>(xx) | | Dosing Error (specify) | xxxxxxxxxx xxxxxxx | xxxxxxxxx | xxxxx xxx xxxx | No | |
| | XXXXXX | DDMMMYYYY<br>(xx) | DDMMMYYYY<br>(xx) | Х | Dosing Error (specify) | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXX | XXX XXXXX | No | |
| xxxxx | XXXXXX | DDMMMYYYY<br>(xx) | DDMMMYYYY<br>(xx) | | Inclusion/Exclusion Criteria | x xxxxxxx xxxxxxxx | xxx xxxxxxx | xxxxx xxxxxxxx | No | |
| | | DDMMMYYYY<br>(xx) | DDMMMYYYY<br>(xx) | | Dosing Error (specify) | xxxxxxxxxxx | xxxxxxxx | XXXXXXX XXXXX | No | |

Abbreviations: Excl from PP Pop? = Subject Excluded from Per-Protocol Population? [1] Study Day is calculated relative to the date of the first dose of study drug.

**Programming Note:** Use data from SDTM.DV and SDTM.SUPPDV. This listing only includes those deviations which are identified as "Important" or "Important – Non Evaluable". Present 'Y' or 'N' in the Excl from PP Pop? column.


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

## Listing 16.4.1 Demographics and Baseline Information Intent-to-Treat Population

Treatment: <Maralixibat or Placebo>

| PFIC | | Age at<br>Consent<br>(Years,<br>Months) | Age at<br>Baseline<br>(Years,<br>Months) | | | Baseline<br>Weight | Baseline<br>Height | Baseline<br>BMI | | | ItchRO<br>in | eDiary |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Туре | Subject | [1] | [1] | Country | Sex | (kg) | (cm) | (kg/m2) | Ethnicity | Race | Paper? | Restrictions |
| xxxxx | XXXXXX | 10, 4 | 10, 5 | GBR | Male | xx.x | xxx | xx.x | Hispanic or<br>Latino | White | No | No |
| | XXXXXX | 1, 11 | 2, 0 | USA | Female | xx.x | xxx | xx.x | Not Hispanic<br>or Latino | Asian | No | No |
| xxxxx | xxxxxx | 5, 5 | 5, 7 | FRA | Female | XX.X | xxx | xx.x | Not Hispanic<br>or Latino | Black or<br>African<br>American | No | No |

Abbreviations: ARG = Argentina; AUT = Austria; BEL = Belgium; BRA = Brazil; CAN = Canada; COL = Columbia; DEU = Germany; FRA = France; GBR = United Kingdom; ITA = Italy; LBN = Lebanon; MEX = Mexico; POL = Poland; SGP = Singapore; TUR = Turkey; USA = United States; BMI = body mass index; ItchRO = Itch Reported Outcomes [1] The subject's age at Screening is used to determine the appropriate age category for the ItchRO, Exploratory Diary Questionnaire, Patient Impression of Severity and PedsQL instruments.

Programming Note: For multiple races, concatenate using ', ' as the delimiter. Use data from CRF.DM and AGE.


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

# Listing 16.4.2 Long-Term Follow-Up Informed Consent and Disease Progression Intent-to-Treat Population

Treatment: <Maralixibat or Placebo>

| | | Date of | | Date of | | | | | | | _ |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | LTFU | Date of | LTFU | | Disease | | | | | Increase |
| | | Parental | LTFU | Adult | | Progression | Reason | | Occurrence | | in |
| PFIC | | Informed | Informed | Informed | | Assessment | Not | Date of | Of Disease | | Concomitant |
| Туре | Subject | Consent | Assent [1] | Consent [2] | Timepoint | Performed? | Assessed | Assessment | Progression? | Outcome | Medications? |
| xxxxx | xxxxxx | DDMMMYYYY | NA | NA | Annual | Yes | | DDMMMYYYY | Yes: xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | PEBD Surgery | Yes |
| | XXXXXX | DDMMMYYYY | NA | NA | Unscheduled | Yes | | DDMMMYYYY | No | | No |
| xxxxx | XXXXXX | DDMMMYYYY | DDMMMYYYY | DDMMMYYYY | xxxxxxxx | No | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | No |

Abbreviations: LTFU = long-term follow-up; NA = not applicable

**Programming Note:** For Occurrence of Disease Progression, if CRF.DP.DPORRES = YES then concatenate DPORRES||': '||DPSPEC. For Outcome, if CRF.DP.DPOUTO = OTHER then concatenate 'OTHER: '||DPOUTOSP. Use data from CRF.DP.


<sup>[1]</sup> Assent is not applicable if the subject is younger than 18 years of age or age of consent at the time of consent.

<sup>[2]</sup> Adult Informed Consent is applicable if subject turned 18 years old or the age of consent during study participation.

Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

### Listing 16.4.3 Informed Consent Intent-to-Treat Population

Treatment: <Maralixibat or Placebo>

| | | Date of | | Subject | | Re-consented | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Parental | Date of | Turn 18 or | | For Major | | | Re-consent |
| PFIC | | Informed | Informed | Age of Consent?/ | | Protocol | Re-consent | Re-consent | Protocol |
| Type | Subject | Consent | Assent [1] | Sign AIC? | Date of AIC [2] | Amendment? | Туре | Date | Version |
| xxxxx | XXXXXX | DDMMMYYYY | NA | No | NA | Yes | Parental/Caregiver<br>Informed Consent | DDMMMYYYY | Amendment 1C –<br>05AUG2019 |
| | XXXXXX | DDMMMYYYY | DDMMMYYYY | No | NA | xx | | | |
| | XXXXXX | DDMMMYYYY | NA | Yes/Yes | DDMMMYYYY | xx | | | |

Abbreviation: AIC = Adult Informed Consent

[1] Assent is not applicable if the subject is younger than 18 years of age or age of consent at the time of consent.

[2] Adult Informed Consent is applicable if subject turned 18 years old or the age of consent during study participation.

**Programming Note:** Use data from CRF.DM, ICR and AIC.


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

### Listing 16.4.4 Medical History Intent-to-Treat Population

Treatment: <Maralixibat or Placebo>

| PFIC<br>Type | Subject | Any<br>History? | System Organ Class | Preferred Term | Verbatim Term | Start Date | End Date |
|---|---|---|---|---|---|---|---|
| xxxxx | XXXXXX | Yes | xxxxxxxxxxxxxxxx | XXXXXXXXXXX | xxxxxxxxxxx | DDMMMYYYY | ONGOING |
| | xxxxxx | No | | | | | |
| | xxxxxx | Yes | xxxxxxxxxxxxxxxx | xxxxxxxxxxxx | xxxxxxxxxx | YYYY | MMMYYYY |
| | | | xxxxxxxxxxxxxx | xxxxxxxxxxx | xxxxxxxxxx | MMMYYYY | ONGOING |
| xxxxx | XXXXXX | Yes | XXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXX | XXXXXXXXXXXX | DDMMMYYYY | DDMMMYYYY |

Note: Events coded using MedDRA version 22.1.

**Programming Note:** Sort medical histories (within subject) by SOC, PT and Verbatim Term. If event is marked as Ongoing, then put "ONGOING" for End Date. Do not include 'UN' or 'UNK' in dates. If entire start or end date is missing then report as 'Unknown'. Use data from CRF.MH.


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

# Listing 16.4.5 Prior and Concomitant Medications/Therapies Intent-to-Treat Population

Treatment: <Maralixibat or Placebo>

| PFIC<br>Type | Subject | Date of<br>Informed<br>Consent | Any<br>Meds? | Ongoing<br>At Time<br>Of IC<br>[1] | Anatomic Therapeutic Class/<br>Preferred Term/<br>Verbatim Term | Start Date/<br>End Date | Indication | Dose (Unit)/<br>Route/<br>Frequency |
|---|---|---|---|---|---|---|---|---|
| xxxxx | xxxxxx | DDMMMYYYY | Yes | Yes | XXXXXXXXX/<br>XXXXXX/<br>XXXXXXXXXXXXXXXXXXX | DDMMMYYYY/<br>ONGOING | XXXXXXXXXXX | XXXX (XXXX)/<br>XXXXXXX/<br>XXXXXXX |
| | XXXXXX | DDMMMYYYY | No | | | | | |
| xxxxx | XXXXXX | DDMMMYYYY | Yes | Yes | xxxxxxxxx/<br>xxxxxx/<br>xxxxxxxxxxxxxxxxxxx | DDMMMYYYY/<br>ONGOING | xxxxxxxxxx | xxxx (xx)/<br>xxxxxxx/<br>xxxxxxx |
| | | | | No | XXXXXXXXX/<br>XXXXXX/<br>XXXXXXXXXXXXXXXXXXX | DDMMMYYYY/<br>DDMMMYYYY | XXXXXXXXXXXX | XXXX (XXXX)/<br>XXXXXXX/<br>XXXXXXX |

Abbreviation: IC = Informed Consent

Note: Medication coded using WHO-DD (Enhanced version September 2019), Anatomic Therapeutic Class (ATC) Level 2. Preferred term is ATC Level 5.

[1] Indicates whether the medication was ongoing at the time of Informed Consent. Medications that are stopped prior to the time of informed consent are not recorded. Only therapies administered for liver disease should be captured prior to baseline.

**Programming Note:** Sort medications (within subject) by start date and then by end date. For any field where answer is "Other", concatenate the specify (e.g., OTHER: mmol) . Use data from CRF.CM.


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4) PCN Number: MIRU8967

### Listing 16.5.1 Liver Imaging Intent-to-Treat Population

Treatment: <Maralixibat or Placebo>

| | | Method of | | | | Masses | |
|---|---|---|---|---|---|---|---|
| PFIC | | Liver | Date of | Masses | | in the | |
| Туре | Subject | Imaging | Imaging | Observed? | If Masses Observed, Specify | Liver? | If Masses in the Liver, Specify |
| xxxxx | XXXXXX | Ultrasound | DDMMMYYYY | Yes | XXXXXX | | |
| | | Ultrasound | DDMMMYYYY | No | | | |
| | XXXXXX | Ultrasound | DDMMMYYYY | | | Yes | XXXXXXXX |
| | | Ultrasound | DDMMMYYYY | | | Yes | XXXXXXXX |
| | XXXXXX | MRI | DDMMMYYYY | No | | | |
| xxxxx | XXXXXX | Ultrasound | DDMMMYYYY | | | No | |

**Programming Note:** Use data from CRF.IM where formnam = IM and IM2.


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4) PCN Number: MIRU8967

### Listing 16.5.2 **Liver-Associated Events** Intent-to-Treat Population

| | | Liver- | | |
|-------|---------|------------|------------------------|-------------------|
| | | Associated | | Event |
| PFIC | | Event | | Start Date |
| Туре | Subject | Reported? | Event | (Study Day) [1] |
| xxxxx | XXXXXX | No | | |
| | XXXXXX | Yes | OTHER: xxxxxxxxxxxxxxx | DDMMMYYYY<br>(xx) |
| xxxxx | XXXXXX | Yes | PEBD SURGERY | DDMMMYYYY<br>(xx) |

<sup>[1]</sup> Study Day is calculated relative to the date of the first dose of study drug.

**Programming Note:** Use data from CRF.LAE.


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4) PCN Number: MIRU8967

### Listing 16.5.3 Liver Transplant List Intent-to-Treat Population

Treatment: <Maralixibat or Placebo>

| | | Placed on<br>Liver | Date Placed<br>On Liver | Still on<br>Liver | | Date Removed<br>From Liver |
|---|---|---|---|---|---|---|
| PFIC | | Transplant | Transplant | Transplant | | Transplant |
| Type | Subject | List? | List | List? | Reason for Removal | List |
| xxxxx | XXXXXX | No | | | | |
| | XXXXXX | Yes | DDMMMYYYY | Yes | | |
| xxxxx | XXXXXX | Yes | DDMMMYYYY | No | xxxxxxxxxxxxxxxxx | DDMMMYYYY |

**Programming Note:** Use data from CRF.LT.


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

## Listing 16.6.1 Study Drug Supplied and Compliance Safety Population

Treatment: <Maralixibat or Placebo>

| | | Study | Study Drug | Study Drug | Reason | Bottle | Date of Do | osing Error | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| PFIC | | <b>Drug Quantity</b> | Supplied via | Taken as | Not Fully | ID | Start | End | Type of | | Compliance |
| Туре | Subject | Sufficient? | Shipment? | Prescribed? | Supplied | Numbers | (Study Day) [1] | (Study Day) [1] | Dosing Error | Comments | % [2] |
| xxxx | XXXXXX | Yes | No | No | | xxxxx,<br>xxxxx | DDMMMYYYY<br>(xx) | DDMMMYYYY<br>(xx) | xxxxxx | XXXXXX | xx.x% |
| | | Yes | No | No | | xxxxx | DDMMMYYYY<br>(xx) | DDMMMYYYY<br>(xx) | XXXXXXXX | XXXXXXXX | |
| | | Yes | No | Yes | | xxxxx | | | | | |
| | | Yes | No | Yes | | xxxxx | | | | | |
| | | Yes | No | Yes | | xxxxx | | | | | |
| | | Yes | No | Yes | | xxxxx | | | | | |
| | | No | Yes | Yes | xxxxxxxx | | | | | | |
| | | Yes | No | Yes | | xxxxxx | | | | | |

Abbreviation: ID = identification

Note: Listing includes all dosing deviations, including those due to an adverse event.

**Programming Note:** Use data from CRF.DA, formnam = DA3 and SDC. % Compliance is in ADEX.


<sup>[1]</sup> Study Day is calculated relative to the date of the first dose of study drug.

<sup>[2]</sup> Compliance (%) = 100\* (Treatment duration in days – Number of days both morning and evening doses were missed) / Treatment duration in days), where Treatment duration (days) = Date of last dose of study drug – Date of first dose of study drug + 1 day. For subject that are missing the date of last dose of study drug, the last known contact date is used to calculate treatment duration.

Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

### Listing 16.6.2 Study Drug Exposure Safety Population

Treatment: <Maralixibat or Placebo>

| | | Body<br>Weight at | Admini-<br>stered | | | | Treatment | |
|---|---|---|---|---|---|---|---|---|
| PFIC | | Screening | Study | Dosage | Start Date | Stop Date | Duration | Total Dose |
| Туре | Subject | (kg) | Drug? | (μg/kg) | (Study Day) [1] | (Study Day) [1] | (days) | (μg/kg) [2] |
| xxxxx | XXXXXX | xx.x | Yes | 150 | DDMMMYYYY (xx) | DDMMMYYYY (xx) | х | xxx |
| | | | Yes | 300 | DDMMMYYYY (xx) | DDMMMYYYY (xx) | x | xxx |
| | | | Yes | 450 | DDMMMYYYY (xx) | DDMMMYYYY (xx) | x | xxxx |
| | | | Yes | 600 | DDMMMYYYY (xx) | DDMMMYYYY (xx) | x | XXXXX |
| XXXXX | XXXXXX | xx.x | xxx | xxx | DDMMMYYYY (xx) | DDMMMYYYY (xx) | х | xxx |
| | | | xxx | xxx | DDMMMYYYY (xx) | DDMMMYYYY (xx) | x | xxx |
| | | | xxx | xxx | DDMMMYYYY (xx) | DDMMMYYYY (xx) | x | xxxxx |
| | | | xxx | xxx | DDMMMYYYY (xx) | DDMMMYYYY (xx) | xx | xxxxxx |
| | | | xxx | XXX | DDMMMYYYY (xx) | DDMMMYYYY (xx) | XX | xxxxxx |

<sup>[1]</sup> Study Day is calculated relative to the date of the first dose of study drug.

**Programming Note:** Use data fromSDTM.EX.


<sup>[2]</sup> Total Dose ( $\mu$ g /kg) = Dose ( $\mu$ g/kg) x Number of doses taken between start and stop dates. For subjects who are missing the date of last dose of study drug, the last known contact date is used in the calculation of treatment duration and study drug exposure.

Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4) PCN Number: MIRU8967

### Listing 16.6.3 Study Drug Accountability Safety Population

Treatment: <Maralixibat or Placebo>

| PFIC<br>Type | Subject | Study Drug Dispensed?/ If No, Reason | Kit Number | Clinic<br>Visit | Dispense<br>Date<br>(Study Day) [2] | Volume<br>Dispensed<br>(mL) | Return<br>Date<br>(Study Day) [1] | Volume<br>Returned<br>(mL) | Comments |
|---|---|---|---|---|---|---|---|---|---|
| | - | | | | | | | | |
| XXXXX | XXXXXX | Yes | XXXXX | VISIT 1 | DDMMMYYYY (x) | XX | DDMMMYYYY (x) | XX.X | |
| | | Yes | XXXXX | VISIT 2 | DDMMMYYYY (xx) | XX | DDMMMYYYY (xx) | XX.X | |
| | | Yes<br>No/xxxxx | xxxxx | VISIT 3 | DDMMMYYYY (xx) | xx | DDMMMYYYY (xx) | xx.x | |

[1] Study Day is calculated relative to the date of the first dose of study drug.

**Programming Note:** Use data from CRF.DA, formnam = DA2.


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

## Listing 16.7.1 Total Serum Bile Acid Intent-to-Treat Population

Treatment: <Maralixibat or Placebo>

| PFIC | | Age [1]/ | Clinic | Analysis | Collection Date | Total<br>sBA | Flag | Chango fron | n Baseline [4] |
|---|---|---|---|---|---|---|---|---|---|
| Туре | Subject | Sex | Visit | Visit | (Study Day) [2] | (umol/L) | [3] | Observed | Percent |
| xxxx | XXXXXX | xx/M | Screening | Screening | DDMMMYYYY (-x) | xxx.x | | | |
| | | | Week 0 | Baseline | DDMMMYYYY (xx) | xxx.x | | xx.x | xx.x |
| | | | Week x | Week 2 | DDMMMYYYY (xx) | xxx.x | В | xx.x | XX.X |
| | | | Week x | Week 6 | DDMMMYYYY (xx) | xxx.x | х | xx.x | xx.x |
| | | | Week x | Week 10 | DDMMMYYYY (xx) | xxx.x | х | xx.x | xx.x |
| | | | Week x | Week 14 | DDMMMYYYY (xxx) | xxx.x | х | xx.x | XX.X |
| | | | Week x | Week 18 | DDMMMYYYY (xxx) | xxx.x | х | xx.x | xx.x |
| | | | Week x | Week 22 | DDMMMYYYY (xxx) | xxx.x | х | xx.x | XX.X |
| | | | Week x | Week 26 | | | | | |

Note: Baseline and all post-baseline sBA samples are assayed at Frontage Laboratories, while screening sBA samples are assayed at ACM Global Laboratories. Only pre-dose samples assayed at Frontage Laboratories are used as a baseline sample.

- [1] Age (years) at Baseline.
- [2] Study Day is calculated relative to the date of the first dose of study drug.
- [3] 'b' indicates ≥ 75% reduction from baseline OR sBA < 102 umol/L
- [4] Baseline is Day 0 value (prior to first dose of study drug).

**Programming Note:** Add footnote for sBA column if needed to explain abbreviation (eg, 'ND = Not Done'); report sBA, observed CFB, and %CFB values to 1 decimal place. Use data from ADaM.ADLB.


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

#### Listing 16.7.2 Serum Bile Acid Subspecies Intent-to-Treat Population

Treatment: <Maralixibat or Placebo>

| | | Age [1]/ | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PFIC | | Sex/ | Clinic | Study | | | | | | | | | | | | | | | |
| Type | Subject | Country | Visit | Day [2] | CDCA | CHA | DCA | GCA | GCDCA | GDCA | GLCA | GUDCA | LCA | TCA | TCDCA | TDCA | TLCA | TUDCA | UDCA |
| | • | | | • | • | | | | • | | | • | • | | • | • | | | • |
| XXXXX | XXXXXX | 3/M/GBR | Screening | -x | x.xx | x.xx | x.xx | xxx.xx | xx.xx | x.xx | x.xx | xxx.xx | x.xx | xx.xx | xx.xx | x.xx | x.xx | xx.xx | x.xx |
| | | | Day 0 | -x | x.xx | X.XX | x.xx | xxx.xx | xx.xx | x.xx | x.xx | xxx.xx | x.xx | xx.xx | xx.xx | x.xx | x.xx | xx.xx | x.xx |
| | | | Week 2 | XX | x.xx | x.xx | x.xx | xxx.xx | XX.XX | x.xx | x.xx | XXX.XX | x.xx | xx.xx | xx.xx | x.xx | x.xx | xx.xx | x.xx |

#### (Continue for all clinic visits)

.

Abbreviations: ARG = Argentina; AUT = Austria; BEL = Belgium; BRA = Brazil; CAN = Canada; COL = Columbia; DEU = Germany; FRA = France; GBR = United Kingdom; ITA = Italy; LBN = Lebanon; MEX = Mexico; POL = Poland; SGP = Singapore; TUR = Turkey; USA = United States; CDCA = Chenodeoxycholic Acid; CHA = Cholic Acid; DCA = Deoxycholic Acid; GCA = Glycocholic Acid; GCDCA = Glycochenodeoxycholic Acid; GCDCA = Glycochenodeoxycholic Acid; GCA = Lithocholic Acid; TCA = Taurocholic Acid; TCDCA = Taurochenodeoxycholic Acid; TDCA = Taurodeoxycholic Acid; TLCA = Taurolithocholic Acid; TUDCA = Tauroursodeoxycholic Acid; UDCA = Ursodeoxycholic; BQL = below quantification limit

Note: Serum bile acid components are presented in units of umol/L. The lower quantification limit is 0.01 μmol/L for CA, GDCA, TDCA, TLCA, CDCA, GLCA, DCA, and LCA. For GCA, TCA, TUDCA, GUDCA, GCDCA, TCDCA, and UDCA, the lower limit is 0.2 μmol/L.

- [1] Age (years) at Baseline.
- [2] Study Day is calculated relative to the date of the first dose of study drug.

Programming Note: Use data from SDTM.LB. If Clinic Visit = 'Week 0' assign 'Day 0'. Use raw values; for example, <0.10, not analysis value.


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

Listing 16.7.3 Clinician Scratch Scale Score Intent-to-Treat Population

Treatment: <Maralixibat or Placebo>

| | | | | Date of | Clinician Scrato | ch Scale Score |
|---|---|---|---|---|---|---|
| PFIC | | | Assessment | Assessment | | Change from |
| Type Subject | Subject | Clinic Visit | Completed? | (Study Day) [1] | Observed [2] | Baseline [3] |
| xxxxx | XXXXXX | Screening | Yes | DDMMMYYYY (-xx) | X | |
| | | Day 0 | Yes | DDMMMYYYY (xx) | Χ | |
| | | Week 2 | No | | | |
| | | Week 4 | Yes | DDMMMYYYY (xx) | Χ | Χ |
| | | Week 6 | Yes | DDMMMYYYY (xx) | Χ | Χ |
| | | Week 10 | Yes | DDMMMYYYY (xx) | Χ | Χ |
| | | Week 14 | Yes | DDMMMYYYY (xx) | Χ | Χ |
| | | Week 18 | Yes | DDMMMYYYY (xx) | Χ | Χ |
| | | Week 22 | Yes | DDMMMYYYY (xx) | Χ | Χ |
| | | Week 26 | Yes | DDMMMYYYY (xx) | Χ | X |

<sup>[1]</sup> Study Day is calculated relative to the date of the first dose of study drug.

**Programming Note:** Use data from SDTM.QS.


<sup>[2] 0 =</sup> None; 1 = Rubbing or mild scratching when undistracted; 2 = Active scratching without evident skin abrasions; 3 = Abrasion evident; 4 = Cutaneous mutilation, haemorrhage and scarring evident.

<sup>[3]</sup> Baseline is Day 0 value (prior to first dose of study drug). If Day 0 value is not available, the last value obtained during Screening is used as the baseline value.
Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

Listing 16.7.4
Itch Reported Outcomes (Subject and Caregiver) Average Morning and Evening Scores
Intent-to-Treat Population

Treatment: <Maralixibat or Placebo>

| | | | Analysis | <u>Itch</u> | nRO (Pt) | [3] Morni | ng | <u>Itch</u> | RO (Pt) | [3] Eveni | ng | <u>ItchF</u> | O (Obs | ) Mornir | <u>ıg</u> | | ItchRO (0 | Obs) Evenin | g |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PFIC | | Age | Visit | Frequ | ency | Seve | rity | Frequ | ency | Seve | rity | Freque | ency | Seve | rity | Frequ | ency | Seve | erity |
| Туре | Subject | [1] | Period [2] | Score | CFB | Score | CFB | Score | CFB | Score | CFB | Score | CFB | Score | CFB | Score | CFB | Score | CFB |
| xxxx | XXXXXX | Х | Baseline | x.xx | | x.xx | | x.xx | | x.xx | | x.xx | | x.xx | | x.xx | | x.xx | |
| | | | Wks 1-6 | X.XX | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | X.XX | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | X.XX | X.X |
| | | | Wks 7-10 | X.XX | x.xx | X.XX | X.XX | X.XX | x.xx | x.xx | X.XX | X.XX | x.xx | x.xx | X.XX | x.xx | x.xx | X.XX | X.X |
| | | | Wks 11-14 | X.XX | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | X.XX | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | X.XX | x.x |
| | | | Wks 15-18 | X.XX | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | X.XX | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | X.XX | X.X |
| | | | Wks 19-22 | X.XX | X.XX | X.XX | X.XX | X.XX | x.xx | x.xx | X.XX | X.XX | x.xx | x.xx | X.XX | x.xx | x.xx | X.XX | x.x |
| | | | Wks 23-26 | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | X.XX | X.XX | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | X.X |
| (XXXX | XXXXXX | Х | Baseline | | | | | | | | | x.xx | | x.xx | | x.xx | | x.xx | |
| | | | Wks 1-6 | | | | | | | | | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.x |

(Continue for all analysis visit periods)

Abbreviation: ItchRO = Itch Reported Outcome; CFB = Change from Baseline, defined as post-baseline value minus baseline value; Pt = Patient; Obs = Observer Note: ItchRO scores have a range from 0 to 4, with the higher score indicating increasing itch frequency/severity.

**Programming Note:** Use data from ADAM.ADQS


<sup>[1]</sup> Age (years) at Screening.

<sup>[2]</sup> Average scores are calculated for each time period, averaging 7-day weekly averages. For each time period, the average of the 4 weekly scores is presented; or 6 weekly scores for Weeks 1-6. The baseline score is calculated as the average of the 4 weekly average scores before the first dose of study drug.

<sup>[3] &#</sup>x27;--' indicates assessment is not applicable for subject age (i.e., if a subject was < 9 years old).

Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

Listing 16.7.5
Exploratory Diary Questionnaire (Subject and Caregiver) Average Morning and Evening Scores
Intent-to-Treat Population

Treatment: <Maralixibat or Placebo>

| | | | Analysis | EDQ (Pt) [4] | Morning | | EDQ (Pt) | [4] Eveni | n <u>g</u> | EDQ (Obs) | Morning | EDQ (Obs) | Evening |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PFIC | | Age | Visit | Seve | rity | Free | quency | Se | verity | Sev | erity | Seve | erity |
| Туре | Subject | [2] | Period [3] | Score | CFB | Score | CFB | Score | CFB | Score | CFB | Score | CFB |
| xxxx | XXXXXX | Х | Baseline | x.xx | | x.xx | | x.xx | | x.xx | | x.xx | |
| | | | Wks 1-6 | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx |
| | | | Wks 7-10 | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx |
| | | | Wks 11-14 | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx |
| | | | Wks 15-18 | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx |
| | | | Wks 19-22 | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx |
| | | | Wks 23-26 | x.xx | x.xx | x.xx | x.xx | X.XX | x.xx | x.xx | X.XX | x.xx | x.xx |
| xxxx | XXXXXX | Х | Baseline | | | | | | | x.xx | | x.xx | |
| | | | Wks 1-6 | | | | | | | x.xx | x.xx | x.xx | x.xx |

Abbreviation: EDQ = Exploratory Diary Questionnaire; CFB = Change from Baseline, defined as post-baseline value minus baseline value; Pt = Patient; Obs = Observer Note: EDQ scores have a range from 1 to 5, with the higher score indicating increasing itch frequency/severity.

**Programming Note:** Use data from ADAM.ADQS


<sup>[1]</sup> Age (years) at Screening.

<sup>[2]</sup> Average scores are calculated for each time period, averaging 7-day weekly averages. For each time period, the average of the 4 weekly scores is presented; or 6 weekly scores for Weeks 1-6. The baseline score is calculated as the average of the 4 weekly average scores before the first dose of study drug.

<sup>[3] &#</sup>x27;--' indicates assessment is not applicable for subject age (i.e., if a subject was < 9 years old).

Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

### Listing 16.7.6.1 PIC and CIC Intent-to-Treat Population

Treatment: <Maralixibat or Placebo>

| | | | Patient | Impression of Change | (PIC) | Cai | regiver Impression of ( | Change (CIC) | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | Date of | | | Date of | | |
| PFIC | | Clinic | | Assessment | | | Assessment | Itch | Xanthoma |
| Type | Subject | Visit | Completed? | (Study Day) [1] | Score [2] | Completed? | (Study Day) [1] | Score [2] | Score [2] |
| XXXXX | XXXXXX | Week 26 EOT | Yes | DDMMMYYYY (xx) | X | Yes | DDMMMYYYY (xx) | Χ | X |
| XXXXX | XXXXXX | Week 26 EOT | Yes | DDMMMYYYY (xx) | Χ | Yes | DDMMMYYYY (xx) | Χ | Χ |

### (Continue for all clinic visits)

Note: PIC is completed by subjects who are 9 years of age or older.

**Programming note:** Merge records within a subject together by study visit; remove Visit column if there are visit discrepancies between assessments. Use data from SDTM.QS.


<sup>[1]</sup> Study Day is calculated relative to the date of the first dose of study drug.

<sup>[2] 1 =</sup> Much better; 2 = Better; 3 = A little better; 4 = No change; 5 = A little worse; 6 = Worse; 7 = Much worse

Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

# Listing 16.7.6.2 PIS and CIS Intent-to-Treat Population

Treatment: <Maralixibat or Placebo>

| | | | Patient Impre | ession of Severity of Pr | uritus (PIS) | Caregiver Imp | ression of Severity of I | Pruritus (CIS |
|---|---|---|---|---|---|---|---|---|
| | | • | | Date of | | | Caregiver Impression of Severity of Prince Date of Assessment Completed? (Study Day) [1] Yes DDMMMYYYY (xx) Yes DDMMMYYYY (xx) No Yes DDMMMYYYY (xx) | |
| PFIC | | Clinic | | Assessment | | | Assessment | |
| Туре | Subject | Visit | Completed? | (Study Day) [1] | Score [2] | Completed? | (Study Day) [1] | Score [3] |
| xxxx | XXXXXX | Day 0 | Yes | DDMMMYYYY (xx) | X | Yes | DDMMMYYYY (xx) | х |
| | | Week 4 | Yes | DDMMMYYYY (xx) | X | Yes | DDMMMYYYY (xx) | Χ |
| | | Week 6 | No | | | No | | |
| | | Week 10 | Yes | DDMMMYYYY (xx) | X | Yes | DDMMMYYYY (xx) | Χ |
| | | Week 14 | Yes | DDMMMYYYY (xx) | X | Yes | DDMMMYYYY (xx) | Χ |
| | | Week 18 | Yes | DDMMMYYYY (xx) | X | Yes | DDMMMYYYY (xx) | Χ |
| | | Week 22 | Yes | DDMMMYYYY (xx) | X | Yes | DDMMMYYYY (xx) | Χ |
| | | Week 26 EOT | Yes | DDMMMYYYY (xx) | Х | Yes | DDMMMYYYY (xx) | Χ |

<sup>[1]</sup> Study Day is calculated relative to the date of the first dose of study drug.

**Programming note:** Merge records within a subject together by study visit; remove Visit column if there are visit discrepancies between assessments. Use data from SDTM.QS.


<sup>[2] 0 =</sup> I didn't feel itchy at all; 1 = I felt a little bit itchy; 2 = I felt pretty itchy; 3 = I felt very itchy; 4 = I felt very, very itchy

<sup>[3] 0 =</sup> None; 1 = Mild; 2 = Moderate; 3 = Severe; 4 = Very severe

Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

## Listing 16.7.7 Efficacy Laboratory Tests Intent-to-Treat Population

Treatment: <Maralixibat or Placebo>

| | | | | | | | | | Local | | | Standa | ard | Change |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PFIC | | Age [1]/ | Laboratory Test | Laboratory | Clinic | Analysis | Collection Date | Fasting? | Lab?/ | Test | Re | ference | Range | from |
| Туре | Subject | Sex | Category | Test (units) | Visit | Visit | (Study Day) [2] | [3] | Visit [4] | Result [5] | Low | High | Flag [6] | Baseline [7] |
| xxxxx | XXXXXX | xx/M | Cholestasis | Serum Bile Acid (μmol/L) | Week 0 | Baseline | DDMMMYYYY<br>(-x) | X | No | xxx | | | | |
| | | | Biomarkers | | | | | | | | | | | |
| | | | | 7α hydroxyl-4-cholesten-3-one<br>(C4) (ng/mL) | Week 0 | Baseline | DDMMMYYYY<br>(-x) | Х | No | XXX | | | | |
| | | | Liver Enzymes | Alanine aminotransferase (U/L) | xxxxxx | Baseline | DDMMMYYYY<br>(-x) | Х | Yes/Baseline | e xxx | xx | xx | | |
| | | | | Bilirubin (mg/dL) | xxxxxx | Baseline | DDMMMYYYY<br>(-x) | Х | | xxx | xx | xx | | |

#### (Continue for lab categories and lab tests specified in Programming Note)

- [1] Age (years) at Baseline.
- [2] Study Day is calculated relative to the date of the first dose of study drug.
- [3] Y = Yes; N = No; U = Unknown
- [4] Were the labs collected for a protocol-related visit in place of central lab collection?/If yes, for which visit?
- [5] 'x' indicates a concentration reported as below the minimum quantitation limit. Half of the minimum quantitation limit is used as the analysis value.
- [6] H = (High) The result is above the upper limit of the reference range for normal subjects; L = (Low) The result is below the lower limit of the reference range for normal subjects.
- [7] Baseline is Day 0 value (prior to first dose of study drug). If Day 0 value is not available, the last value obtained during Screening is used as the baseline value.

**Programming Note:** See Appendix 1 of SAP for list of efficacy lab tests (15 lab tests in total); do <u>not</u> include the 15 sBA subspecies since they are in Listing 16.7.2. Round PELD and MELD to integers; round sBA (BILEAC), FIB-4 and APRI to 2 decimal places. Use data from ADaM.ADLB.


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

# Listing 16.7.8 Height, Weight, and BMI z-Score Intent-to-Treat Population

Treatment: <Maralixibat or Placebo>

| PFIC<br>Type | Subject | Age [1]/<br>Sex | Clinic<br>Visit | Analysis<br>Visit | Vital<br>Signs<br>Collected? | Date of<br>Measurement<br>(Study Day) [2] | Height<br>(cm) | Weight<br>(kg) | BMI<br>(kg/m²) | Height<br>z-Score | Weight<br>z-Score | BMI<br>z-Score |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxxx | XXXXXX | 1/M | Screening | Screening | Yes | DDMMMYYYY (xx) | XXX | xx.x | xx.x | x.xx | x.xx | x.xx |
| | | | Week 0 | Baseline | Yes | DDMMMYYYY (xx) | xxx | xx.x | xx.x | x.xx | x.xx | x.xx |
| | | | xxxxx | Week 2 | Yes | DDMMMYYYY (xx) | XXX | xx.x | xx.x | x.xx | x.xx | x.xx |
| | | | xxxxx | Week 4 | Yes | DDMMMYYYY (xx) | xxx | xx.x | xx.x | x.xx | x.xx | x.xx |
| | | | xxxxxx | Week 6 | Yes | DDMMMYYYY (xx) | xxx | xx.x | xx.x | x.xx | x.xx | x.xx |
| xxxxx | xxxxxx | x/X | xxxxxxx | Baseline | Yes | DDMMMYYYY (xx) | xxx | XX.X | xx.x | x.xx | x.xx | x.xx |
| | | | xxxxxxx | Week xx | Yes | DDMMMYYYY (xx) | xxx | xx.x | xx.x | x.xx | x.xx | x.xx |
| | | | XXXXXX | Week xx | Yes | DDMMMYYYY (xx) | xxx | xx.x | xx.x | x.xx | x.xx | x.xx |
| | | | xxxxxxx | Week xx | Yes | DDMMMYYYY (xx) | xxx | xx.x | xx.x | x.xx | x.xx | x.xx |

(Continue for all analysis visits)

Abbreviation: BMI = Body Mass Index

Note: Listing includes all records used for analysis purposes. A subject's sex and age (at each analysis visit) are used to derive z-scores.

**Programming Note:** Use data from ADAM.ADVS.


<sup>[1]</sup> Age (years) at Baseline.

<sup>[2]</sup> Study Day is calculated relative to the date of the first dose of study drug.

Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

Listing 16.7.9
Exploratory Diary Questionnaire (Caregiver) Average Morning Scores in Sleep Disturbance
Intent-to-Treat Population

Treatment: <Maralixibat or Placebo>

| | | Age at | | Sleep Disturk | oance Score |
|-------|---------|-----------|----------------|---------------|-------------|
| PFIC | | Screening | Analysis Visit | | Change from |
| Туре | Subject | (years) | Period [1] | Observed [3] | Baseline |
| | | | - " | | |
| XXXXX | XXXXXX | XX | Baseline | x.xx | |
| | | | Wks 1-6 | x.xx | x.xx |
| | | | Wks 7-10 | x.xx | x.xx |
| | | | Wks 11-14 | x.xx | x.xx |
| | | | Wks 15-18 | X.XX | X.XX |
| | | | Wks 19-22 | X.XX | X.XX |
| | | | Wks 23-26 | x.xx | x.xx |

Note: Caregivers for all subjects aged <9 years complete the EDQ(Obs) instrument. Sleep disturbance is scored in the morning, in which the caregiver scores the following question: "Because of itch, my child had trouble staying asleep.".

[1] Average scores are calculated for each time period, averaging 7-day weekly averages. For each time period, the average of the 4 weekly scores is presented; or 6 weekly scores for Weeks 1-6. The baseline score is calculated as the average of the 4 weekly average scores before the first dose of study drug.

[2] Study Day is calculated relative to the date of the first dose of study drug.

[3] 1 = Never; 2 = Rarely; 3 = Sometime; 4 = Often; 5 = Almost Always

**Programming Note:** Use ADAM.ADQS


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

Listing 16.8.1 Adverse Events Safety Population

Treatment: <Maralixibat or Placebo>

| PFIC<br>Type | Subject | Any<br>AEs? | PFIC<br>Rec<br>[1] | System Organ Class/<br>Preferred Term/<br>Verbatim Term | TEAE? | Start Date<br>(Study Day)<br>[2] | End Date<br>(Study Day)<br>[2] | Event<br>Duration<br>(days) | Severity Grade/<br>Relationship to<br>Study Drug | Med PFIC Rec?/<br>Outcome/<br>Study Drug<br>Action Taken | Serious?/<br>Criteria<br>Met [3] | Hospitalization<br>Start Date-<br>End Date/<br>Comment |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxxx | XXXXXX | Yes | xxx | xxxxxxxxx xxxxx xxxxx/<br>xxxxxxxxxxxxxxxx | Yes | DDMMMYYYY<br>(xx) | DDMMMYYYY<br>(xx) | xx | Grade 1 (Mild)/<br>Not Related | Yes/<br>Recovered/Resolved/<br>Dose Not Changed | No/<br>None | N/A/<br>None |
| xxxxx | xxxxxx | Yes | xxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | No | DDMMMYYYY<br>(xx) | DDMMMYYYY<br>(xx) | XX | Grade x (xxxx)/<br>Related | xxx/<br>xxxxxxxx/<br>xxxx xxx xxxxxxx | Yes/<br>HOSP; LT | DDMMMYYYY-<br>DDMMMYYYY/<br>xxxxxxxxx xxxxx<br>xxxxxxxx; xxxxx |

Abbreviations: TEAE = Treatment-Emergent Adverse Event; Med PFIC Rec? = Medical Treatment Received?

Note: Adverse events coded using MedDRA version 22.1. In determining TEAEs and study day, partial dates were imputed based on the SAP. Treatment-emergent adverse events are AEs with a start date on or after the first dose of study drug and started prior to the last dose of study drug plus 7 days. For any subjects who die during the study and the date of death is between the date of first dose of study drug and the date of study discontinuation, all AEs that occur during the study are considered as TEAEs irrespective of the last dose.

- [1] Treatment received at the onset of the event; MRX dose reported in units of  $\mu g/kg/day$ . For AEs that started within 7 days after the last dose of study drug, the last MRX dose received is listed. For AEs that started > 7 days after the last dose of study drug, treatment received is blank. NT = Not Treated (for AEs that started prior to 1st dose of study drug)
- [2] Study Day is calculated relative to the date of the first dose of study drug.
- [3] CONG = Resulted in congenital anomaly or birth defect; DISAB = Resulted in significant incapacity or substantial disruption of normal life functions; FATAL = Resulted in death; HOSP = Required or prolonged hospitalization; LT = Was life-threatening; OTHER = Other medically important event that may jeopardize the subject.

**Programming Note:** Sort AEs (within treatment received, cohort and subject) by start date and then by end date; events that are ongoing would be listed after those with end dates (for those events with the same start date). For Comment, concatenate CRF.AE.AENARF1-4 with a '; ' delimiter. Use data from ADAM.ADAE.


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

Listing 16.8.2.1
Adverse Events of Clinical Interest: Diarrhoea Events
Safety Population

Same shell as Listing 16.8.1, except remove 'Any AEs?' column

Listing 16.8.2.2

Adverse Events of Clinical Interest: Lipid Soluble Vitamin Deficiency Events
Safety Population

Same shell as Listing 16.8.1, except remove 'Any AEs?' column

Listing 16.8.2.3

Adverse Events of Clinical Interest: Elevated Transaminases Events

Safety Population

Same shell as Listing 16.8.1, except remove 'Any AEs?' column

Listing 16.8.2.4

Adverse Events of Clinical Interest: Elevated Bilirubin Events

Safety Population

Same shell as Listing 16.8.1, except remove 'Any AEs?' column

Listing 16.8.3
Treatment Related Adverse Events
Safety Population

Same shell as Listing 16.8.1, except remove 'Any AEs?' column


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

Listing 16.8.4.1 Serious Adverse Events Safety Population

Same shell as Listing 16.8.1, except remove 'Any AEs?' column

Listing 16.8.4.2
Serious Related Adverse Events
Safety Population

Same shell as Listing 16.8.1, except remove 'Any AEs?' column

Listing 16.8.5
Adverse Events Leading to Study Drug Discontinuation
Safety Population

Same shell as Listing 16.8.1, except remove 'Any AEs?' column

Listing 16.8.6 Severe Adverse Events Safety Population

Same shell as Listing 16.8.1, except remove 'Any AEs?' column

Listing 16.8.7 Adverse Events Resulting in Death Safety Population

Same shell as Listing 16.8.1, except remove 'Any AEs?' column


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

Listing 16.9.1 Vital Signs Safety Population

Treatment: <Maralixibat or Placebo>

| PFIC<br>Type | Subject | Age [1] | Clinic<br>Visit | Vital<br>Signs<br>Collected? | Date of<br>Measurement<br>(Study Day) [2] | Heart<br>Rate<br>(beats/min) | Respiratory<br>Rate<br>(rpm) | Systolic<br>Blood<br>Pressure<br>(mmHg) | Diastolic<br>Blood<br>Pressure<br>(mmHg) | Temperature<br>(degrees C) |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxx | XXXXXX | xx | Screening | Yes | DDMMMYYYY (-xx) | XX | XX | XXX | XX | XX.X |
| | | | Day 0 | Yes | DDMMMYYYY (xx) | XX | XX | XXX | XX | XX.X |
| | | | Week 2 | Yes | DDMMMYYYY (xx) | XX | XX | XXX | XX | XX.X |
| | | | Week 4 | No | | | | | | |
| | | | Week 6 | Yes | DDMMMYYYY (xx) | XX | XX | XXX | XX | XX.X |

### (Continue for all clinic visits)

Abbreviations: H = High: The result is above the upper limit of the reference range for normal subjects; L = Low: The result is below the lower limit of the reference range for normal subjects

Note: Normal reference ranges for heart rate, respiratory rate and blood pressure are based on the subject's age at time of the measurement.

- [1] Age (years) at Baseline.
- [2] Study Day is calculated relative to the date of the first dose of study drug.

**Programming Note:** Use data from SDTM.VS. If Clinic Visit = 'WEEK 0' assign 'Day 0'.


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

### Listing 16.9.2 **Physical Examination** Safety Population

Treatment: <Maralixibat or Placebo>

| | | | | Examination | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| PFIC | | Clinic | Examination | Date | Any/Changed | | | | Clinically |
| Туре | Subject | Visit | Performed? | (Study Day) [1] | Abnormalities? [2] | Body System | Result | Abnormal Finding | Significant? |
| xxxxx | XXXXXX | Screening | Yes | DDMMMYYYY (-xx) | Yes | System 1 | Abnormal | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Yes |
| | | | | | | System 2 | Normal | | |
| | | | | | | System 3 | Normal | | |
| | | Day 0 | Yes | DDMMMYYYY (xx) | No | | | | |
| | | Week 2 | Yes | DDMMMYYYY (xx) | No | | | | |
| | | Week 4 | Yes | DDMMMYYYY (xx) | Yes | System 6 | | XXXXXXXXXXXX | |
| | | Week 6 | Yes | DDMMMYYYY (xx) | Yes | System 6 | | XXXXXXXXXXXXXXXXXX | |
| | | Week 10 | Yes | DDMMMYYYY (xx) | No | | | | |
| xxxxx | XXXXXX | Screening | Yes | DDMMMYYYY (-xx) | No | | | | |
| | | Day 0 | Yes | DDMMMYYYY (xx) | No | | | | |
| | | Week 2 | Yes | DDMMMYYYY (xx) | No | | | | |
| | | Week 4 | Yes | DDMMMYYYY (xx) | No | | | | |
| | | (Continue fo | or all clinic visits) | | | | | | |

Programming Note: For multiple Abnormal Findings within a Body System, separate text using a ";". Use data from SDTM.PE. If Clinic Visit = 'WEEK 0' assign 'Day 0'.

CONFIDENTIALPage 40 of 51

<sup>[1]</sup> Study Day is calculated relative to the date of the first dose of study drug.

<sup>[2]</sup> For Screening Visit, any abnormal findings are presented; for other visits, newly diagnosed or worsened clinically significant findings since previous visit are indicated.

Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4) PCN Number: MIRU8967

### Listing 16.9.3 12-Lead Safety ECG Safety Population

Treatment: <Maralixibat or Placebo>

| | | | | | Heart | RR | PR | QRS | Uncorrected | | | Investigator | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PFIC | | | ECG | Date/Time | Rate | Interval | Interval | Duration | QT Interval | QTcB | QTcF | Interpretation: | |
| Туре | Subject | Clinic Visit | Performed? | Performed | (bpm) | (ms) | (ms) | (ms) | (ms) | (ms) | (ms) | Abnormality [1] | Comments |
| xxxxx | XXXXXX | Screening | Yes | DDMMMYYYY:hh:mm | 99 | 508 | 120 | 72 | 294 | 438 | 376 | Normal | |
| | | Day 0 | Yes | DDMMMYYYY:hh:mm | xxx | xxx | xxx | XX | xxx | xxx | xxx | A-NCS: xxxxxxxxx | xxxxxxxxxxxxx |
| | | Week 10 | No | | | | | | | | | | |
| | | Week 26 | Yes | DDMMMYYYY:hh:mm | XX | XXX | XXX | XXX | XXX | xxx | XXX | xxxxxxxx | xxxxxxxxxxxxx |
| xxxxx | XXXXXX | Screening | Yes | DDMMMYYYY:hh:mm | xxx | XXX | XXX | xxx | xxx | XXX | xxx | xxx: xxxxxxxxxx | |
| | | Day 0 | Yes | DDMMMYYYY:hh:mm | xxx | xxx | xxx | XXX | xxx | xxx | xxx | XXXXXXXX | |
| | | Week 10 | Yes | DDMMMYYYY:hh:mm | XX | xxx | xxx | XXX | xxx | xxx | xxx | XXXXXXXX | |
| | | Week 26 EOT | Yes | DDMMMYYYY:hh:mm | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXXXXXXX | |

Abbreviations: QTcB = QT interval corrected using Bazett's formula; QTcF = QT interval corrected using Fridericia's formula [1] A-NCS = Abnormal-Not Clinically Significant; A-CS = Abnormal-Clinically Significant

**Programming Note:** Use data from CRF.EG.

CONFIDENTIALPage 41 of 51

Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

## Listing 16.10.1 Clinical Laboratory Tests: Clinical Chemistry Safety Population

Treatment: <Maralixibat or Placebo>

| | | | | | | Local | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PFIC | | Age [1]/ | Laboratory | Clinic | Collection Date | Lab?/ | Fasting? | Test | _ | Rete | rence Rai | nge |
| Гуре | Subject | Sex | Test | Visit | (Study Day) [2] | Visit [3] | [4] | Result [5] | Units | Low | Standard erence Ra High xx | [6] |
| xxxx | XXXXXX | xx/M | xxxxxxxxxxxxx | Screening | DDMMMYYYY (-x) | No | Υ | xxx | XXX | XX | xx | |
| | | | | Day 0 | DDMMMYYYY (x) | No | Υ | xxx | XXX | XX | XX | Х |
| | | | | Week 2 | DDMMMYYYY (xx) | Yes/Week 2 | Υ | xxx | XXX | XX | xx | |
| | | | | Week 6 | DDMMMYYYY (xx) | xx | Υ | xxx | XXX | XX | XX | |
| | | | | Week 10 | DDMMMYYYY (xx) | xx | Υ | xxx | XXX | XX | XX | |
| | | | | Week 14 | DDMMMYYYY (xxx) | xx | Υ | xxx | XXX | XX | XX | |
| | | | | Week 18 | DDMMMYYYY (xxx) | xx | Υ | xxx | XXX | XX | XX | |
| | | | | Week 22 | DDMMMYYYY (xxx) | xx | U | xxx | XXX | XX | XX | |
| | | | | Week 26 | DDMMMYYYY (xxx) | XX | Υ | XXX | XXX | XX | XX | Х |

- [1] Age (years) at Baseline.[2] Study Day is calculated relative to the date of the first dose of study drug.
- [3] Were the labs collected for a protocol-related visit in place of central lab collection?/If yes, for which visit?
- [4] Y = Yes; N = No; U = Unknown
- [5] 'x' indicates a concentration reported as below the minimum quantitation limit. Half of the minimum quantitation limit is used as the analysis value. '+' indicates a concentration reported as above the maximum quantitation limit. The maximum quantitation limit is used as the analysis value. UNL = Unlabeled; SNS = Sample Not Submitted; QNS = Quantity Not Sufficient; NSA = Not Suitable for Analysis; NCAL = Not Calculated
- [6] H = (High) The result is above the upper limit of the reference range for normal subjects; L = (Low) The result is below the lower limit of the reference range for normal subjects.

**Programming Note:** Sort lab records (within subject) by laboratory test and then by collection date. See Appendix 1 of SAP for listing of safety lab tests. Use data from SDTM.LB since labs from all vendors will be consolidated there.


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

Listing 16.10.2
Clinical Laboratory Tests: Hematology
Safety Population

#### Same shell as Listing 16.10.1

Listing 16.10.3 Clinical Laboratory Tests: Urinalysis Safety Population

Same shell as Listing 16.10.1 except remove Local Lab?/Visit column and adjust footnotes accordingly.

Listing 16.10.4
Clinical Laboratory Tests: Lipid Soluble Vitamins
Safety Population

Same shell as Listing 16.10.1

Listing 16.10.5 Clinical Laboratory Tests: Lipid Panel Safety Population

Same shell as Listing 16.10.1

Listing 16.10.6 Clinical Laboratory Tests: Hepatocellular Carcinoma Marker – Alpha-Fetoprotein (AFP) Safety Population

Same shell as Listing 16.10.1 except remove Local Lab?/Visit column and adjust footnotes accordingly


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

### Listing 16.10.7 Clinical Laboratory Tests: Timing of Sample Collection and Last Meal Safety Population

Treatment: <Maralixibat or Placebo>

| | | | | Date of | Date/Time of |
|---|---|---|---|---|---|
| PFIC | | Age [1]/ | Clinic | Sample Collection | Last Meal Prior to |
| Туре | Subject | Sex | Visit | (Study Day) [2] | Sample Collection [3] |
| xxxxx | XXXXXX | xx/M | Screening | DDMMMYYYY (-x) | |
| | | | Day 0 | DDMMMYYYY (x) | |
| | | | Week 2 | DDMMMYYYY (xx) | DDMMMYYYY:hh:mm |
| | | | Week 6 | DDMMMYYYY (xx) | DDMMMYYYY:hh:mm |
| | | | Week 10 | DDMMMYYYY (xx) | DDMMMYYYY:hh:mm |
| | | | Week 14 | DDMMMYYYY (xx) | DDMMMYYYY:hh:mm |
| | | | Week 18 | DDMMMYYYY (xxx) | DDMMMYYYY:hh:mm |
| | | | Week 22 | DDMMMYYYY (xxx) | DDMMMYYYY:hh:mm |
| | | | (Continue fo | r all clinic visits) | |

<sup>[1]</sup> Age (years) at Baseline.

**Programming Note:** For Date/Time columns, may not need to add footnote. For example, "Date/Time of Last Meal Prior to Sample Collection data is collected on the Case Report Form. In cases where an unscheduled visit has the same date/time as a scheduled visit, the Date/Time of Last Meal Prior to Sample Collection was merged in by Sample Collection Date." Use data from CRF.LB.


<sup>[2]</sup> Study Day is calculated relative to the date of the first dose of study drug.

<sup>[3]</sup> Date/time of last meal prior to sample collection is collected on the Case Report Form. In cases where an unscheduled visit has the same date/time as a scheduled visit, the Date/Time of Last Meal Prior to Sample Collection were merged in by Sample Collection Date.

Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

Listing 16.10.8 Microbiology Tests Safety Population

### Treatment: <Maralixibat or Placebo>

| PFIC<br>Type | Subject | Age [1]/<br>Sex | Clinic<br>Visit | Collection Date<br>(Study Day) [2] | Microbiology<br>Test | Test<br>Result [3] | Units |
|---|---|---|---|---|---|---|---|
| | - | | | | | | |
| XXXXX | XXXXXX | xx/M | Screening | DDMMMYYYY (-x) | xxxxxxxxxxxxx | xxx | xxx |
| | | | Day 0 | DDMMMYYYY (x) | | XXX | XXX |
| | | | Week 2 | DDMMMYYYY (xx) | | xxx | XXX |
| | | | Week 6 | DDMMMYYYY (xx) | | xxx | XXX |
| | | | Week 10 | DDMMMYYYY (xx) | | XXX | XXX |
| | | | Week 14 | DDMMMYYYY (xxx) | | XXX | XXX |
| | | | Week 18 | DDMMMYYYY (xxx) | | xxx | XXX |
| | | | Week 22 | DDMMMYYYY (xxx) | | xxx | XXX |
| | | | Week 26 | DDMMMYYYY (xxx) | | xxx | XXX |
| | | | | (Continue for all clin | nic visits) | | |

<sup>[1]</sup> Age (years) at Baseline.

**Programming Note:** Sort microbiology records (within subject) by microbiology test and then by collection date. Include LBCAT = 'EBV PANEL', 'HCV RNA (PCR)', HEP B SURFACE AG', 'HEP C ANTIBODY', 'HEPATITIS A AB, IGM'. Use data from SDTM.MB.


<sup>[2]</sup> Study Day is calculated relative to the date of the first dose of study drug.

<sup>[3]</sup> UNL = Unlabeled; SNS = Sample Not Submitted; QNS = Quantity Not Sufficient; NSA = Not Suitable for Analysis; NCAL = Not Calculated

Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

Listing 16.10.9
Pregnancy Tests
Safety Population

Treatment: <Maralixibat or Placebo>

| | | Age [1]/ | | Sample<br>Collected?/ | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| PFIC | | Childbearing | Clinic | Reason Not | Collection Date/Time | Fasting? | Sample | Test | |
| Туре | Subject | Potential | Visit | Collected? | (Study Day) [2] | [3] | Туре | Result | Units |
| xxxxx | XXXXXX | XX/Yes | Screening | Yes | DDMMMYYYY:hh:mm (-x) | х | Serum | xxx | xxx |
| | | | Day 0 | Yes | DDMMMYYYY:hh:mm (x) | Х | Urine | NEGATIVE | |
| | | | Week 4 | No/xxxxxxx | | | | | |
| | | | Week 10 | Yes | DDMMMYYYY:hh:mm (xx) | Χ | Urine | NEGATIVE | |
| | | | Week 18 | Yes | DDMMMYYYY:hh:mm (xx) | Χ | Urine | NEGATIVE | |
| | | | Week 26 | Yes | DDMMMYYYY:hh:mm (xxx) | X | Urine | NEGATIVE | |
| xxxxx | XXXXXX | XX/xxx | Screening | NA | | | | | |
| | | | Day 0 | NA | | | | | |
| | | | Week 4 | Yes | DDMMMYYYY:hh:mm (xx) | Χ | Urine | NEGATIVE | |
| | | | Week 26 EOT | NA | | | | | |
| | | | (Continue for a | ll clinic visits) | | | | | |

Abbreviation: NA = not applicable

Note: Listing for female subjects only; only females with at least 1 pregnancy test sample are included in the listing.

**Programming Note:** Listing should only include female subjects for which at least 1 pregnancy sample was collected. For these subjects, include each clinic visit.

Use data from SDTM.LB.


<sup>[1]</sup> Age (years) at Baseline.

<sup>[2]</sup> Study Day is calculated relative to the date of the first dose of study drug.

<sup>[3]</sup> Y = Yes; N = No; U = Unknown

Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

# Listing 16.10.10 Plasma Sample Maralixibat Concentrations Safety Population

Treatment: <Maralixibat or Placebo>

| | | | | | | | Date/Time of | |
|---|---|---|---|---|---|---|---|---|
| | | | | | | | Last Meal Prior | Maralixibat |
| PFIC | | Clinic | | Sample | Reason Not | Collection | to Sample | Concentration |
| Туре | Subject | Visit | Time Point | Collected? | Collected | Date/Time | Collection | (ng/mL) |
| xxxx | XXXXXX | Week 10 | PRE-DOSE | Yes | | DDMMMYYYY:hh:mm | | BLQ |
| | | | +2.5H | Yes | | DDMMMYYYY:hh:mm | DDMMMYYYY:hh:mm | XX.XX |
| | | Week 26 | PRE-DOSE | Yes | | DDMMMYYYY:hh:mm | DDMMMYYYY:hh:mm | XX.XX |
| | | | +2.5H | No | xxxxxx xxxx xxx | | | |
| xxxx | XXXXXX | Week 10 | PRE-DOSE | | | DDMMMYYYY:hh:mm | DDMMMYYYY:hh:mm | BLQ |
| | | | +2.5H | | | DDMMMYYYY:hh:mm | DDMMMYYYY:hh:mm | BLQ |
| | | Week 26 EOT | PRE-DOSE | | | DDMMMYYYY:hh:mm | DDMMMYYYY:hh:mm | BLQ |
| | | | +2.5H | | | DDMMMYYYY:hh:mm | DDMMMYYYY:hh:mm | BLQ |

Abbreviations: LLOQ = lower limit of quantitation; BLQ = below quantification limit Note: LLOQ is 0.250 ng/mL. Any concentration below the LLOQ is reported as BLQ.

**Programming Note:** Use data from CRF.PK.


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

# Listing 16.11 Telephone Contact Log Intent-to-Treat Population

Treatment: <Maralixibat or Placebo>

| | | | Subject/ | | Telephone/Email | Any New/ | Report new |
|---|---|---|---|---|---|---|---|
| PFIC | | | Caregiver | Reason Not | Contact Date | Worsening | Concomitant |
| Туре | Subject | Time Point | Contacted? | Contacted | (Study Day) [1] | AEs/SAEs? | Medications |
| xxxxx | XXXXXX | Week 1 | Yes | | DDMMMYYYY (x) | No | No |
| | | Week 3 | Yes | | DDMMMYYYY (xx) | No | No |
| | | Week 5 | No | XXXXXXXXX XXXXX | | | |
| | | Week 8 | Yes | | DDMMMYYYY (xx) | No | No |
| | | Week 12 | Yes | | DDMMMYYYY (xx) | No | No |
| | | Week 16 | No | XXXXXX XXXX | | | |
| | | Week 20 | Yes | | DDMMMYYYY (xx) | No | No |
| | | Week 24 | Yes | | DDMMMYYYY (xx) | Yes | Yes |
| | | Follow-up | Yes | | DDMMMYYYY (NT) | No | No |

(Continue for all time points)

Abbreviation: AEs = Adverse Events; SAEs = Serious Adverse Events

[1] Study Day is calculated relative to the date of the first dose of study drug

Programming Note: If subject was never dosed, Study Day will be reported as "(NT)". Use data from CRF.TC1.


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

# Listing 16.12 Visit Dates and Type Intent-to-Treat Population

Treatment: <Maralixibat or Placebo>

| | | | | | Homecare | | Continuing |
|---|---|---|---|---|---|---|---|
| PFIC | | | Visit Date | Type of | Used?/If No, | Date of Call | to |
| Туре | Subject | Time Point | (Study Day) [1] | Visit | Explain | | Next Visit |
| XXXXX | XXXXXX | Screening | DDMMMYYYY (x) | In Clinic | | DDMMMYYYY | Yes |
| ***** | 70000 | Baseline (Week 0) | DDMMMYYYY (x) | In Clinic | | DDIVIIVIIVII | Yes |
| | | Subject Contact (Week 1) | DDMMMYYYY (x) | Telephone | | | xxx |
| | | Visit 2 (Week 2) | DDMMMYYYY (x) | Remote | Yes | | XXX |
| | | Subject Contact (Week 3) | DDMMMYYYY (x) | XXX | | | XXX |
| | | Visit 3 (Week 4) | DDMMMYYYY (x) | XXXXXX | | | |
| | | | DDMMMYYYY (x) | xxxxx | | | |
| xxxxx | XXXXXX | Screening | DDMMMYYYY (x) | xxxxxxx | | | xxx |
| | | Baseline (Week 0) | DDMMMYYYY (x) | xxxxx | | | XXX |
| | | Subject Contact (Week 1) | DDMMMYYYY (x) | xxxxxx | | | XXX |
| | | Visit 2 (Week 2) | DDMMMYYYY (x) | XXXXXX | | | No |
| | | Early Termination | DDMMMYYYY (x) | | | | |

<sup>[1]</sup> Study Day is calculated relative to the date of the first dose of study drug.

**Programming Note:** Use data from CRF.SV, CONT.


Listing Shells Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4) PCN Number: MIRU8967

### Listing 16.13 Healthcare Utilization Intent-to-Treat Population

Treatment: <Maralixibat or Placebo>

| PFIC<br>Type | Subject | Any<br>Medical<br>Visits? | Type of<br>Visit | Reason for Visit | Admitted<br>to<br>Hospital? | Date of<br>Admission | Date of<br>Surgery/<br>Procedure | Date of<br>Discharge | Discharge<br>Status | Number of<br>Work Days<br>Caregiver<br>Missed |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxx | XXXXXX | No | | | | | | | | |
| xxxxx | XXXXXX | Yes | OUTPATIENT | XXXXXXXXXXXXX | Yes | DDMMMYYYY | DDMMMYYYY | DDMMMYYYY | OTHER: xxxxxxxxxxx | xx |
| | | Yes | XXXXXXXXX | XXXXXXXXXXXX | xxx | DDMMMYYYY | | DDMMMYYYY | | xx |

**Programming Note:** Use data from CRF.HU.


Sponsor: Mirum Pharmaceuticals Inc. Protocol: MRX-502 (Amendment 4)

PCN Number: MIRU8967

Treatment: <Maralixibat or Placebo>

XXXXX

### Listing 16.14 COVID-19 Impact Intent-to-Treat Population

Subject Missed Study Study Affected by/ Type of Assessments? Drug Drug Visit Impacted Visit Efficacy/ Dispensation Administration Additional PFIC ET Reason/ How IP Start Date/ Type Subject by COVID-19? Adjustment Time Point Safety Comments **Impacted End Date** Change Change Comments XXXXXX Yes/Week 14 Yes/Yes Missed **DDMMMYYYY XXXXXXXXXXX** XXXXX Yes/Week 18 Performed via **DDMMMYYYY** No/No Dispensation DDMMMYYYY/ Delivered to telephone Change DDMMMYYYY subject offsite Yes/Week 26 Other: xxxxxxxxxx **DDMMMYYYY** xx/xxx DDMMMYYYY/ XXXXXX **DDMMMYYYY** XXXXXX No

Abbreviations: ET = early termination; IP = investigational product

XXXXXX Yes/Week 10 Missed

Programming Note: If Other, specify is present in data, concatenate Other with specify data (e.g., Other: xxxxxx). Use data from CRF.COVID.

Subject Decision/

XXXXXXXXXXX

Dosing

Interruption

DDMMMYYYY/

**DDMMMYYYY** 

xxxxxxxxxx


**DDMMMYYYY** 

Yes/Yes